Replication of Effects of the angiotensin-receptor blocker telmisartan on cardiovascular events in high-risk patients intolerant to angiotensin-converting enzyme inhibitors: a randomised controlled trial (TRANSCEND trial)

May 13, 2020

#### RCT Details

This section provides a high-level overview of the RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Effects of the angiotensin-receptor blocker telmisartan on cardiovascular events in high-risk patients intolerant to angiotensin-converting enzyme inhibitors: a randomised controlled trial (TRANSCEND trial)

#### 1.2 Intended aim(s)

The primary objective of the study is to determine if treatment with telmisartan 80mg daily is superior to placebo reducing the composite endpoint in patients who are intolerant to Angiotension Converting Enzyme inhibitors.

## 1.3 Primary endpoint for replication and RCT finding

Cardiovascular Death, Non-fatal Myocardial Infarction, Non-fatal Stroke and Hospitalization for Congestive Heart Failure

## 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

An overall sample size of 6000 patients was expected to have 94% power to detect a hazard ratio of 0.81 for telmisartan compared with placebo at a two-sided alpha of 0.05.

### 1.5 Primary trial estimate targeted for replication

HR = 0.92 (95% CI 0.81-1.05) comparing telmisartan to placebo (Yusuf et al., 2008, Lancet)

#### 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D. implemented the study design in the Aetion Evidence Platform. S/he is not responsible for the validity of the design and analytic choices. All implementation steps are recorded and the implementation history is archived in the platform.

## 3. Data Source(s)

United/Optum, MarketScan

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

#### Design Diagram - TRANSCEND TRIAL REPLICATION



#### 5. Cohort Identification

## 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing telmisartan to other antihypertensives, including loop diuretics, thiazides, and dihydropyridines. Although the trial compared telmisartan with placebo added to usual care, we selected an active comparator for this study because non-user comparator groups are known to often lead to confounding by indication and biased treatment effect estimates. This group of other antihypertensives were selected as the primary comparator because intolerance to ACEi was a primary inclusion criteria for the trial. Therefore, patients in both arms were on a mix of non-ACEi and non-ARB antihypertensives as background therapy.

The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of telmisartan or a comparator drug (cohort entry).

#### 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

### 5.2.1 Eligible cohort entry dates

Market availability of telmistartan in the U.S. started on November 10, 1998, however, the Marketscan and Optum data are available at BWH only from Jan 1, 2003 and Jan 1, 2004, respectively.

- For Marketscan: Jan 1, 2003 -Dec 2017 (end of data availability).
- For Optum: Jan 1, 2004-June 30, 2019 (end of data availability).

## 5.2.2 Specify inclusion/exclusion criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

## 5.3 Flowchart of the study cohort assembly

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| | Optum | | MarketScan | |
|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less Excluded Patients | Remaining<br>Patients |
| All patients in the database | | 75,524,500 | | 191,990,035 |
| Did not meet cohort entry criteria | -75,483,721 | 40,779 | -191,937,915 | 52,120 |
| Final cohort | | 40,779 | | 52,120 |

#### 6. Variables

#### 6.1 Exposure-related variables:

## Study drug:

The study exposure of interest is initiation of telmisartan. Initiation will be defined by no use of telmisartan or a comparator in the prior 6 months before treatment initiation (washout period).

#### Comparator agents-

- · Initiators of telmisartan will be compared to initiators of-
  - Loop/Dihydropyridines/Thiazides

### 6.2 Preliminary Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the default baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B). These covariates are based on those used by Patorno et al. (2019).

## 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- <u>Primary outcome</u>: Composite of non-fatal myocardial infarction, non-fatal stroke, or CV mortality, hospital admission for heart failure
- Secondary outcomes: Individual components:
  - o Hospital admission for heart failure
  - o Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  - Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  - All-cause mortality/CV mortality:
    - Information on CV mortality through data linkage with the National Death Index (NDI) will only be available for Optum Clinformatics.
    - All-cause inpatient mortality identified using discharge status codes will be used as a proxy for "CV mortality" in commercial databases

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on day of cohort entry. Because adherence in the real world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of telmisartan and comparator and will continue until the earliest date of the following events:

- · The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission

- Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (telmisartan
  and comparator) plus a defined grace period (i.e., 30 days after the end of the last prescription's days' supply in main
  analyses).
- The date of augmentation or switching from the comparator group to the exposure group (initiation of telmisartan in the comparator group).

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

## 7. Initial Feasibility Analysis

#### Aetion report name:

Optum- https://bwh-dope.aetion.com/projects/details/868/results/52960/result/14

MarketScan- https://bwh-dope.aetion.com/projects/details/853/results/52961/result/14

## Date conducted: 04/27/2020

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Complete study flowchart from Section 5.3
- Report patient characteristics by treatment group
- Report summary parameters of study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

#### Aetion report name:

Optum- https://bwh-dope.aetion.com/projects/details/868/results/37656/result/0
MarketScan- https://bwh-dope.aetion.com/projects/details/853/results/37657/result/0

Date conducted: 08/04/2019

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the
analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons
for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and
reported in the subsequent sections, after incorporating feedback and refining the protocol.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 8/16/19 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 8/31/19 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

#### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/868/results/52962/result/0">https://bwh-dope.aetion.com/projects/details/868/results/52962/result/0</a>
MarketScan- <a href="https://bwh-dope.aetion.com/projects/details/853/results/52963/result/0">https://bwh-dope.aetion.com/projects/details/853/results/52962/result/0</a>

Date conducted: 04/27/2020

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

· Provide plot of PS distributions stratified by treatment group.

Note- Please refer to Appendix B.

Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 303 (0.76%) | 214 (1.07%) | 89 (0.44%) |
| Switch from referent drug to<br>telmisartan | 104 (0.26%) | 104 (0.52%) | 0 (0.00%) |
| Discontinuation of telmisartan | 9,119 (22.77%) | 0 (0.00%) | 9,119 (45.54%) |
| Specified date reached | 7,198 (17.97%) | 3,903 (19.49%) | 3,295 (16.46%) |
| End of patient enrollment | 6,003 (14.99%) | 3,976 (19.86%) | 2,027 (10.12%) |
| Discontinuation of<br>Loop/Dihydropyridines/Thiazides<br>+ nursing home + Pharmacy<br>disenrollment | 17,321 (43.25%) | 11,827 (59.06%) | 5,494 (27.44%) |

· Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | |
|------------------------------------|--------------|--------------|
| Patient Group Optum MarketScan | | |
| Overall Patient Population | 113 [59-229] | 150 [77-380] |

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Referent | 122 [66-304] | 204 [84-522] |
|----------|--------------|--------------|
| Exposure | 106 [58-178] | 118 [66-273] |

· Report overall risk of the primary outcome.

| | Optum | Marketscan | Pooled |
|---|---|---|---|
| Risk per 1,000 patients (Composite endpoint including death | | | |
| from cardiovascular causes, myocardial infarction, stroke, and | | | |
| hospitalization for heart failure) | 51.95 | 73.72 | 64.1 |

#### 9.1 Final Power Assessment

Date conducted: 04/27/2020

- Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9.
   All other parameters in the table should be the same as in Section 8. If the study is to be implemented in more than one database, copy and paste excel sheet to report power for each database separately and for the pooled analysis that uses data from all databases together. Power calculations are based on the formulas from Chow et al. (2008).
  - Pooled

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | |
| Reference | 20,024 |
| Exposed | 20,024 |
| Risk per 1,000 patients | 64.10 |
| Desired HR from RCT | 0.81 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 2567.0768 |
| Power | 0.999635278 |

## Optum

| 8,710 |
|-------------|
| 8,710 |
| 51.95 |
| 0.81 |
| 0.05 |
| 904.969 |
| 0.886777233 |

#### MarketScan

| Superiority Analysis | |
|----------------------------|-------------|
| Number of patients matched | |
| _ | |
| Reference | 11,314 |
| Exposed | 11,314 |
| Risk per 1,000 patients | 73.72 |
| Desired HR from RCT | 0.81 |
| Alpha (2-sided) | 0.05 |
| Number of events expected | 1668.13616 |
| Power | 0.990441892 |

Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of
advisory board. Reviewers evaluate the results of the analyses described above in Sections 9 and 10, including numbers of
patients, balance in patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates
of outcomes and study power.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 5/13/20 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 3/20/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

## 10. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u>
<u>Date votes and concerns are summarized:</u>

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

### 11. Register study protocol on clinicalTrials.gov

#### Date conducted:

Register the study on <u>clinicalTrials.gov</u> and upload this document.

#### 12. Comparative Analyses

#### Aetion report name:

Date conducted:

## 12.1 For primary analysis:

• In the PS-matched cohort of telmisartan and loop/dihydropyridines/thiazides\_initiators from Section 9, calculate the HR for each outcome for telmisartan versus referent patients using a Cox proportional hazards model.

#### 12.2 For secondary analyses:

## 13. Requested Results

#### 13.1 Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | | After adjusti | nent | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |

Effectiveness research with Real World Data to support FDA's regulatory decision making

| Age categories |
|----------------|

## 13.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

## 13.3 Table 3: Censoring events

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

## 13.4 Table 4: Results from primary analyses;

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

Effectiveness research with Real World Data to support FDA's regulatory decision making: Protocol Template

HR, Hazard Ratio; CI, Confidence Interval.

## 13.5 Table 5: Results from secondary analyses;

#### 14. References

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Patorno E, Pawar A, Franklin JM, et al. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISE) Study. Circulation. 2019; in press. (https://www.ahajournals.org/doi/pdf/10.1161/CIRCULATIONAHA.118.039177)

| # | # TRANSCEND trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| | Trial details- 3- Failed 5- No Ni margin specified - 3 : | weeks run in | Pie see see the following Google Drive for further details or any missing information: https://drive.google.com/open?id=1WD63itwnge//idaXeft.TcuX-VCmb6b-gV/ | Diteria |
| | EXPOSURE vs. COMPARISON | | ICD-10 codes are not listed in this document because of excel cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will be swellable in the above Google Ports Folder (link above). ICD-01 to ICD-01 code conversions were completed using a SAS macro that implements forward/ backward mapping based on the CMS ICD-0 to ICD-10 mapping: <a href="https://www.nbsr.cres/data/lcd0-1cd-10-cm-md-pcs-rosswall-gaseral-equivalence-mapping.html">https://www.nbsr.cres/data/lcd0-1cd-10-cm-md-pcs-rosswall-gaseral-equivalence-mapping.html</a> | Adequate mapping in claims |
| | TRANSCEND: Almed to determine if telmisertan is superior to placebo in patients who are intolerant of ACE inhibitors No Loc | or Transcend trial, Inhisatran + Loop/Dihydropyridines/Thiazides vs. oop/Dihydropyridines/Thiazides (Please see Comparison sheet for drug list) ew-use of Telmisartan (Exposure group) PLUS oop/Dihydropyridines/Thiazides (days supply overlap on the index date) vs. ew-use of Loop/Dihydropyridines/Thiazides (Reference group) | | Intermediate mapping in claims |
| | PRIMARY OUTCOME | | | Poor mapping or cannot be measured in claims. |
| | lang Could life Country of the Count | petitent cars acting: smooth in offend mortality/Mi/Stroke/CHF — spirital admission for CHF (Inpetient only, any position) ICD-9 diagnosis: 428.x, 88.93, 402.01, 402.11, 402.91, 404.01, 404.11, 404.93, 404.03, 404.13, 404.93 [[(inpetient only, any position) ICD-9 diagnosis: 410.x excluding 410.x2 roke [Inpetient only, primary position only) ICD-9 diagnosis: 430.xx, 431.xx, 13.x1, 434.xx (excluding 434.x0), 436.x ortality: See Mortality Sheet. | For Mb: →PPV 94% in Medicare claims data Kiyota Y, Schneewelss S, Glynn RJ, Cannuscio CC, Avern J, Solomon DM. Accuracy of Medicare claims-based diagnosis of acute myocardial inferction: estimating positive predictive value on the basis of review of hospital records. American heart journal 2004; 148:99-104.] →PPV 88.4% in commercial ly-insured population (Wahl PM, Rodgers K, Schneewelss S, et al. Validation of claims-based diagnostic and procedure codes for cardiovascular and gastrointestinal serious advance events in a commercially-insured population. Pharmacospiciemiology and Drug Safety 2010;19:396-603.] For atroba: PPV 68.5% or higher for ischemic stroke PPV ranging from 80% to 86% for hemorrhagic stroke →Jendrade SC, Hieroid LE, Tjia J, et al. A systematic review of validated methods for identifying cerebrovascular accident or transler in Ischemic attack using administrative data. Pharmacospidemiology and Drug Safety 2012;21 Suppl 1:100-28.] →Jinchwell CL, Longstreth Wr. Ir. Validation administrative data in stroke research. Stroke; a journal of carebral circulation 2002;31:2465-70.] →Jinchwell CL, Unogstreth Wr. Ir. Validation administrative data in stroke research. Stroke; a journal of carebral circulation 2002;31:2465-70.] →Jinchwell of CD-9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | Can't be measured in claims but not important for the analysis |
| F | INCLUSION CRITERIA | | | |
| - | Individuals 55 years of age with 1 of the following: Age 1 Coronary artery disease | e 255 years at drug initiation | | |
| 10 | Me<br>dia<br>Dia | leasured fores the start of all available data to 2 days prior to drug initiation in any<br>agnosis position and the hipselfent or outpatient care setting<br>valuable (CD-9 diagnosis: 412.xx<br>42.ML (CD-9 diagnosis: 412.xx | Patono, Elisabetta et al. "Cardiovascular outcomes associated with canagliflorin versus other non-gliflorin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patono, Elisabetta et al. "Empagliflorin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliflorin Comparative Effectiveness and Safety (IMP RSZ) Study. "Circulation. 2019 Apr B. doi: 10.1161/CIRCULATIONAHA.118.0391.77 | |
| 1Ь | en<br>Accional | leasured from the start of all available data to 30 days prior to drug initiation in<br>wy diagnosis position and the inpatient or outpatient care setting<br><u>37/3/https://groups.ICP-0-diagnosis</u> : 41.xx<br>able anging ICD-0 diagnosis: 413.xx | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflosin versus other non-gliflosin antidiabetic drugs: population based cohort study." BMU 2015;366k.14 http://dx.doi.org/201.1356/kml, kl.19 Patorno, Elisabetta et al. "Impagliflosin and the Risk of Heart Pallure Mospitalization in Routine Clinical Care: A First Analysis from the Empagliflosin Comparative Effectiveness and Safety (EMP RISE) Study. "Circulation. 2019 Apr E. doi: 10.1161/CIRCULATIONAHA.118.039177 | |

| | | Managed from the start of all models is determined and a second s | |
|---|---|---|---|
| 1e | Multi-vessel PTCA >30 days before informed consent | Measured from the start of all available data to 30 days prior to drug initiation in any procedure position and the care setting indicated below: PTCA [Inpatient only] CPT-4: 29373, 92982, 92984, 92995, 92996, 92920 – 92921, 92924 – 92925, 92937, 92938, 92941, 92943, 92944 [Inpatient on outpatient] ICD-9 procedure: 00.66, 36.03, 36.03, 36.03, 36.05, 36.05 Saming [Inpatient only] CPT-4: 92980, 92981, 92928 – 92929, 92933 – 92934 [Inpatient or outpatient] ICD-9 procedure: 36.05, 36.07 Transmoscaff in resocularization [Inpatient only] CPT-4: 33140, 33141 [Inpatient or outpatient] ICD-9 procedure: 36.31-36.34 | Patorno, Elisabetta et al. "Cardiovecular outcomes associated with canagliflodin versus other non-gliflodin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/pm.k119 Patorno, Elisabetta et al. "Empagliflorin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliflorin Comparative Effectiveness and Safety (EMPS 23) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAMA.118.039177 |
| 1d | Multi-vessel CABG surgery > 4 years before informed consent, or with recurrent angine following surgery | Measured from the start of all evallable data to 1460 days (4 years) prior to drug initiation in any procedure position and the inpatient care setting CASO CPT-4: 33530 – 33536, 33545, 33572. ICD-9 procedure: 36.1x, 36.2x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflodin versus other non-gliflodin antidiabetic drugs: population based cohort study." BMJ 2015;180/k119 http://dx.dol.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflorin and the Risk of Heart Fallure Mospitalization in Routine Clinical Care: A Pirth Analysis from the Empagliflorin Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr II. doi: 10.1161/CRICULATIONAMA.118.039177 |
| 2 | Peripheral artery disease | | |
| 2a | Previous limb bypass surgery or Previous limb bypass surgery or angioplasty | Measured from the start of all available data prior to and including day off day limitation in any procedure position and the inpatient or outpetient care setting Previous limb has an surresview/outs/limb has an surresview/outs/limb has an surresview and setting CPT-4: 33536, 35566, 35570, 35570, 35573, 35583-35587, 35623, 35906, 35660, 35671 Lower-satematic and setting | |
| 2b | Previous limb or foot amputation | Measured from the start of all available data prior to and including day of drug initiation in any diagnosis/procedure position and the inpetient or outpatient care setting. Iconomic returns it various action. Iconomic various va | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagificaln versus other non-glifforin antidiabetic drugs: population based cohort study." BMJ 2011;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagificarin and the Risk of Neart Fallure Hospitalization in Routine Clinical Care: A Pint Analysis from the Empagifican Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 2e | Intermittent claudication, with anklearm SP ratio << 0.80 on at least 1 side | Measured from the start of all evaluable data prior to and including day of drug<br>initiation in any diagnosis position and the inpetient or outpatient care setting<br>Adherosciences in finative arteries of the extremities with intermittent claudication.<br>ICD-9 diagnosis: 440.21 | |
| 2d | Significant peripheral artery stenosis ( >50%) documented by angiography or non-invasive testing | Measured from the start of all evallable data prior to and including day of drug initiation as at least two claims on apparate days in any diagnosis/procedure position and the inpatient or outpetient care setting (unless otherwise specified): Preinhers's exactle of Leasure IECD-9 diagnosis: 440.20 – 440.24, 440.29 – 440.32, 440.3, 440.4, 443.9 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflodin versus other non-gliflodin antidiabetic drugs: population based cohort study." BMJ 2016; 360 kl. 19 http://dx.doi.org/10.1136/bm/.kl19 Patorno, Elisabetta et al. "Empagliflodin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflodin Comparative Effectiveness and Safety (EMPRISZ) Study." Circulation. 2019 Apr E. doi: 10.1161/CIRCULATIONAMA.118.039177 |
| - | Cere brovaccular disease | | |
| 3 | Chippion of Control | | |

| 3a<br>3b | Previous stroke Transient ischemic attacks >7 days and <2 year before informed consent | Me soured from the start of all available data prior to and including day of drug initiation in any diagnosis position and the inputient or outpetient care setting Stroke (CD-9 diagnosis: 430.xx, 431.xx, 433.x1, 434.xx (excluding 434.x0), 436.x Measured 365 days prior to drug initiation to 7 days prior to drug initiation in any diagnosis position and the inputient or outpetient care setting TIAI (CD-9 diagnosis: 435.xx | Patorno, Elisabetta et al. "Cardiovaccular outcomes associated with canaglifical neuron estate non-glificaln antidiabetic drugs: population based cohort study." BMJ 2012; 3604:19 http://ex.doi.org/10.1136/bmj.1119 Patorno, Elisabetta et al. "Empaglifical and the Risk of Heart Fallure Hospitalization in Routine Clinical Care." A Flint Analysis from the Empaglifical no Comparative Effectiveness and Safety (EMPS) Study." Circulation. 2019 Apr E. doi: 10.1161/CRCULATIONAMA.118.039177 |
|---|---|---|---|
| 4 | Diabetus me liitus | | |
| 4 | Diabetes mellitus High-risk diabetics with evidence of endorgen damage | Measured at the start of all evallable data prior to and including day of drug initiation in any disposals position and the lapstient or outpetient care setting Disbetic entangleshy (CD-9 diagnosis 35.2.0. Disbetic entangleshy (CD-9 diagnosis 25.0.5 kg (without martion of 35.0.2.0.3.0.0.0.7) 36.6.1., 365.4. Disbetic nearbroathy (CD-9 diagnosis: 250.4x, 583.81 Disbetic nearbroathy (CD-9 diagnosis: 250.4x, 583.81 Disbetic nearbroathy (CD-9 diagnosis: 250.6x, 357.2x, 337.1 Disbetic nearbroathy (CD-9 diagnosis: 707.1x | Patorno, Elisabetta et al. "Cardiovaccular outcomes associated with canaglifical newsus other non-gifficol natidiabetic drugs: population based cohert study." BMJ 2011;396x119 http://dx.doi.org/20.1136/pmj.1219 Patorno, Elisabetta et al. "Empaglifical and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A First Analysis from the Empaglificain Comparative Effectiveness and Safety (EMPISS) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAMA.118.039177 |
| | | Exclusion criteria | |
| 1 | | N/A | |
| 1a | Inability to discontinue ACE inhibitors or ARB | N/A | |
| 1b | Enown hypersensitivity or intolerance to ACE inhibitors or ARB (patient intolerant of ACE inhibitor can be enrolled in<br>TRANSCEND) | N/A | |
| 2 | Cardiovascular disease (HF) | | |
| 2<br>2a | Cardiovascular disease (HF) Synsptomatic congestive heart failure | Measured 180 days prior to and incuding day of drug initiation in any diagnosis position and the inpatient/emergency room care setting-linear full used (serous) requiring hospitalization. ICD-9 diagnosis: 4218, 388,91,402.01,402.11,402.91,404.01,404.01,404.11,404.91,404.03,404.13,404.03,404.13,404.03,404.13,404.03,404.13,404.03,404.13,404.03,404.13,404.03,404.13,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,404.03,4 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflodin versus other non-gliflodin antidiabetic drugs: population based cohort study." BMJ 2018;360:k139 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflodin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflodin Comparative Effectiveness and Safety (EMPISS) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAMA.118.039177 |
| | | position and the input intermediate process are setting-<br>ticast full used intermediate in breat full used in 10.2.01, 404.01, | versus other non-gliftodin antidiabetic drugs: population based cohort study," BMI 2018;380:k119 http://dx.doi.org/10.1136/bm/.k119 Patomo, Elisabetta et al. "Empagliftodin and the Risk of Heart Failure Hospitalization in Routine Clinical Care. A First Analysis from the Empagliftosin Comparative Effectiveness and Safety (EMPSE) Study." Circulation. 2019 Apr E. doi: |
| 2a | Symptomatic congestive heart fallure | position and the inpatient/emergencyroom care setting-<br>ticart fail und identification in the best initiation. ICD-9 diagnosis: 428.x, 398.91.402.01, 402.11, 402.91, 404.01, 404.11, 404.91,<br>404.03, 404.13, 404.93. ICD-10 diagnosis: 92.81, 111.0, 133.0, 133.2, 150.1, 150.20, 150.21, 150.22, 150.23,<br>150.31, 150.32, 150.33, 150.40, 150.41, 150.42, 150.43, 150.9 Measured 180 days prior to and including day of drug initiation in any diagnosis position and the inpatient or outpetient care setting Various and Setting of the Inpatient of Companies 745.4x Insectro bits Cardiamonathy ICD-0 diagnosis: 425.1x Statisticart valval a heart disease ICD-0 diagnosis: 374.x, 385.x, 385.x, 397.x, 398.9x, V42.2, V43.3 ICD-0 grocedure: 35.1x, 35.2x ICD-0 grocedure: 35.1x, 35.2x | waraus other non-gliftodin antidiabetic drugs: population based cohort study." BMJ<br>2018;380:k119 http://dx.doi.org/10.1118/bm/.k119 Patomo, Elisabetta et al. "Empagliflodin and the Risk of Heart Failure Hospitalization<br>in Routine Clinical Care: A First Analysis from the Empagliflodin Comparative<br>Effectiveness and Safety (EMPSE) Study." Circulation. 2019 Apr E. doi: |

| | | Measured 90 days prior to and incuding day of drug initiation in any diagnosis | |
|---|---|---|---|
| | | position and the inpatient or outpatient care setting | |
| 2e | Syncopal episodes of unknown etiology <3 months before informed consent | Syncope and collapse ICD-9 diagnosis: 780.2 | |
| w | Planned cardiac surgery or PTCA <3 months of informed consent | N/A | |
| 41 | Parties Cardia: largery of PTLA G months of informed consent | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| | | position and the inpatient or outpetient care setting | |
| 24 | Uncontrolled hypertension on treatment (eg. BP >150/100 mm Hg) | Malignant Hypertension ICD-9 diagnosis: 401.0, 402.0, 402.00, 402.01, 403.0, | |
| - | | | |
| | | 403.00, 403.01, 404.0, 404.00, 404.01, 404.02, 404.03, 405.0, 405.01, 405.09 | |
| | | Measured 180 days prior to and incuding day of drug initiation in any | |
| | | diagnosis/procedure position and the inpetient or outpetient care setting | |
| 25 | | Heart transplantation | |
| 4 | Heart transplant recipient | ICD-9 diagnosis: V42.1 | |
| | | ICD-9 procedure: 37.51 | |
| | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| | | position and the inpatient or outpetient care setting | |
| 2g | Stroke due to subarachnoid hemorrhage | Subarachnoid hemorrhage (SAH) ICD-9 diagnosis: 430.xx | |
| 3 | Other conditions | | |
| | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| 30 | Significant renal artery disease | position and the inpatient or outpetient care setting | |
| | | Renovascular hypertension ICD-9 diagnosis: 405.01, 405.11, 405.91, 440.1 | |
| | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| | | position and the inpatient or outpatient care setting | |
| _ | | Hepatitis ICD-9 diagnosis: 070.0, 070.1, 070.20, 070.21, 070.30, 070.31, 070.41, | |
| 36 | Hepatic dysfunction | 070.51 | |
| | | Chronic liver disease and cirrhosis ICD-9 diagnosis: 571.x, 572.x, 573.x | |
| 3: | Uncorrected volume or sodium depletion | N/A | |
| | | Measured 150 days prior to and incuding day of drug initiation in any diagnosis | |
| | | position and the inpatient or outpatient care setting | |
| 34 | Primary hyperaldosteronism | Hyperaldosteronism ICD-9 diagnosis: 255.10 | |
| | | Measured 180 days prior to and incuding day of drug initiation in any diagnosis | |
| _ | | position and the inpatient or outpatient care setting | |
| 3e | Hereditary fructose intolerance | Hereditary Fructose Intolerance ICD-9 diagnosis: 271.2 | |
| | | | Gagne, Josh Jet. al. "'A combined comorbidity score predicted mortality in elderly |
| | | | patients better than existing scores." J Clin Epidemiol. 2011 Jul;64(7):749-59. doi: |
| | Other major noncardiac illness expected to reduce life expectancy or interfere with study participation | Measured 180 days prior to and including day of drug initiation- | 10.1016/j.jclinepi.2010.10.004. |
| 38 | | CCI≥10 | and the second of the second o |
| | | | Sun, Jenny Wet. al. "Validation of the Combined Comorbidity Index of Charlson and |
| | | | Elixhauser to Predict 30-Day Mortality Across ICD-9 and ICD-10." Med Care. 2018 |
| | | | Sep;56(9):812. doi: 10.1097/MLR.0000000000000954. |
| 3g | Simultaneously taking another experimental drug | N/A | |
| | Significant disability precluding regular follow-up visits | N/A | |
| | | | 1 |
| 31 | Unable or unwilling to provide written informed consent | N/A | |

| Trial ID | sNDA8 |
|---|---|
| Trial Name (with web links) | TRANSCEND |
| Trial Name (with pdf links) | TRANSCEND |
| NCT | NCT00153101 |
| Trial category | Secondary indication |
| Therapeutic Area | Cardiology/Vascular Diseases |
| Study batch | Antihypertensives (ARBs+aliskiren) |
| RCT Category | 1a- Intended S with label change |
| Brand Name | Micardis |
| Generic Name | Telmisartan |
| Sponsor | BoehringerIngelheim |
| <u>Year</u> | 2009 |
| Measurable endpoint | Composite endpoint including death from cardiovascular causes, myocardial infarction, stroke, and hospitalization for heart failure |
| Exposure | Telmisartan 80 mg/day |
| Comparator | Placebo |
| <u>Population</u> | 55% Statin, 57% β blocker, 75% aspirin & 79% Antiplatelet users |
| Trial finding | HR = 0.92 (95% CI 0.81–1.05) |
| Notes | |
| No. of Patients | 5926 |
| Non-inferiority margin | - |
| Assay Sens. Outcome | |
| Assay Sens. Endpoint (from trial) | |
| Finding for potential Assay Sens. Outcome from trial- | |
| <u>Power</u> | |
| Blinding | Double-blinded |
| Statistical Method | |
| | Reduction of the risk of myocardial infarction, stroke, or death from cardiovascular causes in patients 55 years of age or older at high risk of developing major cardiovascular events who |
| Approval indication | are unable to take ACE inhibitors |

#### **Loop Diuretics**

BUMETANIDE ETHACRYNIC ACID FUROSEMIDE TORSEMIDE

#### Thiazides

BENDROFLUMETHIAZIDE
CHLOROTHIAZIDE
CHLORTHALIDONE
HYDROCHLOROTHIAZIDE
HYDROFLUMETHIAZIDE
INDAPAMIDE
METHYCLOTHIAZIDE
METOLAZONE
POLYTHIAZIDE

#### Dihydropyridines

AMLODIPINE BESYLATE
CLEVIDIPINE BUTYRATE
FELODIPINE
ISRADIPINE
NICARDIPINE HCL
NIFEDIPINE
NIMODIPINE
NISOLDIPINE

AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM

## Mortality-Dependent on data source. 1. All-cause mortality / inpatient mortality Identified using the vital status file-Medicare Identified using the discharge status codes-Optum- 20 = EXPIRED 21 = EXPIRED TO BE DEFINED AT STATE LEVEL 22 = EXPIRED TO BE DEFINED AT STATE LEVEL 23 = EXPIRED TO BE DEFINED AT STATE LEVEL 24 = EXPIRED TO BE DEFINED AT STATE LEVEL 25 = EXPIRED TO BE DEFINED AT STATE LEVEL 26 = EXPIRED TO BE DEFINED AT STATE LEVEL 27 = EXPIRED TO BE DEFINED AT STATE LEVEL 28 = EXPIRED TO BE DEFINED AT STATE LEVEL 29 = EXPIRED TO BE DEFINED AT STATE LEVEL 40 = EXPIRED AT HOME (HOSPICE) 41 = EXPIRED IN A MEDICAL FACILITY (HOSPICE) 42 = EXPIRED - PLACE UNKNOWN (HOSPICE) Truven- 20 - Died 22 - Died 23 - Died • 24 - Died 25 - Died 26 - Died 27 - Died • 28 - Died 29 - Died • 40 - Other died status or Expired at home (Hospice claims only) (depends on year) 41 - Other died status or Expired in medical facility (Hospice claims only) (depends on year) • 42 - Other died status or Expired - place unknown (Hospice claims only) (depends on year) 21 - Died or Disch./Transf. to court/law enforcement (depends on year)



Figure 60: Post-matching propensity score overlap

Figure 59: Post-matching propensity score overlap

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| | | | | Uni | natched | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Opt | tum | | Tru | ven | | POOL | .ED | |
| Variable | Matched Referent | Exposure-Telmisartan | St. Diff. | Matched Referent | Exposure- | St. Diff. | Matched Referent | Exposure- | |
| Number of patients | 30,558 | 10,187 | | 39,090 | 13,030 | | 69,648 | 23,217 | |
| Age | | | | | | | | | |
| mean (sd) | 71.58 (8.24) | 71.42 (8.51) | 0.02 | 70.44 (9.62) | 70.40 (9.83) | 0.00 | 70.94 (9.04) | 70.85 (9.27) | 0.01 |
| median [IQR] | 72.00 [66.00, 78.00] | 72.00 [65.00, 78.00] | 0.00 | 70.00 [62.00, 78.00] | 70.00 [62.00, 78.00] | 0.00 | 70.88 (9.04) | 70.88 (9.27) | 0.00 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0,000 (0.0%) | #DIV/0! |
| 55 - 64; n (%) | 6,649 (21.8%) | 2,401 (23.6%) | -0.04 | 13,962 (35.7%) | 4,648 (35.7%) | 0.00 | 20,611 (29.6%) | 7,049 (30.4%) | -0.02 |
| 65 - 74; n (%) | 12,245 (40.1%) | 3,909 (38.4%) | 0.03 | 10,959 (28.0%) | 3,697 (28.4%) | -0.01 | 23,204 (33.3%) | 7,606 (32.8%) | 0.01 |
| >=75; n (%) | 11,664 (38.2%) | 3,877 (38.1%) | 0.00 | 14,169 (36.2%) | 4,685 (36.0%) | 0.00 | 25,833 (37.1%) | 8,562 (36.9%) | 0.00 |
| Gender | | | | | | | | | |
| Males; n (%) | 12,556 (41.1%) | 4,187 (41.1%) | 0.00 | 17,427 (44.6%) | 5,809 (44.6%) | 0.00 | 29,983 (43.0%) | 9,996 (43.1%) | 0.00 |
| Females; n (%) | 18,002 (58.9%) | 6,000 (58.9%) | 0.00 | 21,663 (55.4%) | 7,221 (55.4%) | 0.00 | 39,665 (57.0%) | 13,221 (56.9%) | 0.00 |
| Region | | | | | | | | | |
| Northeast; n (%) | 2,784 (9.1%) | 924 (9.1%) | 0.00 | 5,473 (14.0%) | 1,598 (12.3%) | 0.05 | 8,257 (11.9%) | 2,522 (10.9%) | 0.03 |
| South; n (%) | 15,070 (49.3%) | 6,451 (63.3%) | -0.29 | 13,295 (34.0%) | 3,338 (25.6%) | 0.18 | 28,365 (40.7%) | 9,789 (42.2%) | -0.03 |
| Midwest; n (%) | 5,614 (18.4%) | 1,127 (11.1%) | 0.21 | 13,822 (35.4%) | 6,022 (46.2%) | -0.22 | 19,436 (27.9%) | 7,149 (30.8%) | -0.06 |
| West; n (%) | 7,090 (23.2%) | 1,685 (16.5%) | 0.17 | 6,317 (16.2%) | 2,009 (15.4%) | 0.02 | 13,407 (19.2%) | 3,694 (15.9%) | 0.09 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 183 (0.5%) | 63 (0.5%) | 0.00 | 183 (0.3%) | 63 (0.3%) | 0.00 |
| CV Covariates | · | | | | | | | | |
| Ischemic heart disease; n (%) | 10,190 (33.3%) | 3,232 (31.7%) | 0.03 | 12,833 (32.8%) | 4,242 (32.6%) | 0.00 | 23,023 (33.1%) | 7,474 (32.2%) | 0.02 |
| Acute MI; n (%) | 763 (2.5%) | 184 (1.8%) | 0.05 | 1,178 (3.0%) | 250 (1.9%) | 0.07 | 1941 (2.8%) | 434 (1.9%) | 0.06 |
| ACS/unstable angina; n (%) | 909 (3.0%) | 250 (2.5%) | 0.03 | 1,582 (4.0%) | 492 (3.8%) | 0.01 | 2491 (3.6%) | 742 (3.2%) | 0.02 |
| Old MI; n (%) | 1,782 (5.8%) | 413 (4.1%) | 0.08 | 1,022 (2.6%) | 224 (1.7%) | 0.06 | 2804 (4.0%) | 637 (2.7%) | 0.07 |
| Stable angina; n (%) | 2,184 (7.1%) | 708 (7.0%) | 0.00 | 2,274 (5.8%) | 767 (5.9%) | 0.00 | 4,458 (6.4%) | 1,475 (6.4%) | 0.00 |
| Coronary atherosclerosis and other forms | 9,135 (29.9%) | 2,910 (28.6%) | 0.03 | 11,369 (29.1%) | 3,744 (28.7%) | 0.01 | 20,504 (29.4%) | 6,654 (28.7%) | 0.02 |
| of chronic ischemic heart disease; n (%) | | | | | | | | | |
| Other atherosclerosis with ICD10; n (%) | 467 (1.5%) | 160 (1.6%) | -0.01 | 715 (1.8%) | 280 (2.1%) | -0.02 | 1182 (1.7%) | 440 (1.9%) | -0.02 |
| Previous cardiac procedure (CABG or PTCA | 460 (1.5%) | 96 (0.9%) | 0.06 | 1,009 (2.6%) | 226 (1.7%) | 0.06 | 1469 (2.1%) | 322 (1.4%) | 0.05 |
| or Stent); n (%) | () | | | | | | | | |
| History of CABG or PTCA; n (%) | 2,592 (8.5%) | 722 (7.1%) | 0.05 | 1,420 (3.6%) | 385 (3.0%) | 0.03 | 4,012 (5.8%) | 1,107 (4.8%) | 0.04 |
| Any stroke; n (%) | 4,439 (14.5%) | 1,358 (13.3%) | 0.03 | 5,684 (14.5%) | 1,919 (14.7%) | -0.01 | 10,123 (14.5%) | 3,277 (14.1%) | 0.01 |
| Ischemic stroke (w and w/o mention of | 4,398 (14.4%) | 1,341 (13.2%) | 0.03 | 5,629 (14.4%) | 1,907 (14.6%) | -0.01 | 10,027 (14.4%) | 3,248 (14.0%) | 0.01 |
| cerebral infarction); n (%) | 140 (0 EW) | 42 (0.4%) | 0.01 | 170 (0 EW) | 41 (0.3%) | 0.03 | 319 (0.5%) | 93 (0.49/) | 0.01 |
| Hemorrhagic stroke; n (%) | 140 (0.5%) | | | 179 (0.5%) | 41 (0.3%) | 0.03 | | 83 (0.4%) | |
| TIA; n (%) Other cerebrovascular disease; n (%) | 1,169 (3.8%) | 332 (3.3%) | 0.03<br>0.04 | 1,563 (4.0%) | 501 (3.8%) | 0.01 | 2732 (3.9%)<br>2206 (3.2%) | 833 (3.6%) | 0.02 |
| Late effects of cerebrovascular disease; n | 1,160 (3.8%) | 315 (3.1%) | 0.04 | 1,046 (2.7%) | 320 (2.5%)<br>226 (1.7%) | 0.01 | 1945 (2.8%) | 635 (2.7%)<br>489 (2.1%) | 0.05 |
| (%) | 1,068 (3.5%) | 263 (2.6%) | 0.05 | 877 (2.2%) | 220 (1.770) | 0.04 | 1343 (2.070) | +07 (2.170) | 0.05 |
| (70)<br>Cerebrovascular procedure; n (%) | 86 (0.3%) | 25 (0.2%) | 0.02 | 198 (0.5%) | 65 (0.5%) | 0.00 | 284 (0.4%) | 90 (0.4%) | 0.00 |
| Heart failure (CHF); n (%) | 3,690 (12.1%) | 1,106 (10.9%) | 0.02 | 3,739 (9.6%) | 1,133 (8.7%) | 0.03 | 7,429 (10.7%) | 2,239 (9.6%) | 0.04 |
| Peripheral Vascular Disease (PVD) or PVD | 3,739 (12.2%) | 1,216 (11.9%) | 0.04 | 3,346 (8.6%) | 1,050 (8.1%) | 0.03 | 7,085 (10.2%) | 2,266 (9.8%) | 0.04 |
| Surgery; n (%) | 3,733 (12.270) | 1,210 (11.5%) | 0.01 | 3,340 (0.070) | 1,030 (0.170) | 0.02 | 7,003 (10.270) | 2,200 (3.070) | 0.01 |
| Atrial fibrillation; n (%) | 3,724 (12,2%) | 962 (9.4%) | 0.09 | 4.091 (10.5%) | 1,194 (9.2%) | 0.04 | 7.815 (11.2%) | 2,156 (9.3%) | 0.06 |
| Other cardiac dysrhythmia; n (%) | 4,907 (16.1%) | 1,375 (13.5%) | 0.07 | 4,006 (10.2%) | 1,242 (9.5%) | 0.04 | 8,913 (12.8%) | 2,617 (11.3%) | 0.05 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Cardiac conduction disorders; n (%) | 1,293 (4.2%) | 360 (3.5%) | 0.04 | 1,066 (2.7%) | 277 (2.1%) | 0.04 | 2359 (3.4%) | 637 (2.7%) | 0.04 | ı |
|---|---|---|---|---|---|---|---|---|---|---|
| Other CVD; n (%) | 3,202 (10.5%) | 960 (9.4%) | 0.04 | 5,927 (15.2%) | 1,945 (14.9%) | 0.01 | 9,129 (13.1%) | 2,905 (12.5%) | 0.02 | ı |
| Diabetes-related complications | | | | | | | | | | ı |
| Diabetic retinopathy; n (%) | 2,260 (7.4%) | 857 (8.4%) | -0.04 | 2,067 (5.3%) | 731 (5.6%) | -0.01 | 4,327 (6.2%) | 1,588 (6.8%) | -0.02 | ı |
| Diabetes with other ophthalmic | 300 (1.0%) | 119 (1.2%) | -0.02 | 1,353 (3.5%) | 470 (3.6%) | -0.01 | 1,653 (2.4%) | 0,589 (2.5%) | -0.01 | ı |
| manifestations; n (%) | | | | | | | | | | ı |
| Retinal detachment, vitreous hemorrhage,<br>vitrectomy; n (%) | 179 (0.6%) | 65 (0.6%) | 0.00 | 199 (0.5%) | 72 (0.6%) | -0.01 | 378 (0.5%) | 137 (0.6%) | -0.01 | ı |
| Retinal laser coagulation therapy; n (%) | 218 (0.7%) | 96 (0.9%) | -0.02 | 396 (1.0%) | 167 (1.3%) | -0.03 | 614 (0.9%) | 263 (1.1%) | -0.02 | ı |
| Occurrence of Diabetic Neuropathy; n (%) | 5,375 (17.6%) | 1,768 (17.4%) | 0.01 | 3,080 (7.9%) | 976 (7.5%) | 0.02 | 8,455 (12.1%) | 2,744 (11.8%) | 0.01 | ı |
| occurrence of Diabetic riculopatiny , in (19) | 3,373 (27.070) | 2,700 (27.170) | 0.01 | 3,000 (7.570) | 570 (7.570) | 0.02 | 0,133 (12.170) | 2,7 11 (22.070) | 0.01 | ı |
| Occurrence of diabetic nephropathy with ICD10; n (%) | 4,097 (13.4%) | 1,564 (15.4%) | -0.06 | 1,963 (5.0%) | 683 (5.2%) | -0.01 | 6,060 (8.7%) | 2,247 (9.7%) | -0.03 | l |
| Hypoglycemia; n (%) | 403 (1.3%) | 133 (1.3%) | 0.00 | 1,016 (2.6%) | 279 (2.1%) | 0.03 | 1,419 (2.0%) | 0,412 (1.8%) | 0.01 | ı |
| Hyperglycemia; n (%) | 1,356 (4.4%) | 438 (4.3%) | 0.00 | 547 (1.4%) | 156 (1.2%) | 0.02 | 1,903 (2.7%) | 0,594 (2.6%) | 0.01 | ı |
| Disorders of fluid electrolyte and acid-base | 3,686 (12.1%) | 1,034 (10.2%) | 0.06 | 2,829 (7.2%) | 798 (6.1%) | 0.04 | 6,515 (9.4%) | 1,832 (7.9%) | 0.05 | ı |
| balance; n (%) | | | | | | | | | | 1 |
| Diabetic ketoacidosis; n (%) | 84 (0.3%) | 18 (0.2%) | 0.02 | 89 (0.2%) | 26 (0.2%) | 0.00 | 173 (0.2%) | 44 (0.2%) | 0.00 | ı |
| Hyperosmolar hyperglycemic nonketotic | 92 (0.3%) | 24 (0.2%) | 0.02 | 54 (0.1%) | 20 (0.2%) | -0.03 | 146 (0.2%) | 44 (0.2%) | 0.00 | ı |
| syndrome (HONK); n (%) | | - | | - | | | - | | | 1 |
| Diabetes with peripheral circulatory disorders with ICD-10; n (%) | 2,053 (6.7%) | 663 (6.5%) | 0.01 | 946 (2.4%) | 310 (2.4%) | 0.00 | 2,999 (4.3%) | 0,973 (4.2%) | 0.00 | l |
| Diabetic Foot; n (%) | 1,262 (4.1%) | 265 (2.6%) | 0.08 | 1,603 (4.1%) | 415 (3.2%) | 0.05 | 2865 (4.1%) | 680 (2.9%) | 0.07 | ı |
| Gangrene; n (%) | 124 (0.4%) | 16 (0.2%) | 0.04 | 111 (0.3%) | 17 (0.1%) | 0.04 | 235 (0.3%) | 33 (0.1%) | 0.04 | ı |
| Lower extremity amputation; n (%) | 312 (1.0%) | 51 (0.5%) | 0.06 | 188 (0.5%) | 33 (0.3%) | 0.03 | 500 (0.7%) | 84 (0.4%) | 0.04 | ı |
| Osteomyelitis; n (%) | 269 (0.9%) | 43 (0.4%) | 0.06 | 323 (0.8%) | 58 (0.4%) | 0.05 | 592 (0.8%) | 101 (0.4%) | 0.05 | ı |
| Skin infections; n (%) | 2,288 (7.5%) | 562 (5.5%) | 0.08 | 2,693 (6.9%) | 807 (6.2%) | 0.03 | 4,981 (7.2%) | 1,369 (5.9%) | 0.05 | ı |
| Erectile dysfunction; n (%) | 634 (2.1%) | 258 (2.5%) | -0.03 | 401 (1.0%) | 152 (1.2%) | -0.02 | 1,035 (1.5%) | 0,410 (1.8%) | -0.02 | ı |
| Diabetes with unspecified complication; n (%) | 1,118 (3.7%) | 382 (3.7%) | 0.00 | 751 (1.9%) | 233 (1.8%) | 0.01 | 1,869 (2.7%) | 0,615 (2.6%) | 0.01 | l |
| Diabetes mellitus without mention of complications; n (%) | 13,676 (44.8%) | 5,038 (49.5%) | -0.09 | 15,361 (39.3%) | 5,474 (42.0%) | -0.05 | 29,037 (41.7%) | 10,512 (45.3%) | -0.07 | l |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 27,536 (90.1%) | 9,735 (95.6%) | -0.21 | 26,419 (67.6%) | 9,876 (75.8%) | -0.18 | 53,955 (77.5%) | 19,611 (84.5%) | -0.18 | l |
| Hyperlipidemia ; n (%) | 19,134 (62.6%) | 6,815 (66.9%) | -0.09 | 14,108 (36.1%) | 4,802 (36.9%) | -0.02 | 33,242 (47.7%) | 11,617 (50.0%) | -0.05 | 1 |
| Edema; n (%) | 5,202 (17.0%) | 1,351 (13.3%) | 0.10 | 4,091 (10.5%) | 1,103 (8.5%) | 0.07 | 9,293 (13.3%) | 2,454 (10.6%) | 0.08 | 1 |
| Renal Dysfunction (non-diabetic); n (%) | 8,373 (27.4%) | 3,032 (29.8%) | -0.05 | 5,789 (14.8%) | 2,163 (16.6%) | -0.05 | 14,162 (20.3%) | 5,195 (22.4%) | -0.05 | ı |
| Occurrence of acute renal disease; n (%) | 1,458 (4.8%) | 374 (3.7%) | 0.05 | 1,270 (3.2%) | 341 (2.6%) | 0.04 | 2728 (3.9%) | 715 (3.1%) | 0.04 | ı |
| Occurrence of chronic renal insufficiency;<br>n (%) | 6,787 (22.2%) | 2,512 (24.7%) | -0.06 | 4,135 (10.6%) | 1,631 (12.5%) | -0.06 | 10,922 (15.7%) | 4,143 (17.8%) | -0.06 | |
| Chronic kidney disease ; n (%) | 6,566 (21.5%) | 2,430 (23.9%) | -0.06 | 3,774 (9.7%) | 1,505 (11.6%) | -0.06 | 10,340 (14.8%) | 3,935 (16.9%) | -0.06 | 1 |
| CKD Stage 3-4; n (%) | 4,689 (15.3%) | 1,764 (17.3%) | -0.05 | 2,418 (6.2%) | 1,002 (7.7%) | -0.06 | 7,107 (10.2%) | 2,766 (11.9%) | -0.05 | ı |
| Occurrence of hypertensive nephropathy; | 3,581 (11.7%) | 1,352 (13.3%) | -0.05 | 1,611 (4.1%) | 643 (4.9%) | -0.04 | 5192 (7.5%) | 1995 (8.6%) | -0.04 | l |
| n (%) | 2 220 /7 20/ | 063 /0 EW1 | 0.04 | 1 979 /4 99/ | 734/E CW1 | -0.04 | 4 107 /E 094) | 1 507 (5 004) | 0.04 | ı |
| Occurrence of miscellaneous renal<br>insufficiency; n (%) | 2,228 (7.3%) | 863 (8.5%) | -0.04 | 1,879 (4.8%) | 734 (5.6%) | -0.04 | 4,107 (5.9%) | 1,597 (6.9%) | -0.04 | ı |
| ** ** | 6,579 (21.5%) | 2,433 (23.9%) | -0.06 | 7,118 (18.2%) | 2,588 (19.9%) | -0.04 | 13,697 (19.7%) | 5,021 (21.6%) | -0.05 | ı |
| Glaucoma or cataracts ; n (%)<br>Cellulitis or abscess of toe; n (%) | 735 (2.4%) | 2,433 (23.9%)<br>133 (1.3%) | 0.08 | 7,118 (18.2%)<br>449 (1.1%) | 2,588 (19.9%)<br>124 (1.0%) | 0.04 | | 257 (1.1%) | 0.05 | 1 |
| | | | | | | | 1184 (1.7%) | | | ı |
| Foot ulcer; n (%) | 1,250 (4.1%) | 268 (2.6%) | 0.08 | 1,648 (4.2%) | 426 (3.3%) | 0.05 | 2898 (4.2%) | 694 (3.0%) | 0.06 | ı |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Bladder stones; n (%) | 44 (0.1%) | 11 (0.1%) | 0.00 | 37 (0.1%) | 9 (0.1%) | 0.00 | 81 (0.1%) | 20 (0.1%) | 0.00 | ı |
|---|---|---|---|---|---|---|---|---|---|---|
| Kidney stones; n (%) | 718 (2.3%) | 224 (2.2%) | 0.01 | 650 (1.7%) | 221 (1.7%) | 0.00 | 1,368 (2.0%) | 0,445 (1.9%) | 0.01 | ı |
| Urinary tract infections (UTIs); n (%) | 3,654 (12.0%) | 1,123 (11.0%) | 0.03 | 3,124 (8.0%) | 873 (6.7%) | 0.05 | 6,778 (9.7%) | 1,996 (8.6%) | 0.04 | ı |
| Dipstick urinalysis; n (%) | 10,731 (35.1%) | 4,047 (39.7%) | -0.10 | 9,218 (23.6%) | 3,227 (24.8%) | -0.03 | 19,949 (28.6%) | 7,274 (31.3%) | -0.06 | ı |
| Non-dipstick urinalysis; n (%) | 7,758 (25.4%) | 3,078 (30.2%) | -0.11 | 4,754 (12.2%) | 1,632 (12.5%) | -0.01 | 12,512 (18.0%) | 4,710 (20.3%) | -0.06 | ı |
| Urine function test; n (%) | 871 (2.9%) | 324 (3.2%) | -0.02 | 1,148 (2.9%) | 406 (3.1%) | -0.01 | 2,019 (2.9%) | 0,730 (3.1%) | -0.01 | ı |
| Cytology; n (%) | 433 (1.4%) | 134 (1.3%) | 0.01 | 709 (1.8%) | 191 (1.5%) | 0.02 | 1142 (1.6%) | 325 (1.4%) | 0.02 | ı |
| Cystos; n (%) | 576 (1.9%) | 184 (1.8%) | 0.01 | 936 (2.4%) | 270 (2.1%) | 0.02 | 1512 (2.2%) | 454 (2.0%) | 0.01 | ı |
| Other Covariates | | | | | | | | | | ı |
| Liver disease; n (%) | 1,031 (3.4%) | 336 (3.3%) | 0.01 | 378 (1.0%) | 92 (0.7%) | 0.03 | 1,409 (2.0%) | 0,428 (1.8%) | 0.01 | ı |
| Osteoarthritis; n (%) | 6,896 (22.6%) | 2,198 (21.6%) | 0.02 | 5,701 (14.6%) | 1,857 (14.3%) | 0.01 | 12,597 (18.1%) | 4,055 (17.5%) | 0.02 | ı |
| Other arthritis, arthropathies and | 13,531 (44.3%) | 4,208 (41.3%) | 0.06 | 13,759 (35.2%) | 4,457 (34.2%) | 0.02 | 27,290 (39.2%) | 8,665 (37.3%) | 0.04 | ı |
| musculoskeletal pain; n (%) | | | | | | | | | | ı |
| Dorsopathies; n (%) | 8,371 (27.4%) | 2,675 (26.3%) | 0.02 | 7,865 (20.1%) | 2,610 (20.0%) | 0.00 | 16,236 (23.3%) | 5,285 (22.8%) | 0.01 | ı |
| Fractures; n (%) | 1,359 (4.4%) | 308 (3.0%) | 0.07 | 1,687 (4.3%) | 466 (3.6%) | 0.04 | 3,046 (4.4%) | 0,774 (3.3%) | 0.06 | ı |
| Falls; n (%) | 1,768 (5.8%) | 379 (3.7%) | 0.10 | 341 (0.9%) | 82 (0.6%) | 0.03 | 2109 (3.0%) | 461 (2.0%) | 0.06 | ı |
| Osteoporosis; n (%) | 2,841 (9.3%) | 963 (9.5%) | -0.01 | 3,457 (8.8%) | 1,173 (9.0%) | -0.01 | 6,298 (9.0%) | 2,136 (9.2%) | -0.01 | ı |
| Hyperthyroidism; n (%) | 228 (0.7%) | 85 (0.8%) | -0.01 | 169 (0.4%) | 66 (0.5%) | -0.01 | 397 (0.6%) | 151 (0.7%) | -0.01 | ı |
| Hypothyroidism; n (%) | 5,256 (17.2%) | 1,768 (17.4%) | -0.01 | 3,261 (8.3%) | 1,046 (8.0%) | 0.01 | 8,517 (12.2%) | 2,814 (12.1%) | 0.00 | ı |
| Other disorders of thyroid gland; n (%) | 1,209 (4.0%) | 470 (4.6%) | -0.03 | 870 (2.2%) | 348 (2.7%) | -0.03 | 2,079 (3.0%) | 0,818 (3.5%) | -0.03 | ı |
| Depression; n (%) | 2,922 (9.6%) | 699 (6.9%) | 0.10 | 2,210 (5.7%) | 572 (4.4%) | 0.06 | 5,132 (7.4%) | 1,271 (5.5%) | 0.08 | ı |
| Anxiety; n (%) | 3,025 (9.9%) | 832 (8.2%) | 0.06 | 1,405 (3.6%) | 376 (2.9%) | 0.04 | 4,430 (6.4%) | 1,208 (5.2%) | 0.05 | ı |
| SleepDisorder; n (%) | 1,872 (6.1%) | 667 (6.5%) | -0.02 | 3,366 (8.6%) | 1,261 (9.7%) | -0.04 | 5,238 (7.5%) | 1,928 (8.3%) | -0.03 | ı |
| Dementia; n (%) | 1,867 (6.1%) | 443 (4.3%) | 0.08 | 1,454 (3.7%) | 350 (2.7%) | 0.06 | 3321 (4.8%) | 793 (3.4%) | 0.07 | ı |
| Delirium; n (%) | 615 (2.0%) | 125 (1.2%) | 0.06 | 559 (1.4%) | 109 (0.8%) | 0.06 | 1174 (1.7%) | 234 (1.0%) | 0.06 | ı |
| Psychosis; n (%) | 427 (1.4%) | 89 (0.9%) | 0.05 | 433 (1.1%) | 86 (0.7%) | 0.04 | 860 (1.2%) | 175 (0.8%) | 0.04 | ı |
| Obesity; n (%) | 5,506 (18.0%) | 2,014 (19.8%) | -0.05 | 2,043 (5.2%) | 630 (4.8%) | 0.02 | 7,549 (10.8%) | 2,644 (11.4%) | -0.02 | ı |
| Overweight; n (%) | 1,809 (5.9%) | 697 (6.8%) | -0.04 | 203 (0.5%) | 92 (0.7%) | -0.03 | 2,012 (2.9%) | 0,789 (3.4%) | -0.03 | ı |
| Smoking; n (%) | 4,399 (14.4%) | 1,083 (10.6%) | 0.12 | 1,540 (3.9%) | 385 (3.0%) | 0.05 | 5,939 (8.5%) | 1,468 (6.3%) | 0.08 | ı |
| Alcohol abuse or dependence; n (%) | 386 (1.3%) | 66 (0.6%) | 0.07 | 180 (0.5%) | 36 (0.3%) | 0.03 | 566 (0.8%) | 102 (0.4%) | 0.05 | ı |
| Drug abuse or dependence; n (%) | 678 (2.2%) | 169 (1.7%) | 0.04 | 191 (0.5%) | 38 (0.3%) | 0.03 | 869 (1.2%) | 207 (0.9%) | 0.03 | ı |
| COPD; n (%) | 4,635 (15.2%) | 1,287 (12.6%) | 0.08 | 4,322 (11.1%) | 1,224 (9.4%) | 0.06 | 8,957 (12.9%) | 2,511 (10.8%) | 0.07 | ı |
| Asthma; n (%) | 2,178 (7.1%) | 749 (7.4%) | -0.01 | 1,919 (4.9%) | 687 (5.3%) | -0.02 | 4,097 (5.9%) | 1,436 (6.2%) | -0.01 | ı |
| Obstructive sleep apnea; n (%) | 2,861 (9.4%) | 1,030 (10.1%) | -0.02 | 2,220 (5.7%) | 842 (6.5%) | -0.03 | 5,081 (7.3%) | 1,872 (8.1%) | -0.03 | ı |
| Pneumonia; n (%) | 1,212 (4.0%) | 284 (2.8%) | 0.07 | 1,603 (4.1%) | 401 (3.1%) | 0.05 | 2,815 (4.0%) | 0,685 (3.0%) | 0.05 | ı |
| Imaging, n (%) | 61 (0.2%) | 13 (0.1%) | 0.03 | 7,118 (18.2%) | 17 (0.1%) | 0.66 | 122 (0.2%) | 30 (0.1%) | 0.03 | ı |
| Other Medications | | | | | | | | | | ı |
| Use of ACE inhibitors; n (%) | 12,465 (40.8%) | 1,969 (19.3%) | 0.48 | 16,962 (43.4%) | 3,692 (28.3%) | 0.32 | 29,427 (42.3%) | 5,661 (24.4%) | 0.39 | ı |
| Use of ARBs; n (%) | 9,547 (31.2%) | 10,187 (100.0%) | -2.10 | 11,259 (28.8%) | 13,030 (100.0%) | -2.22 | 20,806 (29.9%) | 23,217 (100.0%) | -2.17 | ı |
| Use of Loop Diuretics - ; n (%) | 12,256 (40.1%) | 3,193 (31.3%) | 0.18 | 18,355 (47.0%) | 4,966 (38.1%) | 0.18 | 30,611 (44.0%) | 8,159 (35.1%) | 0.18 | ı |
| Use of other diuretics-; n (%) | 1,140 (3.7%) | 452 (4.4%) | -0.04 | 1,556 (4.0%) | 607 (4.7%) | -0.03 | 2,696 (3.9%) | 1,059 (4.6%) | -0.03 | ı |
| Use of nitrates-; n (%) | 2,848 (9.3%) | 918 (9.0%) | 0.01 | 5,406 (13.8%) | 1,759 (13.5%) | 0.01 | 8,254 (11.9%) | 2,677 (11.5%) | 0.01 | 1 |
| Use of other hypertension drugs; n (%) | 3,696 (12.1%) | 1,741 (17.1%) | -0.14 | 4,858 (12.4%) | 2,168 (16.6%) | -0.12 | 8,554 (12.3%) | 3,909 (16.8%) | -0.13 | ı |
| Use of digoxin-; n (%) | 691 (2.3%) | 211 (2.1%) | 0.01 | 1,888 (4.8%) | 610 (4.7%) | 0.00 | 2579 (3.7%) | 821 (3.5%) | 0.01 | L |
| Use of Anti-arrhythmics; n (%) | 835 (2.7%) | 250 (2.5%) | 0.01 | 1,365 (3.5%) | 447 (3.4%) | 0.01 | 2200 (3.2%) | 697 (3.0%) | 0.01 | ı |
| Use of COPD/asthma meds-; n (%) | 5,867 (19.2%) | 2,136 (21.0%) | -0.04 | 7,725 (19.8%) | 2,699 (20.7%) | -0.02 | 13,592 (19.5%) | 4,835 (20.8%) | -0.03 | ı |
| Use of statins; n (%) | 19,124 (62.6%) | 6,880 (67.5%) | -0.10 | 23,989 (61.4%) | 8,315 (63.8%) | -0.05 | 43,113 (61.9%) | 15,195 (65.4%) | -0.07 | ı |
| Use of other lipid-lowering drugs; n (%) | 2,786 (9.1%) | 1,173 (11.5%) | -0.08 | 5,338 (13.7%) | 2,163 (16.6%) | -0.08 | 8,124 (11.7%) | 3,336 (14.4%) | -0.08 | ı |
| • | - | | | | | | | | | ~ |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Use of oral anticoagulants (Dabigatran, | 3,235 (10.6%) | 837 (8.2%) | 0.08 | 4,611 (11.8%) | 1,329 (10.2%) | 0.05 | 7,846 (11.3%) | 2,166 (9.3%) | 0.07 |
|---|---|---|---|---|---|---|---|---|---|
| Rivaroxaban, Apixaban, Warfarin); n (%) | | | | | | | | | |
| Use of heparin and other low-molecular | 191 (0.6%) | 42 (0.4%) | 0.03 | 25 (0.1%) | 2 (0.0%) | 0.04 | 216 (0.3%) | 44 (0.2%) | 0.02 |
| weight heparins; n (%) | | () | | | () | | | | |
| Use of NSAIDs; n (%) | 4,843 (15.8%) | 1,727 (17.0%) | -0.03 | 5,571 (14.3%) | 1,988 (15.3%) | -0.03 | 10,414 (15.0%) | 3,715 (16.0%) | -0.03 |
| Use of oral corticosteroids; n (%) | 6,288 (20.6%) | 2,072 (20.3%) | 0.01 | 7,586 (19.4%) | 2,503 (19.2%) | 0.01 | 13,874 (19.9%) | 4,575 (19.7%) | 0.01 |
| Use of bisphosphonate (); n (%) | 1,423 (4.7%) | 481 (4.7%) | 0.00 | 2,556 (6.5%) | 889 (6.8%) | -0.01 | 3979 (5.7%) | 1370 (5.9%) | -0.01 |
| Use of opioids- ; n (%) | 8,944 (29.3%) | 2,651 (26.0%) | 0.07 | 13,182 (33.7%) | 4,088 (31.4%) | 0.05 | 22,126 (31.8%) | 6,739 (29.0%) | 0.06 |
| Use of antidepressants; n (%) | 8,217 (26.9%) | 2,446 (24.0%) | 0.07 | 9,879 (25.3%) | 3,102 (23.8%) | 0.03 | 18,096 (26.0%) | 5,548 (23.9%) | 0.05 |
| Use of antipsychotics; n (%) | 847 (2.8%) | 202 (2.0%) | 0.05 | 984 (2.5%) | 257 (2.0%) | 0.03 | 1,831 (2.6%) | 0,459 (2.0%) | 0.04 |
| Use of anticonvulsants; n (%) | 5,915 (19.4%) | 1,744 (17.1%) | 0.06 | 5,485 (14.0%) | 1,691 (13.0%) | 0.03 | 11,400 (16.4%) | 3,435 (14.8%) | 0.04 |
| Use of lithium- ; n (%) | 52 (0.2%) | 5 (0.0%) | 0.06 | 43 (0.1%) | 10 (0.1%) | 0.00 | 95 (0.1%) | 15 (0.1%) | 0.00 |
| Use of Benzos- ; n (%) | 3,815 (12.5%) | 1,286 (12.6%) | 0.00 | 6,652 (17.0%) | 2,308 (17.7%) | -0.02 | 10,467 (15.0%) | 3,594 (15.5%) | -0.01 |
| Use of anxiolytics/hypnotics-; n (%) | 2,091 (6.8%) | 718 (7.0%) | -0.01 | 3,734 (9.6%) | 1,335 (10.2%) | -0.02 | 5,825 (8.4%) | 2,053 (8.8%) | -0.01 |
| Use of dementia meds-; n (%) | 994 (3.3%) | 321 (3.2%) | 0.01 | 1,308 (3.3%) | 392 (3.0%) | 0.02 | 2302 (3.3%) | 713 (3.1%) | 0.01 |
| Use of antiparkinsonian meds-; n (%) | 1,061 (3.5%) | 271 (2.7%) | 0.05 | 1,276 (3.3%) | 402 (3.1%) | 0.01 | 2,337 (3.4%) | 0,673 (2.9%) | 0.03 |
| Entresto (sacubitril/valsartan); n (%) | 62 (0.2%) | 2 (0.0%) | 0.06 | 4 (0.0%) | 0 (0.0%) | #DIV/0! | 66 (0.1%) | 2 (0.0%) | 0.04 |
| Labs | | | | | | | 0 | 0 | |
| Lab values- HbA1c (%); n (%) | 6,661 (21.8%) | 2,606 (25.6%) | -0.09 | 566 (1.4%) | 139 (1.1%) | 0.03 | 7,227 (10.4%) | 2,745 (11.8%) | -0.04 |
| Lab values- HbA1c (%) (within 3 months) ; n<br>(%) | 4,616 (15.1%) | 1,790 (17.6%) | -0.07 | 407 (1.0%) | 91 (0.7%) | 0.03 | 5,023 (7.2%) | 1,881 (8.1%) | -0.03 |
| Lab values- HbA1c (%) (within 6 months); n | 6,661 (21.8%) | 2,606 (25.6%) | -0.09 | 566 (1.4%) | 139 (1.1%) | 0.03 | 7,227 (10.4%) | 2,745 (11.8%) | -0.04 |
| (%) | | | | | | | | | |
| Lab values- BNP; n (%) | 398 (1.3%) | 111 (1.1%) | 0.02 | 15 (0.0%) | 5 (0.0%) | #DIV/0! | 413 (0.6%) | 116 (0.5%) | 0.01 |
| Lab values- BNP (within 3 months); n (%) | 315 (1.0%) | 75 (0.7%) | 0.03 | 12 (0.0%) | 1 (0.0%) | #DIV/0! | 327 (0.5%) | 76 (0.3%) | 0.03 |
| Lab values- BNP (within 6 months); n (%) | 398 (1.3%) | 111 (1.1%) | 0.02 | 15 (0.0%) | 5 (0.0%) | #DIV/0! | 413 (0.6%) | 116 (0.5%) | 0.01 |
| Lab values- BUN (mg/dl); n (%) | 9,795 (32.1%) | 3,628 (35.6%) | -0.07 | 415 (1.1%) | 169 (1.3%) | -0.02 | 10,210 (14.7%) | 3,797 (16.4%) | -0.05 |
| Lab values-BUN (mg/dl) (within 3 months); | 7,233 (23.7%) | 2,633 (25.8%) | -0.05 | 300 (0.8%) | 120 (0.9%) | -0.01 | 7,533 (10.8%) | 2,753 (11.9%) | -0.03 |
| n (%) | | | | | | | | | |
| Lab values-BUN (mg/dl) (within 6 months); | 9,795 (32.1%) | 3,628 (35.6%) | -0.07 | 415 (1.1%) | 169 (1.3%) | -0.02 | 10,210 (14.7%) | 3,797 (16.4%) | -0.05 |
| n (%) | | | | | | | | | |
| Lab values- Creatinine (mg/dl); n (%) | 10,174 (33.3%) | 3,760 (36.9%) | -0.08 | 439 (1.1%) | 182 (1.4%) | -0.03 | 10,613 (15.2%) | 3,942 (17.0%) | -0.05 |
| Lab values- Creatinine (mg/dl) (within 3<br>months) ; n (%) | 7,531 (24.6%) | 2,722 (26.7%) | -0.05 | 322 (0.8%) | 130 (1.0%) | -0.02 | 7,853 (11.3%) | 2,852 (12.3%) | -0.03 |
| Lab values- Creatinine (mg/dl) (within 6<br>months) ; n (%) | 10,174 (33.3%) | 3,760 (36.9%) | -0.08 | 439 (1.1%) | 182 (1.4%) | -0.03 | 10,613 (15.2%) | 3,942 (17.0%) | -0.05 |
| Lab values- HDL level (mg/dl); n (%) | 7,125 (23.3%) | 2,794 (27.4%) | -0.09 | 485 (1.2%) | 126 (1.0%) | 0.02 | 7,610 (10.9%) | 2,920 (12.6%) | -0.05 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 4,750 (15.5%) | 1,815 (17.8%) | -0.06 | 326 (0.8%) | 77 (0.6%) | 0.02 | 5,076 (7.3%) | 1,892 (8.1%) | -0.03 |
| Lab values-HDL level (mg/dl) (within 6 months); n (%) | 7,125 (23.3%) | 2,794 (27.4%) | -0.09 | 485 (1.2%) | 126 (1.0%) | 0.02 | 7,610 (10.9%) | 2,920 (12.6%) | -0.05 |
| Lab values-LDL level (mg/dl); n (%) | 7,501 (24.5%) | 2,923 (28.7%) | -0.10 | 541 (1.4%) | 132 (1.0%) | 0.04 | 8,042 (11.5%) | 3,055 (13.2%) | -0.05 |
| Lab values-LDL level (mg/dl) (within 3 months); n (%) | 4,974 (16.3%) | 1,901 (18.7%) | -0.06 | 369 (0.9%) | 79 (0.6%) | 0.03 | 5,343 (7.7%) | 1,980 (8.5%) | -0.03 |
| | 7 504 (04 50) | 2,923 (28.7%) | -0.10 | 541 (1.4%) | 132 (1.0%) | 0.04 | 8,042 (11.5%) | 3,055 (13.2%) | -0.05 |
| Lab values- LDL level (mg/dl) (within 6<br>months) ; n (%) | 7,501 (24.5%) | 2,525 (20.770) | | | | | | | |
| | 7,501 (24.5%)<br>86 (0.3%) | 19 (0.2%) | 0.02 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 86 (0.1%) | 19 (0.1%) | 0.00 |
| months); n (%) | | | 0.02<br>0.03 | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | #DIV/0!<br>#DIV/0! | 86 (0.1%)<br>71 (0.1%) | 19 (0.1%)<br>9 (0.0%) | 0.00<br>0.04 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Lab values-NT-proBNP (within 6 months);<br>n (%) | 86 (0.3%) | 19 (0.2%) | 0.02 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 86 (0.1%) | 19 (0.1%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values-Total cholesterol (mg/dl); n (%) | 7,363 (24.1%) | 2,895 (28.4%) | -0.10 | 499 (1.3%) | 134 (1.0%) | 0.03 | 7,862 (11.3%) | 3,029 (13.0%) | -0.05 |
| Lab values-Total cholesterol (mg/dl)<br>(within 3 months); n (%) | 4,900 (16.0%) | 1,885 (18.5%) | -0.07 | 340 (0.9%) | 81 (0.6%) | 0.03 | 5,240 (7.5%) | 1,966 (8.5%) | -0.04 |
| Lab values-Total cholesterol (mg/dl)<br>(within 6 months); n (%) | 7,363 (24.1%) | 2,895 (28.4%) | -0.10 | 499 (1.3%) | 134 (1.0%) | 0.03 | 7,862 (11.3%) | 3,029 (13.0%) | -0.05 |
| Lab values-Triglyceride level (mg/dl); n (%) | 7,248 (23.7%) | 2,860 (28.1%) | -0.10 | 487 (1.2%) | 132 (1.0%) | 0.02 | 7,735 (11.1%) | 2,992 (12.9%) | -0.06 |
| Lab values-Triglyceride level (mg/dl)<br>(within 3 months); n (%) | 4,827 (15.8%) | 1,864 (18.3%) | -0.07 | 325 (0.8%) | 79 (0.6%) | 0.02 | 5,152 (7.4%) | 1,943 (8.4%) | -0.04 |
| Lab values-Triglyceride level (mg/dl)<br>(within 6 months); n (%) | 7,248 (23.7%) | 2,860 (28.1%) | -0.10 | 487 (1.2%) | 132 (1.0%) | 0.02 | 7,735 (11.1%) | 2,992 (12.9%) | -0.06 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 6,534 | 2,568 | | 419 | 139 | | 0 | 0 | |
| mean (sd) | 6.97 (1.55) | 6.86 (1.37) | 0.08 | 7.42 (1.63) | 7.36 (1.68) | 0.04 | 7.22 (1.60) | 7.14 (1.55) | 0.05 |
| median [IQR] | 6.60 [5.90, 7.60] | 6.50 [5.90, 7.47] | 0.07 | 7.00 [6.40, 8.00] | 6.90 [6.20, 8.00] | 0.06 | 6.82 (1.60) | 6.72 (1.55) | 0.06 |
| Missing; n (%) | 24,024 (78.6%) | 7,619 (74.8%) | 0.09 | 38,671 (98.9%) | 12,891 (98.9%) | 0.00 | 62,695 (90.0%) | 20,510 (88.3%) | 0.05 |
| Lab result number- BNP mean | 398 | 111 | | 15 | 5 | | 0 | 0 | |
| mean (sd) | 185.26 (253.16) | 135.34 (198.32) | 0.22 | 208.58 (332.19) | 52.80 (38.49) | 0.66 | 198.35 (300.09) | 89.02 (134.49) | 0.47 |
| median [IQR] | 94.00 [41.27, 239.25] | 67.60 [30.80, 147.97] | 0.12 | 56.00 [21.00,<br>260.00] | 60.00 [17.50, 84.50] | -0.02 | 72.67 (300.09) | 63.33 (134.49) | 0.04 |
| Missing; n (%) | 30,160 (98.7%) | 10,076 (98.9%) | -0.02 | 39,075 (100.0%) | 13,025 (100.0%) | #DIV/0! | 69,235 (99.4%) | 23,101 (99.5%) | -0.01 |
| Lab result number- BUN (mg/dl) mean | 9,795 | 3,628 | | 415 | 169 | | 0 | 0 | |
| mean (sd) | 20.16 (10.19) | -71.24 (5,534.18) | 0.02 | 20.45 (9.55) | 21.61 (12.44) | -0.10 | 20.32 (9.84) | -19.13 (3665.83) | 0.02 |
| median [IQR] | 18.00 [14.00, 23.50] | 18.00 [14.00, 24.00] | 0.00 | 19.00 [14.00, 24.00] | 19.00 [14.00, 24.00] | 0.00 | 18.56 (9.84) | 18.56 (3665.83) | 0.00 |
| Missing; n (%) | 20,763 (67.9%) | 6,559 (64.4%) | 0.07 | 38,675 (98.9%) | 12,861 (98.7%) | 0.02 | 59,438 (85.3%) | 19,420 (83.6%) | 0.05 |
| Lab result number- Creatinine (mg/dl)<br>mean (only 0.1 to 15 included) | 9,940 | 3,657 | | 414 | 169 | | 0 | 0 | |
| mean (sd) | 1.14 (0.64) | 1.16 (0.63) | -0.03 | 1.15 (0.61) | 1.25 (1.04) | -0.12 | 1.15 (0.62) | 1.21 (0.88) | -0.08 |
| median [IQR] | 1.00 [0.82, 1.26] | 1.02 [0.84, 1.30] | -0.03 | 1.00 [0.83, 1.29] | 1.00 [0.83, 1.27] | 0.00 | 1.00 (0.62) | 1.01 (0.88) | -0.01 |
| Missing; n (%) | 20,618 (67.5%) | 6,530 (64.1%) | 0.07 | 38,676 (98.9%) | 12,861 (98.7%) | 0.02 | 59,294 (85.1%) | 19,391 (83.5%) | 0.04 |
| Lab result number- HDL level (mg/dl) mean<br>(only =<5000 included) | 7,125 | 2,794 | | 485 | 126 | | 0 | 0 | |
| mean (sd) | 50.65 (17.42) | 50.72 (17.23) | 0.00 | 47.35 (14.16) | 46.74 (13.38) | 0.04 | 48.80 (15.67) | 48.49 (15.19) | 0.02 |
| median [IQR] | 49.00 [40.00, 60.00] | 49.00 [40.00, 60.00] | 0.00 | 45.00 [37.00, 55.00] | 44.25 [36.75, 54.25] | 0.05 | 46.75 (15.67) | 46.33 (15.19) | 0.03 |
| Missing; n (%) | 23,433 (76.7%) | 7,393 (72.6%) | 0.09 | 38,605 (98.8%) | 12,904 (99.0%) | -0.02 | 62,038 (89.1%) | 20,297 (87.4%) | 0.05 |
| Lab result number-LDL level (mg/dl) mean (only =<5000 included) | 7,380 | 2,882 | | 494 | 129 | | 0 | 0 | |
| mean (sd) | -182.77 (16,462.54) | -1,476.42 (38,379.52) | 0.04 | 86.53 (36.62) | 85.79 (40.20) | 0.02 | -31.63 (10904.49) | -599.67 (25422.45) | 0.03 |
| median [IQR] | 84.00 [64.00, 110.50] | 82.00 [63.00, 105.00] | 0.00 | 82.00 [65.00,<br>107.00] | 80.50 [58.33,<br>112.00] | 0.04 | 82.88 (10904.49) | 81.16 (25422.45) | 0.00 |
| Missing; n (%) | 23,178 (75.8%) | 7,305 (71.7%) | 0.09 | 38,596 (98.7%) | 12,901 (99.0%) | -0.03 | 61,774 (88.7%) | 20,206 (87.0%) | 0.05 |
| Lab result number-Total cholesterol | 7,362 | 2,891 | | 499 | 134 | | 0 | 0 | |
| (mg/dl) mean (only =<5000 included) | | _, | | | | | - | _ | ı |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| mean (sd) | 167.59 (49.65) | 165.07 (48.23) | 0.05 | 168.89 (43.43) | 171.93 (55.24) | -0.06 | 168.32 (46.26) | 168.92 (52.28) | -0.01 |
|---|---|---|---|---|---|---|---|---|---|
| | 165.00 [139.00, | 163.00 [139.00, | 0.05 | 162.00 [140.00, | 162.00 [140.25, | 0.00 | 163.32 (46.26) | 162.44 (52.28) | 0.02 |
| median [IQR] | 195.00] | 191.00] | 0.04 | 192.00] | 195.75] | 0.00 | 163.32 (46.26) | 162.44 (52.28) | 0.02 |
| Missing; n (%) | 23,196 (75.9%) | 7,296 (71.6%) | 0.10 | 38,591 (98.7%) | 12,896 (99.0%) | -0.03 | 61,787 (88.7%) | 20,192 (87.0%) | 0.05 |
| Lab result number-Triglyceride level | 7,248 | 2,860 | | 487 | 132 | | 0 | 0 | - 1 |
| (mg/dl) mean (only =<5000 included) | | | | | | | | | - 1 |
| mean (sd) | 142.17 (87.70) | 141.97 (89.94) | 0.00 | 165.50 (146.50) | 195.76 (371.54) | -0.11 | 155.26 (124.18) | 172.16 (284.65) | -0.08 |
| median [IQR] | 122.00 [88.00,<br>172.00] | 122.00 [88.00,<br>170.00] | 0.00 | 137.00 [97.00,<br>190.00] | 140.50 [95.25,<br>205.00] | -0.01 | 130.42 (124.18) | 132.38 (284.65) | -0.01 |
| Missing; n (%) | 23,310 (76.3%) | 7,327 (71.9%) | 0.10 | 38,603 (98.8%) | 12,898 (99.0%) | -0.02 | 61,913 (88.9%) | 20,225 (87.1%) | 0.06 |
| Lab result number- Hemoglobin mean | 7,384 | 2,785 | | 291 | 118 | | 0 | 0 | |
| (only >0 included) | ,, | - | | | | | | | - 1 |
| mean (sd) | 12.98 (1.77) | 12.93 (1.70) | 0.03 | 12.88 (1.90) | 84,758.66<br>(920,573.33) | -0.13 | 12.92 (1.84) | 47574.50<br>(689651.34) | -0.10 |
| median [IQR] | 13.00 [11.90, 14.17] | 12.93 [11.80, 14.05] | 0.04 | 12.95 [11.90, 14.10] | 13.10 [11.90, 14.35] | 0.00 | 12.97 (1.84) | 13.03 (689651.34) | 0.00 |
| Missing; n (%) | 23,174 (75.8%) | 7,402 (72.7%) | 0.07 | 38,799 (99.3%) | 12,912 (99.1%) | 0.02 | 61,973 (89.0%) | 20,314 (87.5%) | 0.05 |
| Lab result number- Serum sodium mean<br>(only >90 and <190 included) | 9,645 | 3,620 | | 373 | 154 | | 0 | 0 | |
| mean (sd) | 140.31 (3.03) | 140.44 (2.92) | -0.04 | 139.48 (2.89) | 139.94 (2.67) | -0.17 | 139.84 (2.95) | 140.16 (2.78) | -0.11 |
| median [IQR] | 140.67 [139.00,<br>142.00] | 141.00 [139.00,<br>142.00] | -0.11 | 140.00 [138.00,<br>141.00] | 140.00 [138.38,<br>142.00] | 0.00 | 140.29 (2.95) | 140.44 (2.78) | -0.05 |
| Missing; n (%) | 20,913 (68.4%) | 6,567 (64.5%) | 0.08 | 38,717 (99.0%) | 12,876 (98.8%) | 0.02 | 59,630 (85.6%) | 19,443 (83.7%) | 0.05 |
| Lab result number- Albumin mean (only >0 | 8,891 | 3,390 | | 335 | 148 | | 0 | 0 | |
| and <=10 included) | · · | • | | | | | | | |
| mean (sd) | 4.15 (0.37) | 4.20 (0.36) | -0.14 | 4.07 (0.48) | 4.13 (0.38) | -0.14 | 4.11 (0.44) | 4.16 (0.37) | -0.12 |
| median [IQR] | 4.20 [3.95, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.10 [3.90, 4.40] | 4.18 [4.00, 4.37] | -0.18 | 4.14 (0.44) | 4.19 (0.37) | -0.12 |
| Missing; n (%) | 21,667 (70.9%) | 6,797 (66.7%) | 0.09 | 38,755 (99.1%) | 12,882 (98.9%) | 0.02 | 60,422 (86.8%) | 19,679 (84.8%) | 0.06 |
| Lab result number- Glucose (fasting or | 9,589 | 3,608 | | 356 | 153 | | 0 | 0 | - 1 |
| random) mean (only 10-1000 included) | | | | | | | | | |
| mean (sd) | 125.63 (52.72) | 123.59 (46.97) | 0.04 | 144.13 (58.68) | 144.99 (59.74) | -0.01 | 136.01 (56.14) | 135.60 (54.51) | 0.01 |
| median [IQR] | 108.50 [94.00,<br>141.00] | 109.00 [95.00,<br>138.00] | -0.01 | 129.25 [103.44,<br>166.88] | 133.00 [106.50,<br>165.25] | -0.06 | 120.15 (56.14) | 122.47 (54.51) | -0.04 |
| Missing; n (%) | 20,969 (68.6%) | 6,579 (64.6%) | 0.08 | 38,734 (99.1%) | 12,877 (98.8%) | 0.03 | 59,703 (85.7%) | 19,456 (83.8%) | 0.05 |
| Lab result number- Potassium mean (only<br>1-7 included) | 9,892 | 3,674 | | 420 | 169 | | 0 | 0 | |
| mean (sd) | 4.42 (0.48) | 4.37 (0.48) | 0.10 | 4.31 (0.51) | 4.28 (0.48) | 0.06 | 4.36 (0.50) | 4.32 (0.48) | 0.08 |
| median [IQR] | 4.40 [4.10, 4.70] | 4.35 [4.07, 4.65] | 0.10 | 4.30 [4.00, 4.60] | 4.30 [4.00, 4.60] | 0.00 | 4.34 (0.50) | 4.32 (0.48) | 0.04 |
| Missing; n (%) | 20,666 (67.6%) | 6,513 (63.9%) | 0.08 | 38,670 (98.9%) | 12,861 (98.7%) | 0.02 | 59,336 (85.2%) | 19,374 (83.4%) | 0.05 |
| Comorbidity Scores | , ,, | , ,, | | , | , | | , | , ,, | |
| CCI (180 days)-ICD9 and ICD10 | | | | | | | | | |
| mean (sd) | 3.10 (2.10) | 3.04 (2.00) | 0.03 | 2.11 (1.80) | 2.08 (1.69) | 0.02 | 2.54 (1.94) | 2.50 (1.83) | 0.02 |
| median [IQR] | 3.00 [1.00, 4.00] | 3.00 [1.00, 4.00] | 0.00 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 2.44 (1.94) | 2.44 (1.83) | 0.00 |
| Frailty Score (mean): Empirical Version 365 days, | , | ,, | | ,, | | | | | |
| mean (sd) | 0.19 (0.06) | 0.18 (0.06) | 0.17 | 0.17 (0.06) | 0.17 (0.05) | 0.00 | 0.18 (0.06) | 0.17 (0.05) | 0.18 |
| mean (so)<br>median [IQR] | 0.18 [0.14, 0.22] | 0.18 (0.06) | 0.17 | 0.16 [0.13, 0.20] | 0.16 [0.14, 0.19] | 0.00 | 0.17 (0.06) | 0.17 (0.05) | 0.18 |
| median [iQK] Healthcare Utilization | 0.10 [0.14, 0.22] | 0.17 [0.14, 0.21] | 0.17 | 0.10 [0.13, 0.20] | 0.10 [0.14, 0.15] | 0.00 | 0.17 (0.06) | 0.10 (0.05) | 0.10 |
| Any hospitalization; n (%) | 4,339 (14.2%) | 939 (9.2%) | 0.16 | 7,950 (20.3%) | 1,950 (15.0%) | 0.14 | 12,289 (17.6%) | 2,889 (12.4%) | 0.15 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| la | 2.455/40.49() | 730 (7 00/) | 0.11 | E 0E4 (4E 00/) | 4 545 (44 00/) | 0.10 | 0.447/43.40/ | 2 204 (0 00) | 0.10 | |
|---|---|---|---|---|---|---|---|---|---|---|
| Any hospitalization during prior 31-180 | 3,166 (10.4%) | 738 (7.2%) | 0.11 | 5,951 (15.2%) | 1,546 (11.9%) | 0.10 | 9,117 (13.1%) | 2,284 (9.8%) | 0.10 | ı |
| days; n (%) | 0.040 (5.70/) | ner (n ray) | 0.07 | 0.400/5.50/ | 007 (5 00/) | | 4.030 (5.40) | 4 750 /7 50/ | 0.05 | ı |
| Endocrinologist Visit; n (%) | 2,048 (6.7%) | 865 (8.5%) | -0.07 | 2,190 (5.6%) | 897 (6.9%) | -0.05 | 4,238 (6.1%) | 1,762 (7.6%) | -0.06 | ı |
| Endocrinologist Visit (30 days prior); n (%) | 730 (2.4%) | 285 (2.8%) | -0.03 | 784 (2.0%) | 346 (2.7%) | -0.05 | 1,514 (2.2%) | 0,631 (2.7%) | -0.03 | ı |
| Endocrinologist Visit (31 to 180 days | 1,793 (5.9%) | 782 (7.7%) | -0.07 | 1,959 (5.0%) | 801 (6.1%) | -0.05 | 3,752 (5.4%) | 1,583 (6.8%) | -0.06 | ı |
| prior); n (%) | | | | | | | | | | ı |
| Internal medicine/family medicine visits; n<br>(%) | 26,121 (85.5%) | 8,580 (84.2%) | 0.04 | 30,158 (77.2%) | 10,465 (80.3%) | -0.08 | 56,279 (80.8%) | 19,045 (82.0%) | -0.03 | l |
| Internal medicine/family medicine visits | 16,528 (54.1%) | 5,661 (55.6%) | -0.03 | 18,789 (48.1%) | 6,950 (53.3%) | -0.10 | 35,317 (50.7%) | 12,611 (54.3%) | -0.07 | ı |
| (30 days prior); n (%) | 10,528 (54.1%) | 3,001 (33.0%) | -0.03 | 10,705 (40.1%) | 0,550 (55.5%) | 4.10 | 33,317 (30.770) | 12,011 (54.5%) | -0.07 | ı |
| Internal medicine/family medicine visits | 24,292 (79.5%) | 7,939 (77.9%) | 0.04 | 27,875 (71.3%) | 9,655 (74.1%) | -0.06 | 52,167 (74.9%) | 17,594 (75.8%) | -0.02 | ı |
| (31 to 180 days prior); n (%) | | | | | | | | | | ı |
| Cardiologist visit; n (%) | 12,308 (40.3%) | 4,133 (40.6%) | -0.01 | 13,821 (35.4%) | 5,000 (38.4%) | -0.06 | 26,129 (37.5%) | 9,133 (39.3%) | -0.04 | ı |
| Number of Cardiologist visits (30 days prior); n (%) | 5,503 (18.0%) | 1,788 (17.6%) | 0.01 | 6,180 (15.8%) | 2,310 (17.7%) | -0.05 | 11,683 (16.8%) | 4,098 (17.7%) | -0.02 | l |
| Number of Cardiologist visits (31 to 180 | 10,090 (33.0%) | 3,429 (33.7%) | -0.01 | 11,449 (29.3%) | 4,188 (32.1%) | -0.06 | 21,539 (30.9%) | 7,617 (32.8%) | -0.04 | ı |
| days prior); n (%) | 10,050 (55.0%) | 3,423 (33.770) | 0.01 | 11,445 (25.5%) | 4,100 (32.1%) | 0.00 | 21,333 (30.370) | 7,017 (52.070) | 0.01 | ı |
| Electrocardiogram ; n (%) | 12,530 (41.0%) | 3,952 (38.8%) | 0.04 | 16,188 (41.4%) | 5,594 (42.9%) | -0.03 | 28,718 (41.2%) | 9,546 (41.1%) | 0.00 | ı |
| Use of glucose test strips; n (%) | 699 (2.3%) | 271 (2.7%) | -0.03 | 692 (1.8%) | 278 (2.1%) | -0.02 | 1,391 (2.0%) | 0,549 (2.4%) | -0.03 | ı |
| Dialysis; n (%) | 100 (0.3%) | 33 (0.3%) | 0.00 | 179 (0.5%) | 58 (0.4%) | 0.01 | 279 (0.4%) | 91 (0.4%) | 0.00 | ı |
| number of different/distinct medication | 100 (0.3%) | 33 (0.5%) | 0.00 | 175 (0.5%) | 36 (0.470) | 0.01 | 275 (0.4%) | 31 (0.4%) | 0.00 | ı |
| prescriptions | | | | | | | | | | ı |
| mean (sd) | 10.39 (5.17) | 11.81 (5.25) | -0.27 | 10.90 (5.24) | 11.95 (5.36) | -0.20 | 10.68 (5.21) | 11.89 (5.31) | -0.23 | ı |
| | 10.00 [7.00, 13.00] | 11.00 [8.00, 15.00] | -0.19 | 10.00 [7.00, 14.00] | 11.00 [8.00, 15.00] | -0.19 | 10.00 (5.21) | 11.00 (5.31) | -0.19 | ı |
| median [IQR] | 10.00 [7.00, 15.00] | 11.00 [0.00, 15.00] | -0.15 | 10.00 [7.00, 14.00] | 11.00 [0.00, 15.00] | -0.15 | 10.00 (5.21) | 11.00 (5.51) | -0.15 | ı |
| Number of Hospitalizations | | | | | | | | | | ı |
| mean (sd) | 0.18 (0.49) | 0.11 (0.38) | 0.16 | 0.24 (0.52) | 0.17 (0.44) | 0.15 | 0.21 (0.51) | 0.14 (0.41) | 0.15 | ı |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.51) | 0.00 (0.41) | 0.00 | ı |
| Number of hospital days | , , , , , , | | | | . , , | | | , | | ı |
| mean (sd) | 1.08 (4.26) | 0.57 (2.56) | 0.15 | 1.41 (4.54) | 0.94 (3.46) | 0.12 | 1.27 (4.42) | 0.78 (3.10) | 0.13 | ı |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (4.42) | 0.00 (3.10) | 0.00 | ı |
| Number of Emergency Department (ED) | | | | | | | (/ | | | ı |
| visits | | | | | | | | | | ı |
| mean (sd) | 0.58 (1.36) | 0.44 (1.38) | 0.10 | 0.26 (1.50) | 0.14 (1.12) | 0.09 | 0.40 (1.44) | 0.27 (1.24) | 0.10 | ı |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.44) | 0.00 (1.24) | 0.00 | ı |
| Number of Office visits | | | | | | | | | | ı |
| mean (sd) | 5.90 (4.60) | 6.12 (4.55) | -0.05 | 6.16 (5.13) | 6.65 (5.08) | -0.10 | 6.05 (4.90) | 6.42 (4.85) | -0.08 | ı |
| median [IQR] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 0.00 | 5.00 [3.00, 8.00] | 6.00 [3.00, 9.00] | -0.20 | 5.00 (4.90) | 5.56 (4.85) | -0.11 | ۱ |
| Number of Endocrinologist visits | | | | | | | | | | ı |
| mean (sd) | 0.30 (1.74) | 0.40 (2.08) | -0.05 | 0.27 (1.69) | 0.34 (1.91) | -0.04 | 0.41 (1.55) | 0.38 (1.70) | 0.02 | ۱ |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.55) | 0.00 (1.70) | 0.00 | 1 |
| Number of internal medicine/family | | | | | | | | | | ı |
| medicine visits | | | | | | | | | | 1 |
| mean (sd) | 11.25 (15.95) | 10.71 (15.22) | 0.03 | 7.00 (11.52) | 7.51 (11.09) | -0.05 | 8.86 (13.64) | 8.91 (13.06) | 0.00 | 1 |
| median [IQR] | 6.00 [2.00, 14.00] | 6.00 [2.00, 13.00] | 0.00 | 4.00 [1.00, 9.00] | 4.00 [1.00, 10.00] | 0.00 | 4.88 (13.64) | 4.88 (13.06) | 0.00 | ı |
| Number of Cardiologist visits | | | | | | | | | | ۱ |
| mean (sd) | 2.14 (4.97) | 2.09 (4.45) | 0.01 | 1.96 (4.61) | 2.13 (4.53) | -0.04 | 2.04 (4.77) | 2.11 (4.50) | -0.02 | ı |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 (4.77) | 0.00 (4.50) | 0.00 | ı |
| F-3-1 | | | | | | | | | | |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Number electrocardiograms received | 1 | | | | | | | | - 1 |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 0.87 (1.60) | 0.75 (1.41) | 0.08 | 0.81 (1.43) | 0.79 (1.32) | 0.01 | 0.84 (1.51) | 0.77 (1.36) | 0.05 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.51) | 0.00 (1.36) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 0.69 (0.88) | 0.82 (0.93) | -0.14 | 0.34 (0.69) | 0.35 (0.72) | -0.01 | 0.49 (0.78) | 0.56 (0.82) | -0.09 |
| median [IQR] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | -1.10 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.78) | 0.44 (0.82) | -0.55 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.34 (2.36) | 0.35 (2.08) | 0.00 | 0.23 (0.92) | 0.23 (1.41) | 0.00 | 0.28 (1.71) | 0.28 (1.74) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.71) | 0.00 (1.74) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 0.75 (0.93) | 0.86 (0.96) | -0.12 | 0.43 (0.89) | 0.43 (0.90) | 0.00 | 0.57 (0.91) | 0.62 (0.93) | -0.05 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.44 (0.91) | 0.44 (0.93) | 0.00 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.10 (0.48) | 0.08 (0.40) | 0.05 | 0.14 (0.67) | 0.06 (0.38) | 0.15 | 0.12 (0.59) | 0.07 (0.39) | 0.10 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.59) | 0.00 (0.39) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.07 (0.54) | 0.06 (0.50) | 0.02 | 0.09 (0.59) | 0.05 (0.44) | 0.08 | 0.08 (0.57) | 0.05 (0.47) | 0.06 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.57) | 0.00 (0.47) | 0.00 |
| Number of tests for microal buminuria | | | | | | | | | |
| mean (sd) | 0.48 (1.07) | 0.60 (1.16) | -0.11 | 0.18 (0.64) | 0.20 (0.67) | -0.03 | 0.31 (0.86) | 0.38 (0.92) | -0.08 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.86) | 0.00 (0.92) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at | | | | | | | | | |
| the 3rd digit level | | | | 4 1 | | | | | |
| mean (sd) | 8.34 (9.97) | 7.64 (8.67) | 0.07 | 1.77 (4.44) | 1.41 (3.76) | 0.09 | 4.65 (7.39) | 4.14 (6.40) | 0.07 |
| median [IQR] | 6.00 [0.00, 12.00] | 5.00 [0.00, 12.00] | 0.11 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 2.63 (7.39) | 2.19 (6.40) | 0.06 |
| For PS | 4 222 (4 221) | 200 (2 00) | | 4 () | () | | | (n) | |
| Hemorrhagic stroke+Other | 1,288 (4.2%) | 362 (3.6%) | 0.03 | 1,308 (3.3%) | 392 (3.0%) | 0.02 | 2596 (3.7%) | 754 (3.2%) | 0.03 |
| cerebrovascular disease+Cerebrovascular<br>procedure (for PS); n (%) | | | | | | | | | |
| Occurrence of creatinine tests ordered (for PS); n (%) | 1,980 (6.5%) | 542 (5.3%) | 0.05 | 2,949 (7.5%) | 562 (4.3%) | 0.14 | 4,929 (7.1%) | 1,104 (4.8%) | 0.10 |
| Occurrence of BUN tests ordered (for PS); n<br>(%) | 1,146 (3.8%) | 339 (3.3%) | 0.03 | 1,852 (4.7%) | 411 (3.2%) | 80.0 | 2,998 (4.3%) | 0,750 (3.2%) | 0.06 |
| Occurrence of chronic renal insufficiency<br>w/o CKD (for PS); n (%) | 2,436 (8.0%) | 840 (8.2%) | -0.01 | 1,704 (4.4%) | 660 (5.1%) | -0.03 | 4,140 (5.9%) | 1,500 (6.5%) | -0.02 |
| Chronic kidney disease Stage 1-2 (for PS); n<br>(%) | 1,248 (4.1%) | 514 (5.0%) | -0.04 | 443 (1.1%) | 214 (1.6%) | -0.04 | 1691 (2.4%) | 728 (3.1%) | -0.04 |
| Chronic kidney disease Stage 3-6 (for PS); n<br>(%) | 4,943 (16.2%) | 1,843 (18.1%) | -0.05 | 2,782 (7.1%) | 1,114 (8.5%) | -0.05 | 7,725 (11.1%) | 2,957 (12.7%) | -0.05 |
| Bladder stones+Kidney stones (for PS); n<br>(%) | 738 (2.4%) | 228 (2.2%) | 0.01 | 670 (1.7%) | 227 (1.7%) | 0.00 | 1,408 (2.0%) | 0,455 (2.0%) | 0.00 |
| Diabetes with peripheral circulatory disorders+Gangrene+Osteomyelitis(for PS) with ICD10; n (%) | 2,248 (7.4%) | 700 (6.9%) | 0.02 | 1,251 (3.2%) | 367 (2.8%) | 0.02 | 3,499 (5.0%) | 1,067 (4.6%) | 0.02 |
| Alcohol abuse or dependence+Drug abuse<br>or dependence (for PS); n (%) | 1,014 (3.3%) | 227 (2.2%) | 0.07 | 340 (0.9%) | 71 (0.5%) | 0.05 | 1354 (1.9%) | 298 (1.3%) | 0.05 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Diabetes with other ophthalmic manifestations+Retinal detachment, vitreous hemorrhage, vitrectomy+Retinal | 645 (2.1%) | 257 (2.5%) | -0.03 | 1,738 (4.4%) | 616 (4.7%) | -0.01 | 2,383 (3.4%) | 0,873 (3.8%) | -0.02 |
|---|---|---|---|---|---|---|---|---|---|
| laser coagulation therapy (for PS); n (%) Other atherosclerosis+Cardiac conduction disorders+Other CVD (for PS); n (%) | 4,574 (15.0%) | 1,386 (13.6%) | 0.04 | 7,157 (18.3%) | 2,324 (17.8%) | 0.01 | 11,731 (16.8%) | 3,710 (16.0%) | 0.02 |
| Previous cardiac procedure (CABG or PTCA<br>or Stent) + History of CABG or PTCA (for PS)<br>; n (%) | 2,735 (9.0%) | 748 (7.3%) | 0.06 | 2,029 (5.2%) | 527 (4.0%) | 0.06 | 4,764 (6.8%) | 1,275 (5.5%) | 0.05 |
| Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland (for PS); n (%) | 6,115 (20.0%) | 2,123 (20.8%) | -0.02 | 3,989 (10.2%) | 1,338 (10.3%) | 0.00 | 10,104 (14.5%) | 3,461 (14.9%) | -0.01 |
| Delirium + Psychosis (for PS); n (%) | 943 (3.1%) | 200 (2.0%) | 0.07 | 893 (2.3%) | 178 (1.4%) | 0.07 | 1836 (2.6%) | 378 (1.6%) | 0.07 |
| Any use of Meglitinides (for PS); n (%) | 169 (0.6%) | 89 (0.9%) | -0.03 | 426 (1.1%) | 202 (1.6%) | -0.04 | 595 (0.9%) | 291 (1.3%) | -0.04 |
| Any use of AGIs (for PS); n (%) | 56 (0.2%) | 19 (0.2%) | 0.00 | 87 (0.2%) | 43 (0.3%) | -0.02 | 11,731 (16.8%) | 3,710 (16.0%) | 0.02 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 4,953 (16.2%) | 1,845 (18.1%) | -0.05 | 2,814 (7.2%) | 1,121 (8.6%) | -0.05 | 7,767 (11.2%) | 2,966 (12.8%) | -0.05 |
| Use of thiazide; n (%) | 11,780 (38.5%) | 3,002 (29.5%) | 0.19 | 14,978 (38.3%) | 3,878 (29.8%) | 0.18 | 36,428 (52.3%) | 12,835 (55.3%) | -0.06 |
| Use of beta blockers; n (%) | 15,394 (50.4%) | 5,625 (55.2%) | -0.10 | 21,034 (53.8%) | 7,210 (55.3%) | -0.03 | 41,604 (59.7%) | 16,258 (70.0%) | -0.22 |
| Use of calcium channel blockers; n (%) | 18,948 (62.0%) | 7,400 (72.6%) | -0.23 | 22,656 (58.0%) | 8,858 (68.0%) | -0.21 | 24,505 (35.2%) | 9,196 (39.6%) | -0.09 |
| All antidiabetic medications except<br>Insulin; n (%) | 11,225 (36.7%) | 4,342 (42.6%) | -0.12 | 13,280 (34.0%) | 4,854 (37.3%) | -0.07 | 26,758 (38.4%) | 6,880 (29.6%) | 0.19 |
| DM Medications - Insulin ; n (%) | 4,651 (15.2%) | 1,738 (17.1%) | -0.05 | 6,406 (16.4%) | 2,156 (16.5%) | 0.00 | 11,057 (15.9%) | 3,894 (16.8%) | -0.02 |
| Use of Low Intensity Statins; n (%) | 9,976 (32.6%) | 3,348 (32.9%) | -0.01 | 13,646 (34.9%) | 4,367 (33.5%) | 0.03 | 23622 (33.9%) | 7,715 (33.2%) | 0.01 |
| Use of High Intensity Statins; n (%) | 9,219 (30.2%) | 3,433 (33.7%) | -0.08 | 9,307 (23.8%) | 3,330 (25.6%) | -0.04 | 18526 (26.6%) | 6,763 (29.1%) | -0.06 |
| Malignant hypertension; n (%) | 1,065 (3.5%) | 303 (3.0%) | 0.03 | 16,602 (42.5%) | 5,939 (45.6%) | -0.06 | 17667 (25.4%) | 6,242 (26.9%) | -0.03 |
| Cardiovascular stress test; n (%) | 52 (0.2%) | 25 (0.2%) | 0.00 | 180 (0.5%) | 59 (0.5%) | 0.00 | 0,232 (0.3%) | 84 (0.4%) | -0.02 |
| Echocardiogram; n (%) | 4,440 (14.5%) | 1,292 (12.7%) | 0.05 | 8,540 (21.8%) | 2,793 (21.4%) | 0.01 | 12,980 (18.6%) | 4085 (17.6%) | 0.03 |
| Number of BNP tests | | | | | | | | | |
| mean (sd) | 0.08 (0.35) | 0.06 (0.32) | 0.06 | 0.05 (0.29) | 0.04 (0.26) | 0.04 | 0.06 (0.32) | 0.05 (0.29) | 0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.32) | 0.00 (0.29) | 0.00 |
| Number of Cardiac biomarkers tests | | | | | | | | | |
| (tropnin, CK-MBs, Myoglobin, CPK) | | | | | | | | | |
| mean (sd) | 0.24 (0.97) | 0.20 (0.85) | 0.04 | 0.21 (0.97) | 0.19 (0.94) | 0.02 | 0.22 (0.97) | 0.19 (0.90) | 0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.97) | 0.00 (0.90) | 0.00 |
| Number of Ambulatory Blood pressure<br>monitoring tests | | | | | | | | | |
| mean (sd) | 0.00 (0.04) | 0.00 (0.05) | 0.00 | 0.00 (0.06) | 0.00 (0.08) | 0.00 | 0.00 (0.05) | 0.00 (0.07) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.05) | 0.00 (0.07) | 0.00 |
| N of days on antihypertensive medications | | | | | | | | | ı |
| during baseline | | | | | | | | | |
| mean (sd) | 133.67 (59.83) | 157.56 (44.97) | -0.45 | 136.86 (58.07) | 151.84 (48.50) | -0.28 | 135.46 (58.85) | 154.35 (46.98) | -0.35 |
| median [IQR] | 168.00 [89.00,<br>181.00] | 180.00 [160.00,<br>181.00] | -0.23 | 169.00 [103.00,<br>181.00] | 177.00 [147.00,<br>181.00] | -0.15 | 168.56 (58.85) | 178.32 (46.98) | -0.18 |
| N of days in database anytime prior | | | | | | | | | |
| mean (sd) | 1,995.86 (1,453.10) | 2,000.22 (1,451.36) | 0.00 | 1,703.15 (1,098.06) | 1,702.21 (1,073.87) | 0.00 | 1831.58 (1266.15) | 1832.97 (1253.58) | 0.00 |
| median [IQR] | 1,624.00 [863.00,<br>2,765.00] | 1,603.00 [870.00,<br>2,760.00] | 0.01 | 1,489.50 [821.00,<br>2,387.00] | 1,512.00 [823.00,<br>2,435.00] | -0.02 | 1548.51 (1266.15) | 1551.93 (1253.58) | 0.00 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Mean Copay for per prescription cost | 1 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (charges in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 27.35 (36.41) | 27.57 (33.60) | -0.01 | 24.94 (27.07) | 25.76 (27.05) | -0.03 | 26.00 (31.51) | 26.55 (30.10) | -0.02 |
| median [IQR] | 18.09 [7.38, 34.53] | 18.83 [7.21, 35.75] | -0.02 | 19.14 [8.16, 34.09] | 20.24 [8.02, 35.24] | -0.04 | 18.68 (31.51) | 19.62 (30.10) | -0.03 |
| | 20.05 [7.50, 51.55] | 20.03 [7.22, 33.73] | 0.02 | 25.21 [0.20, 5 1.05] | 20.21 [0.02, 33.21] | 0.01 | 20.00 (32.32) | 15.02 (50.10) | 0.03 |
| Missing; n (%) | 35 (0.1%) | 125 (1.2%) | -0.14 | 25 (0.1%) | 155 (1.2%) | -0.14 | 0,060 (0.1%) | 280 (1.2%) | -0.14 |
| Colonos; n (%) | 1,397 (4.6%) | 507 (5.0%) | -0.02 | 2,205 (5.6%) | 691 (5.3%) | 0.01 | 3,602 (5.2%) | 1198 (5.2%) | 0.00 |
| Fecal occult blood (FOB) test; n (%) | 1,279 (4.2%) | 451 (4.4%) | -0.01 | 1,375 (3.5%) | 423 (3.2%) | 0.02 | 2,654 (3.8%) | 874 (3.8%) | 0.00 |
| Flu vaccine; n (%) | 5,716 (18.7%) | 1,888 (18.5%) | 0.01 | 4,264 (10.9%) | 1,381 (10.6%) | 0.01 | 9,980 (14.3%) | 3269 (14.1%) | 0.01 |
| Mammogram; n (%) | 3,758 (12.3%) | 1,366 (13.4%) | -0.03 | 4,463 (11.4%) | 1,576 (12.1%) | -0.02 | 8,221 (11.8%) | 2942 (12.7%) | -0.03 |
| Pap smear; n (%) | 864 (2.8%) | 337 (3.3%) | -0.03 | 1,502 (3.8%) | 527 (4.0%) | -0.01 | 2,366 (3.4%) | 864 (3.7%) | -0.02 |
| Pneumonia vaccine; n (%) | 5,084 (16.6%) | 1,661 (16.3%) | 0.01 | 1,174 (3.0%) | 369 (2.8%) | 0.01 | 6,258 (9.0%) | 2030 (8.7%) | 0.01 |
| PSA test or Prostate exam for DRE; n (%) | 3,599 (11.8%) | 1,374 (13.5%) | -0.05 | 3,005 (7.7%) | 1,010 (7.8%) | 0.00 | 6,604 (9.5%) | 2384 (10.3%) | -0.03 |
| Bone mineral density; n (%) | 1,387 (4.5%) | 501 (4.9%) | -0.02 | 1,099 (2.8%) | 410 (3.1%) | -0.02 | 2,486 (3.6%) | 911 (3.9%) | -0.02 |
| Use of Sympatomimetic agents; n (%) | 241 (0.8%) | 88 (0.9%) | -0.01 | 690 (1.8%) | 245 (1.9%) | -0.01 | 0,931 (1.3%) | 333 (1.4%) | -0.01 |
| Use of CNS stimulants; n (%) | 175 (0.6%) | 59 (0.6%) | 0.00 | 338 (0.9%) | 116 (0.9%) | 0.00 | 0,513 (0.7%) | 175 (0.8%) | -0.01 |
| Use of estrogens, progestins, androgens; n | 1,157 (3.8%) | 444 (4.4%) | -0.03 | 2,529 (6.5%) | 936 (7.2%) | -0.03 | 3,686 (5.3%) | 1380 (5.9%) | -0.03 |
| (%) | 2,227 (3.2.7) | () | 0.02 | 2,525 (5.515) | 220 (2.4) | | 2,000 (2.2.0) | 2500 (5.570) | 0.02 |
| Use of Angiogenesis inhibitors; n (%) | 17 (0.1%) | 2 (0.0%) | 0.04 | 41 (0.1%) | 7 (0.1%) | 0.00 | 0,058 (0.1%) | 9 (0.0%) | 0.04 |
| Use of Oral Immunosuppressants; n (%) | 106 (0.3%) | 42 (0.4%) | -0.02 | 283 (0.7%) | 68 (0.5%) | 0.03 | 0,389 (0.6%) | 110 (0.5%) | 0.01 |
| Cardiomegaly, LVH, and other cardiopathy | | 1,372 (13.5%) | -0.06 | 3,537 (9.0%) | 1,413 (10.8%) | -0.06 | 7,052 (10.1%) | 2785 (12.0%) | -0.06 |
| due to hypertension; n (%) | 5,515 (11.570) | 1,572 (15.570) | 0.00 | 3,337 (3.070) | 1,115 (10.0%) | 0.00 | 7,032 (20.270) | 2703 (22.0%) | 0.00 |
| Ultrasound; n (%) | 6,328 (20.7%) | 1,957 (19.2%) | 0.04 | 9,576 (24.5%) | 3,275 (25.1%) | -0.01 | 15,904 (22.8%) | 5232 (22.5%) | 0.01 |
| Symptomatic hypotension; n (%) | 808 (2.6%) | 171 (1.7%) | 0.06 | 711 (1.8%) | 155 (1.2%) | 0.05 | 1,519 (2.2%) | 326 (1.4%) | 0.06 |
| Syncopal episodes; n (%) | 913 (3.0%) | 256 (2.5%) | 0.03 | 586 (1.5%) | 211 (1.6%) | -0.01 | 1,499 (2.2%) | 467 (2.0%) | 0.01 |
| N of Generic name drugs only | 515 (5.0%) | 250 (2.5%) | 0.03 | 300 (1.3%) | 211 (1.0%) | 0.01 | 2,455 (2.270) | 407 (2.0%) | 0.01 |
| mean (sd) | 16.93 (12.96) | 19.19 (14.62) | -0.16 | 13.57 (10.14) | 13.52 (10.76) | 0.00 | 15.04 (11.46) | 16.01 (12.60) | -0.08 |
| median [IQR] | 14.00 [8.00, 22.00] | 16.00 [10.00, 25.00] | -0.14 | 11.00 [7.00, 18.00] | 11.00 [6.00, 18.00] | 0.00 | 12.32 (11.46) | 13.19 (12.60) | -0.07 |
| median [lok] | 14.00 [8.00, 22.00] | 16.00 [10.00, 25.00] | -0.14 | 11.00 [7.00, 18.00] | 11.00 [6.00, 16.00] | 0.00 | 12.32 (11.40) | 13.19 (12.60) | -0.07 |
| N of Brand name drugs only | | | | | | | | | |
| mean (sd) | 4.58 (6.39) | 5.69 (7.35) | -0.16 | 7.70 (7.53) | 8.69 (8.23) | -0.13 | 6.33 (7.05) | 7.37 (7.86) | -0.14 |
| median [IQR] | 2.00 [0.00, 6.00] | 3.00 [0.00, 8.00] | -0.15 | 6.00 [2.00, 11.00] | 7.00 [3.00, 12.00] | -0.13 | 4.25 (7.05) | 5.24 (7.86) | -0.13 |
| Number of distinct antihypertensive | | | | | | | | | |
| generic medications (180-1 days before | | | | | | | | | |
| index) | | | | | | | | | |
| mean (sd) | 3.01 (1.39) | 2.98 (1.50) | 0.02 | 3.12 (1.45) | 2.80 (1.57) | 0.21 | 3.07 (1.42) | 2.88 (1.54) | 0.13 |
| median [IQR] | 3.00 [2.00, 4.00] | 3.00 [2.00, 4.00] | 0.00 | 3.00 [2.00, 4.00] | 3.00 [2.00, 4.00] | 0.00 | 3.00 (1.42) | 3.00 (1.54) | 0.00 |
| Number of distinct antihypertensive | | | | | | | | | |
| generic medications on CED | | | | | | | | | |
| mean (sd) | 0.08 (0.34) | 1.40 (0.75) | -2.27 | 0.08 (0.35) | 1.50 (0.83) | -2.23 | 0.08 (0.35) | 1.46 (0.80) | -2.23 |
| median [IQR] | 0.00 [0.00, 0.00] | 1.00 [1.00, 2.00] | -1.72 | 0.00 [0.00, 0.00] | 1.00 [1.00, 2.00] | -1.57 | 0.00 (0.35) | 1.00 (0.80) | -1.62 |
| Hypertensive retinopathy; n (%) | 345 (1.1%) | 182 (1.8%) | -0.06 | 194 (0.5%) | 77 (0.6%) | -0.01 | 0,539 (0.8%) | 259 (1.1%) | -0.03 |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code - CORRECT ONE -<br>TRUVEN | | | | | | | | | |
| | | | | | | | | ***** | |
| Commercial; n (%) | 7,018 (23.0%) | 2,863 (28.1%) | -0.12 | 25,554 (65.4%) | 8,518 (65.4%) | 0.00 | 32,572 (46.8%) | 11381 (49.0%) | 0.00 |
| Medicare Advantage; n (%) | 23,540 (77.0%) | 7,324 (71.9%) | 0.12 | 13,536 (34.6%) | 4,512 (34.6%) | 0.00 | 37,076 (53.2%) | 11836 (51.0%) | 0.00 |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code | l | | | | | | | | |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| COM = COMMERCIAL; n (%) | 7,018 (23.0%) | 2,863 (28.1%) | -0.12 | - | - | #VALUE! | 7,018 (23.0%) | 2,863 (28.1%) | -0.12 |
|---|---|---|---|---|---|---|---|---|---|
| MCR = MEDICARE; n (%) | 23,540 (77.0%) | 7,324 (71.9%) | 0.12 | - | - | #VALUE! | 23,540 (77.0%) | 7,324 (71.9%) | 0.12 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| in 2015); n (%) | | | | | | | | | - 1 |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data | | | | | | | | | |
| Type | | | | | | | | | - 1 |
| 1 - Fee For Service; n (%) | - | - | #VALUE! | 11,302 (28.9%) | 4,122 (31.6%) | -0.06 | 11,302 (28.9%) | 4,122 (31.6%) | -0.06 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 2,234 (5.7%) | 390 (3.0%) | 0.13 | 2,234 (5.7%) | 390 (3.0%) | 0.13 |
| 3 - Medicare; n (%) | - | - | #VALUE! | 21,958 (56.2%) | 8,038 (61.7%) | -0.11 | 21,958 (56.2%) | 8,038 (61.7%) | -0.11 |
| 4 - Medicare Encounter; n (%) | - | - | #VALUE! | 3,596 (9.2%) | 480 (3.7%) | 0.23 | 3,596 (9.2%) | 480 (3.7%) | 0.23 |
| Metropolitan Statistical Area - Urban (any | | | | | | | | | - 1 |
| MSA) vs Rural (non-MSA) | | | | | | | | | - 1 |
| Urban; n (%) | - | - | #VALUE! | 29,715 (76.0%) | 9,885 (75.9%) | 0.00 | 29,715 (76.0%) | 9,885 (75.9%) | 0.00 |
| Rural; n (%) | - | - | #VALUE! | 298 (0.8%) | 75 (0.6%) | 0.02 | 298 (0.8%) | 75 (0.6%) | 0.02 |
| Unknown/Missing; n (%) | - | - | #VALUE! | 9,077 (23.2%) | 3,070 (23.6%) | -0.01 | 9,077 (23.2%) | 3,070 (23.6%) | -0.01 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| | | | F | 'S-matched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Opt | tum | | Truv | en | | POOL | .ED | |
| Variable | Matched Referent | Exposure- | St. Diff. | Matched Referent | Exposure- | St. Diff. | Matched Referent | Exposure- | St. Diff. |
| Number of patients | 8,710 | 8,710 | | 11,314 | 11,314 | | 20,024 | 20,024 | |
| Age | | | | | | | | | |
| mean (sd) | 71.46 (8.13) | 71.49 (8.51) | 0.00 | 70.45 (9.52) | 70.46 (9.87) | 0.00 | 70.89 (8.94) | 70.91 (9.30) | 0.00 |
| median [IQR] | 72.00 [66.00, 77.00] | 72.00 [65.00, 78.00] | 0.00 | 70.00 [62.00, | 70.00 [62.00, | 0.00 | 70.87 (8.94) | 70.87 (9.30) | 0.00 |
| Age categories | | | | | | | | | |
| 18 - 54; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 0,000 (0.0%) | 0,000 (0.0%) | #DIV/0! |
| 55 - 64; n (%) | 1,942 (22.3%) | 2,029 (23.3%) | -0.02 | 4,003 (35.4%) | 4,024 (35.6%) | 0.00 | 5,945 (29.7%) | 6,053 (30.2%) | -0.01 |
| 65 - 74; n (%) | 3,515 (40.4%) | 3,353 (38.5%) | 0.04 | 3,208 (28.4%) | 3,184 (28.1%) | 0.01 | 6,723 (33.6%) | 6,537 (32.6%) | 0.02 |
| >=75; n (%) | 3,253 (37.3%) | 3,328 (38.2%) | -0.02 | 4,103 (36.3%) | 4,106 (36.3%) | 0.00 | 7,356 (36.7%) | 7,434 (37.1%) | -0.01 |
| Gender | | | | | | | | | |
| Males; n (%) | 3,477 (39.9%) | 3,537 (40.6%) | -0.01 | 5,008 (44.3%) | 5,001 (44.2%) | 0.00 | 8,485 (42.4%) | 8,538 (42.6%) | 0.00 |
| Females; n (%) | 5,233 (60.1%) | 5,173 (59.4%) | 0.01 | 6,306 (55.7%) | 6,313 (55.8%) | 0.00 | 11,539 (57.6%) | 11,486 (57.4%) | 0.00 |
| Region | , , , , , , | | | | , , , | | | | |
| _ | | | | | | | | | |
| Northeast; n (%) | 831 (9.5%) | 800 (9.2%) | 0.01 | 1,465 (12.9%) | 1,447 (12.8%) | 0.00 | 2,296 (11.5%) | 2,247 (11.2%) | 0.01 |
| South; n (%) | 5,271 (60.5%) | 5,276 (60.6%) | 0.00 | 3,087 (27.3%) | 3,085 (27.3%) | 0.00 | 8,358 (41.7%) | 8,361 (41.8%) | 0.00 |
| Midwest; n (%) | 1,077 (12.4%) | 1,070 (12.3%) | 0.00 | 5,011 (44.3%) | 5,001 (44.2%) | 0.00 | 6,088 (30.4%) | 6,071 (30.3%) | 0.00 |
| West; n (%) | 1,531 (17.6%) | 1,564 (18.0%) | -0.01 | 1,688 (14.9%) | 1,723 (15.2%) | -0.01 | 3,219 (16.1%) | 3,287 (16.4%) | -0.01 |
| Unknown+missing; n (%) | N/A | N/A | #VALUE! | 63 (0.6%) | 58 (0.5%) | 0.01 | 63 (0.3%) | 58 (0.3%) | 0.00 |
| CV Covariates | | | | | | | | | |
| schemic heart disease; n (%) | 2,835 (32.5%) | 2,813 (32.3%) | 0.00 | 3,786 (33.5%) | 3,714 (32.8%) | 0.01 | 6,621 (33.1%) | 6,527 (32.6%) | 0.01 |
| Acute MI; n (%) | 162 (1.9%) | 163 (1.9%) | 0.00 | 242 (2.1%) | 227 (2.0%) | 0.01 | 404 (2.0%) | 390 (1.9%) | 0.01 |
| ACS/unstable angina; n (%) | 225 (2.6%) | 221 (2.5%) | 0.01 | 423 (3.7%) | 421 (3.7%) | 0.00 | 648 (3.2%) | 642 (3.2%) | 0.00 |
| Old MI; n (%) | 381 (4.4%) | 386 (4.4%) | 0.00 | 193 (1.7%) | 205 (1.8%) | -0.01 | 574 (2.9%) | 591 (3.0%) | -0.01 |
| Stable angina; n (%) | 630 (7.2%) | 632 (7.3%) | 0.00 | 675 (6.0%) | 655 (5.8%) | 0.01 | 1,305 (6.5%) | 1,287 (6.4%) | 0.00 |
| Coronary atherosclerosis and other forms | 2,585 (29.7%) | 2,529 (29.0%) | 0.02 | 3,393 (30.0%) | 3,285 (29.0%) | 0.02 | 5,978 (29.9%) | 5,814 (29.0%) | 0.02 |
| of chronic ischemic heart disease; n (%) | () | | | () | () | | | () | |
| Other atherosclerosis with ICD10; n (%) | 137 (1.6%) | 138 (1.6%) | 0.00 | 209 (1.8%) | 245 (2.2%) | -0.03 | 346 (1.7%) | 383 (1.9%) | -0.02 |
| Previous cardiac procedure (CABG or PTCA<br>or Stent); n (%) | 98 (1.1%) | 88 (1.0%) | 0.01 | 188 (1.7%) | 205 (1.8%) | -0.01 | 286 (1.4%) | 293 (1.5%) | -0.01 |
| History of CABG or PTCA; n (%) | 656 (7.5%) | 652 (7.5%) | 0.00 | 366 (3.2%) | 343 (3.0%) | 0.01 | 1,022 (5.1%) | 0,995 (5.0%) | 0.00 |
| Any stroke; n (%) | 1,188 (13.6%) | 1,174 (13.5%) | 0.00 | 1,660 (14.7%) | 1,648 (14.6%) | 0.00 | 2,848 (14.2%) | 2,822 (14.1%) | 0.00 |
| schemic stroke (w and w/o mention of | 1,178 (13.5%) | 1,159 (13.3%) | 0.01 | 1,650 (14.6%) | 1,637 (14.5%) | 0.00 | 2,828 (14.1%) | 2,796 (14.0%) | 0.00 |
| cerebral infarction); n (%) | 1,170 (13.370) | 1,133 (13.370) | 0.01 | 1,050 (14.0%) | 1,037 (14.370) | 0.00 | 2,020 (14.170) | 2,750 (14.070) | 0.00 |
| Hemorrhagic stroke; n (%) | 29 (0.3%) | 34 (0.4%) | -0.02 | 32 (0.3%) | 34 (0.3%) | 0.00 | 61 (0.3%) | 68 (0.3%) | 0.00 |
| ΠΑ; n (%) | 307 (3.5%) | 290 (3.3%) | 0.01 | 432 (3.8%) | 446 (3.9%) | -0.01 | 739 (3.7%) | 736 (3.7%) | 0.00 |
| Other cerebrovascular disease; n (%) | 307 (3.5%) | 274 (3.1%) | 0.02 | 300 (2.7%) | 285 (2.5%) | 0.01 | 607 (3.0%) | 559 (2.8%) | 0.01 |
| Late effects of cerebrovascular disease; n | 239 (2.7%) | 231 (2.7%) | 0.00 | 217 (1.9%) | 203 (1.8%) | 0.01 | 456 (2.3%) | 434 (2.2%) | 0.01 |
| (%) | 222 (2.770) | 222 (2.774) | 2.00 | 22. (2.5%) | 202 (2.070) | 2.01 | .55 (2.570) | | 3.01 |
| Cerebrovascular procedure; n (%) | 26 (0.3%) | 23 (0.3%) | 0.00 | 54 (0.5%) | 63 (0.6%) | -0.01 | 80 (0.4%) | 86 (0.4%) | 0.00 |
| Heart failure (CHF); n (%) | 962 (11.0%) | 982 (11.3%) | -0.01 | 1,054 (9.3%) | 1,023 (9.0%) | 0.01 | 2,016 (10.1%) | 2,005 (10.0%) | 0.00 |
| Peripheral Vascular Disease (PVD) or PVD | 1,062 (12.2%) | 1,046 (12.0%) | 0.01 | 922 (8.1%) | 920 (8.1%) | 0.00 | 1,984 (9.9%) | 1,966 (9.8%) | 0.00 |
| Surgery; n (%) | 1,002 (12.2/0) | 1,010 (12.070) | 0.01 | 522 (0.176) | 520 (5.276) | 0.00 | 2,501 (5.570) | 1,500 (5.070) | 0.00 |
| Atrial fibrillation; n (%) | 909 (10.4%) | 882 (10.1%) | 0.01 | 1,066 (9.4%) | 1,071 (9.5%) | 0.00 | 1,975 (9.9%) | 1,953 (9.8%) | 0.00 |
| acidi normacion, ii (70) | 1,248 (14.3%) | 1,224 (14.1%) | 0.01 | 1,095 (9.7%) | 1,090 (9.6%) | 0.00 | 2,343 (11.7%) | 2,314 (11.6%) | 0.00 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Cardiac conduction disorders; n (%) | 313 (3.6%) | 318 (3.7%) | -0.01 | 293 (2.6%) | 240 (2.1%) | 0.03 | 606 (3.0%) | 558 (2.8%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| Other CVD; n (%) | 878 (10.1%) | 839 (9.6%) | 0.02 | 1,698 (15.0%) | 1,716 (15.2%) | -0.01 | 2,576 (12.9%) | 2,555 (12.8%) | 0.00 |
| Diabetes-related complications | | | | | | | | | |
| Diabetic retinopathy; n (%) | 761 (8.7%) | 727 (8.3%) | 0.01 | 656 (5.8%) | 634 (5.6%) | 0.01 | 1,417 (7.1%) | 1,361 (6.8%) | 0.01 |
| Diabetes with other ophthalmic manifestations; n (%) | 101 (1.2%) | 91 (1.0%) | 0.02 | 415 (3.7%) | 410 (3.6%) | 0.01 | 0,516 (2.6%) | 0,501 (2.5%) | 0.01 |
| Retinal detachment, vitreous hemorrhage,<br>vitrectomy; n (%) | 62 (0.7%) | 54 (0.6%) | 0.01 | 51 (0.5%) | 62 (0.5%) | 0.00 | 113 (0.6%) | 116 (0.6%) | 0.00 |
| Retinal laser coagulation therapy; n (%) | 69 (0.8%) | 82 (0.9%) | -0.01 | 131 (1.2%) | 139 (1.2%) | 0.00 | 200 (1.0%) | 221 (1.1%) | -0.01 |
| Occurrence of Diabetic Neuropathy ; n (%) | 1,526 (17.5%) | 1,497 (17.2%) | 0.01 | 839 (7.4%) | 845 (7.5%) | 0.00 | 2,365 (11.8%) | 2,342 (11.7%) | 0.00 |
| Occurrence of diabetic nephropathy with ICD10; n (%) | 1,320 (15.2%) | 1,308 (15.0%) | 0.01 | 581 (5.1%) | 574 (5.1%) | 0.00 | 1,901 (9.5%) | 1,882 (9.4%) | 0.00 |
| Hypoglycemia; n (%) | 113 (1.3%) | 120 (1.4%) | -0.01 | 229 (2.0%) | 237 (2.1%) | -0.01 | 0,342 (1.7%) | 0,357 (1.8%) | -0.01 |
| Hyperglycemia; n (%) | 379 (4.4%) | 364 (4.2%) | 0.01 | 139 (1.2%) | 137 (1.2%) | 0.00 | 0,518 (2.6%) | 0,501 (2.5%) | 0.01 |
| Disorders of fluid electrolyte and acid-base | 932 (10.7%) | 923 (10.6%) | 0.00 | 717 (6.3%) | 707 (6.2%) | 0.00 | 1,649 (8.2%) | 1,630 (8.1%) | 0.00 |
| balance; n (%) | _ | | | | | | | | |
| Diabetic ketoacidosis; n (%) | 20 (0.2%) | 16 (0.2%) | 0.00 | 21 (0.2%) | 23 (0.2%) | 0.00 | 41 (0.2%) | 39 (0.2%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic<br>syndrome (HONK); n (%) | 28 (0.3%) | 21 (0.2%) | 0.02 | 12 (0.1%) | 17 (0.2%) | -0.03 | 40 (0.2%) | 38 (0.2%) | 0.00 |
| Diabetes with peripheral circulatory<br>disorders with ICD-10; n (%) | 593 (6.8%) | 575 (6.6%) | 0.01 | 238 (2.1%) | 273 (2.4%) | -0.02 | 0,831 (4.2%) | 0,848 (4.2%) | 0.00 |
| Diabetic Foot; n (%) | 250 (2.9%) | 240 (2.8%) | 0.01 | 358 (3.2%) | 367 (3.2%) | 0.00 | 608 (3.0%) | 607 (3.0%) | 0.00 |
| Gangrene; n (%) | 18 (0.2%) | 14 (0.2%) | 0.00 | 17 (0.2%) | 16 (0.1%) | 0.03 | 35 (0.2%) | 30 (0.1%) | 0.03 |
| Lower extremity amputation; n (%) | 41 (0.5%) | 49 (0.6%) | -0.01 | 27 (0.2%) | 30 (0.3%) | -0.02 | 68 (0.3%) | 79 (0.4%) | -0.02 |
| Osteomyelitis; n (%) | 51 (0.6%) | 42 (0.5%) | 0.01 | 67 (0.6%) | 54 (0.5%) | 0.01 | 118 (0.6%) | 96 (0.5%) | 0.01 |
| Skin infections ; n (%) | 498 (5.7%) | 504 (5.8%) | 0.00 | 730 (6.5%) | 714 (6.3%) | 0.01 | 1,228 (6.1%) | 1,218 (6.1%) | 0.00 |
| Erectile dysfunction; n (%) | 203 (2.3%) | 215 (2.5%) | -0.01 | 130 (1.1%) | 131 (1.2%) | -0.01 | 0,333 (1.7%) | 0,346 (1.7%) | 0.00 |
| Diabetes with unspecified complication; n | 330 (3.8%) | 338 (3.9%) | -0.01 | 214 (1.9%) | 201 (1.8%) | 0.01 | 0,544 (2.7%) | 0,539 (2.7%) | 0.00 |
| (%) | (, | (, | | | | | -,, | -,, | |
| Diabetes mellitus without mention of complications; n (%) | 4,329 (49.7%) | 4,230 (48.6%) | 0.02 | 4,706 (41.6%) | 4,689 (41.4%) | 0.00 | 9,035 (45.1%) | 8,919 (44.5%) | 0.01 |
| Hypertension: 1 inpatient or 2 outpatient claims within 365 days; n (%) | 8,291 (95.2%) | 8,291 (95.2%) | 0.00 | 8,443 (74.6%) | 8,416 (74.4%) | 0.00 | 16,734 (83.6%) | 16,707 (83.4%) | 0.01 |
| Hyperlipidemia ; n (%) | 5,790 (66.5%) | 5,796 (66.5%) | 0.00 | 4,103 (36.3%) | 4,117 (36.4%) | 0.00 | 9,893 (49.4%) | 9,913 (49.5%) | 0.00 |
| Edema; n (%) | 1,228 (14.1%) | 1,220 (14.0%) | 0.00 | 1,011 (8.9%) | 985 (8.7%) | 0.01 | 2,239 (11.2%) | 2,205 (11.0%) | 0.01 |
| Renal Dysfunction (non-diabetic); n (%) | 2,558 (29.4%) | 2,576 (29.6%) | 0.00 | 1,921 (17.0%) | 1,831 (16.2%) | 0.02 | 4,479 (22.4%) | 4,407 (22.0%) | 0.01 |
| Occurrence of acute renal disease; n (%) | 357 (4.1%) | 338 (3.9%) | 0.01 | 314 (2.8%) | 306 (2.7%) | 0.01 | 671 (3.4%) | 644 (3.2%) | 0.01 |
| Occurrence of chronic renal insufficiency;<br>n (%) | 2,128 (24.4%) | 2,137 (24.5%) | 0.00 | 1,374 (12.1%) | 1,388 (12.3%) | -0.01 | 3,502 (17.5%) | 3,525 (17.6%) | 0.00 |
| Chronic kidney disease ; n (%) | 2,057 (23.6%) | 2,063 (23.7%) | 0.00 | 1,269 (11.2%) | 1,277 (11.3%) | 0.00 | 3,326 (16.6%) | 3,340 (16.7%) | 0.00 |
| CKD Stage 3-4; n (%) | 1,465 (16.8%) | 1,517 (17.4%) | -0.02 | 828 (7.3%) | 850 (7.5%) | -0.01 | 2,293 (11.5%) | 2,367 (11.8%) | -0.01 |
| Occurrence of hypertensive nephropathy;<br>n (%) | 1,135 (13.0%) | 1,134 (13.0%) | 0.00 | 546 (4.8%) | 534 (4.7%) | 0.00 | 1681 (8.4%) | 1668 (8.3%) | 0.00 |
| Occurrence of miscellaneous renal | 685 (7.9%) | 716 (8.2%) | -0.01 | 659 (5.8%) | 606 (5.4%) | 0.02 | 1,344 (6.7%) | 1,322 (6.6%) | 0.00 |
| insufficiency; n (%) | 2,104 (24.2%) | 2,009 (23.1%) | 0.03 | 2,288 (20.2%) | 2,198 (19.4%) | 0.02 | 4,392 (21.9%) | 4,207 (21.0%) | 0.02 |
| Glaucoma or cataracts; n (%) | | | 0.03 | | | | | | |
| Cellulitis or abscess of toe; n (%) | 126 (1.4%) | 124 (1.4%) | | 99 (0.9%) | 110 (1.0%) | -0.01 | 225 (1.1%) | 234 (1.2%) | -0.01 |
| Foot ulcer; n (%) | 243 (2.8%) | 240 (2.8%) | 0.00 | 370 (3.3%) | 378 (3.3%) | 0.00 | 613 (3.1%) | 618 (3.1%) | 0.00 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Bladder stones; n (%) | 10 (0.1%) | 11 (0.1%) | 0.00 | 7 (0.1%) | 7 (0.1%) | 0.00 | 17 (0.1%) | 18 (0.1%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Kidney stones; n (%) | 193 (2.2%) | 192 (2.2%) | 0.00 | 192 (1.7%) | 189 (1.7%) | 0.00 | 0,385 (1.9%) | 0,381 (1.9%) | 0.00 |
| Urinary tract infections (UTIs); n (%) | 987 (11.3%) | 997 (11.4%) | 0.00 | 787 (7.0%) | 788 (7.0%) | 0.00 | 1,774 (8.9%) | 1,785 (8.9%) | 0.00 |
| Dipstick urinalysis; n (%) | 3,368 (38.7%) | 3,400 (39.0%) | -0.01 | 2,729 (24.1%) | 2,756 (24.4%) | -0.01 | 6,097 (30.4%) | 6,156 (30.7%) | -0.01 |
| Non-dipstick urinalysis; n (%) | 2,594 (29.8%) | 2,560 (29.4%) | 0.01 | 1,392 (12.3%) | 1,386 (12.3%) | 0.00 | 3,986 (19.9%) | 3,946 (19.7%) | 0.01 |
| Urine function test; n (%) | 298 (3.4%) | 271 (3.1%) | 0.02 | 410 (3.6%) | 349 (3.1%) | 0.03 | 0,708 (3.5%) | 0,620 (3.1%) | 0.02 |
| Cytology; n (%) | 120 (1.4%) | 113 (1.3%) | 0.01 | 217 (1.9%) | 164 (1.4%) | 0.04 | 337 (1.7%) | 277 (1.4%) | 0.02 |
| Cystos; n (%) | 159 (1.8%) | 147 (1.7%) | 0.01 | 313 (2.8%) | 225 (2.0%) | 0.05 | 472 (2.4%) | 372 (1.9%) | 0.03 |
| Other Covariates | | ( | | , | (, | | , , , , , , | | |
| Liver disease: n (%) | 274 (3.1%) | 289 (3.3%) | -0.01 | 82 (0.7%) | 74 (0.7%) | 0.00 | 0,356 (1.8%) | 0,363 (1.8%) | 0.00 |
| Osteoarthritis; n (%) | 1,892 (21.7%) | 1,895 (21.8%) | 0.00 | 1,575 (13.9%) | 1,625 (14.4%) | -0.01 | 3,467 (17.3%) | 3,520 (17.6%) | -0.01 |
| Other arthritis, arthropathies and | 3,668 (42.1%) | 3,639 (41.8%) | 0.01 | 3,859 (34.1%) | 3,888 (34.4%) | -0.01 | 7,527 (37.6%) | 7,527 (37.6%) | 0.00 |
| musculoskeletal pain; n (%) | -,, | -,(, | | -,, | -,, | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | ,,, | |
| Dorsopathies; n (%) | 2,364 (27.1%) | 2,293 (26.3%) | 0.02 | 2,260 (20.0%) | 2,296 (20.3%) | -0.01 | 4,624 (23.1%) | 4,589 (22.9%) | 0.00 |
| Fractures; n (%) | 297 (3.4%) | 283 (3.2%) | 0.01 | 426 (3.8%) | 421 (3.7%) | 0.01 | 0,723 (3.6%) | 0,704 (3.5%) | 0.01 |
| Falls; n (%) | 353 (4.1%) | 344 (3.9%) | 0.01 | 88 (0.8%) | 78 (0.7%) | 0.01 | 441 (2.2%) | 422 (2.1%) | 0.01 |
| Osteoporosis; n (%) | 823 (9.4%) | 815 (9.4%) | 0.00 | 1,004 (8.9%) | 1,033 (9.1%) | -0.01 | 1,827 (9.1%) | 1,848 (9.2%) | 0.00 |
| Hyperthyroidism; n (%) | 69 (0.8%) | 74 (0.8%) | 0.00 | 50 (0.4%) | 63 (0.6%) | -0.03 | 119 (0.6%) | 137 (0.7%) | -0.01 |
| Hypothyroidism ; n (%) | 1,667 (19.1%) | 1,524 (17.5%) | 0.04 | 901 (8.0%) | 907 (8.0%) | 0.00 | 2,568 (12.8%) | 2,431 (12.1%) | 0.02 |
| Other disorders of thyroid gland; n (%) | 364 (4.2%) | 408 (4.7%) | -0.02 | 251 (2.2%) | 302 (2.7%) | -0.03 | 0,615 (3.1%) | 0,710 (3.5%) | -0.02 |
| Depression; n (%) | 679 (7.8%) | 636 (7.3%) | 0.02 | 511 (4.5%) | 514 (4.5%) | 0.00 | 1,190 (5.9%) | 1,150 (5.7%) | 0.01 |
| Anxiety, n (%) | 773 (8.9%) | 736 (8.5%) | 0.01 | 359 (3.2%) | 340 (3.0%) | 0.01 | 1,132 (5.7%) | 1,076 (5.4%) | 0.01 |
| SleepDisorder; n (%) | 588 (6.8%) | 571 (6.6%) | 0.01 | 1,084 (9.6%) | 1,078 (9.5%) | 0.00 | 1,672 (8.3%) | 1,649 (8.2%) | 0.00 |
| Dementia; n (%) | 413 (4.7%) | 394 (4.5%) | 0.01 | 330 (2.9%) | 321 (2.8%) | 0.01 | 743 (3.7%) | 715 (3.6%) | 0.01 |
| Delirium; n (%) | 109 (1.3%) | 116 (1.3%) | 0.00 | 105 (0.9%) | 104 (0.9%) | 0.00 | 214 (1.1%) | 220 (1.1%) | 0.00 |
| Psychosis; n (%) | 88 (1.0%) | 82 (0.9%) | 0.01 | 83 (0.7%) | 78 (0.7%) | 0.00 | 171 (0.9%) | 160 (0.8%) | 0.01 |
| Obesity; n (%) | 1,722 (19.8%) | 1,689 (19.4%) | 0.01 | 540 (4.8%) | 553 (4.9%) | 0.00 | 2,262 (11.3%) | 2,242 (11.2%) | 0.00 |
| Overweight; n (%) | 584 (6.7%) | 567 (6.5%) | 0.01 | 83 (0.7%) | 80 (0.7%) | 0.00 | 0,667 (3.3%) | 0,647 (3.2%) | 0.01 |
| Smoking; n (%) | 1,014 (11.6%) | 971 (11.1%) | 0.02 | 353 (3.1%) | 347 (3.1%) | 0.00 | 1,367 (6.8%) | 1,318 (6.6%) | 0.01 |
| Alcohol abuse or dependence; n (%) | 66 (0.8%) | 65 (0.7%) | 0.01 | 32 (0.3%) | 34 (0.3%) | 0.00 | 98 (0.5%) | 99 (0.5%) | 0.00 |
| Drug abuse or dependence; n (%) | 165 (1.9%) | 156 (1.8%) | 0.01 | 44 (0.4%) | 33 (0.3%) | 0.02 | 209 (1.0%) | 189 (0.9%) | 0.01 |
| COPD; n (%) | 1,182 (13.6%) | 1,134 (13.0%) | 0.02 | 1,116 (9.9%) | 1,107 (9.8%) | 0.00 | 2,298 (11.5%) | 2,241 (11.2%) | 0.01 |
| Asthma; n (%) | 664 (7.6%) | 654 (7.5%) | 0.00 | 600 (5.3%) | 588 (5.2%) | 0.00 | 1,264 (6.3%) | 1,242 (6.2%) | 0.00 |
| Obstructive sleep apnea; n (%) | 869 (10.0%) | 861 (9.9%) | 0.00 | 733 (6.5%) | 714 (6.3%) | 0.01 | 1,602 (8.0%) | 1,575 (7.9%) | 0.00 |
| Pneumonia; n (%) | 260 (3.0%) | 260 (3.0%) | 0.00 | 377 (3.3%) | 363 (3.2%) | 0.01 | 0,637 (3.2%) | 0,623 (3.1%) | 0.01 |
| Imaging, n (%) | 11 (0.1%) | 11 (0.1%) | 0.00 | 12 (0.1%) | 15 (0.1%) | 0.00 | 23 (0.1%) | 26 (0.1%) | 0.00 |
| Other Medications | (-:) | (0.2.5) | 0.00 | 22 (0.274) | 25 (0.275) | 0.00 | 22 (0.2.0) | 20 (0.274) | 0.00 |
| Use of ACE inhibitors; n (%) | 1,904 (21.9%) | 1,935 (22.2%) | -0.01 | 3,523 (31.1%) | 3,516 (31.1%) | 0.00 | 5,427 (27.1%) | 5,451 (27.2%) | 0.00 |
| Use of ARBs; n (%) | 4,132 (47.4%) | 8,710 (100.0%) | -1.49 | 3,674 (32.5%) | 11,314 (100.0%) | -2.04 | 7,806 (39.0%) | 20,024 (100.0%) | -1.77 |
| Use of Loop Diuretics - ; n (%) | 2,955 (33.9%) | 2,918 (33.5%) | 0.01 | 4,662 (41.2%) | 4,571 (40.4%) | 0.02 | 7,617 (38.0%) | 7,489 (37.4%) | 0.01 |
| Use of other diuretics-; n (%) | 401 (4.6%) | 388 (4.5%) | 0.00 | 528 (4.7%) | 500 (4.4%) | 0.01 | 0,929 (4.6%) | 0,888 (4.4%) | 0.01 |
| Use of nitrates-; n (%) | 821 (9.4%) | 800 (9.2%) | 0.01 | 1,578 (13.9%) | 1,532 (13.5%) | 0.01 | 2,399 (12.0%) | 2,332 (11.6%) | 0.01 |
| Use of other hypertension drugs; n (%) | 1,457 (16.7%) | 1,407 (16.2%) | 0.01 | 1,839 (16.3%) | 1,755 (15.5%) | 0.02 | 3,296 (16.5%) | 3,162 (15.8%) | 0.02 |
| Use of digoxin-; n (%) | 190 (2.2%) | 183 (2.1%) | 0.01 | 547 (4.8%) | 536 (4.7%) | 0.00 | 737 (3.7%) | 719 (3.6%) | 0.01 |
| Use of Anti-arrhythmics; n (%) | 210 (2.4%) | 221 (2.5%) | -0.01 | 411 (3.6%) | 393 (3.5%) | 0.01 | 621 (3.1%) | 614 (3.1%) | 0.00 |
| Use of COPD/asthma meds-; n (%) | 1,837 (21.1%) | 1,805 (20.7%) | 0.01 | 2,441 (21.6%) | 2,343 (20.7%) | 0.02 | 4,278 (21.4%) | 4,148 (20.7%) | 0.02 |
| Use of statins; n (%) | 5,780 (66.4%) | 5,815 (66.8%) | -0.01 | 7,194 (63.6%) | 7,201 (63.6%) | 0.02 | 12,974 (64.8%) | 13,016 (65.0%) | 0.02 |
| Use of other lipid-lowering drugs; n (%) | 938 (10.8%) | 957 (11.0%) | -0.01 | 1,796 (15.9%) | 1,820 (16.1%) | -0.01 | 2,734 (13.7%) | 2,777 (13.9%) | -0.01 |
| oscorodia iipia iowering drugs, ii (70) | 330 (10.070) | 337 (22.070) | -0.01 | 1,750 (15.570) | 1,020 (10.1/0) | 0.01 | 2,134 (13.170) | 2,777 (13.370) | 0.01 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| I | | () | | | | | () | | 1 |
|---|---|---|---|---|---|---|---|---|---|
| Use of oral anticoagulants (Dabigatran, | 770 (8.8%) | 765 (8.8%) | 0.00 | 1,228 (10.9%) | 1,207 (10.7%) | 0.01 | 1,998 (10.0%) | 1,972 (9.8%) | 0.01 |
| Rivaroxaban, Apixaban, Warfarin); n (%) | () | () | | | | | | () | |
| Use of heparin and other low-molecular | 42 (0.5%) | 40 (0.5%) | 0.00 | 2 (0.0%) | 2 (0.0%) | #DIV/0! | 44 (0.2%) | 42 (0.2%) | 0.00 |
| weight heparins; n (%) | 4 440 (45 50/) | 4 454 (45 00/) | | 4 700 (45 00) | 4 705 (45 70) | 0.00 | 3 450 (45 00/) | 2 400 (45 00) | 0.00 |
| Use of NSAIDs; n (%) | 1,440 (16.5%) | 1,464 (16.8%) | -0.01 | 1,720 (15.2%) | 1,726 (15.3%) | 0.00 | 3,160 (15.8%) | 3,190 (15.9%) | 0.00 |
| Use of oral corticosteroids; n (%) | 1,804 (20.7%) | 1,806 (20.7%) | 0.00 | 2,220 (19.6%) | 2,175 (19.2%) | 0.01 | 4,024 (20.1%) | 3,981 (19.9%) | 0.01 |
| Use of bisphosphonate (); n (%) | 419 (4.8%) | 410 (4.7%) | 0.00 | 746 (6.6%) | 784 (6.9%) | -0.01 | 1165 (5.8%) | 1194 (6.0%) | -0.01 |
| Use of opioids-; n (%) | 2,333 (26.8%) | 2,334 (26.8%) | 0.00 | 3,670 (32.4%) | 3,614 (31.9%) | 0.01 | 6,003 (30.0%) | 5,948 (29.7%) | 0.01 |
| Use of antidepressants; n (%) | 2,184 (25.1%) | 2,119 (24.3%) | 0.02 | 2,782 (24.6%) | 2,733 (24.2%) | 0.01 | 4,966 (24.8%) | 4,852 (24.2%) | 0.01 |
| Use of antipsychotics; n (%) | 195 (2.2%) | 183 (2.1%) | 0.01 | 245 (2.2%) | 234 (2.1%) | 0.01 | 0,440 (2.2%) | 0,417 (2.1%) | 0.01 |
| Use of anticonvulsants; n (%) | 1,571 (18.0%) | 1,512 (17.4%) | 0.02 | 1,513 (13.4%) | 1,521 (13.4%) | 0.00 | 3,084 (15.4%) | 3,033 (15.1%) | 0.01 |
| Use of lithium-; n (%) | 15 (0.2%) | 5 (0.1%) | 0.03 | 13 (0.1%) | 9 (0.1%) | 0.00 | 28 (0.1%) | 14 (0.1%) | 0.00 |
| Use of Benzos- ; n (%) | 1,127 (12.9%) | 1,119 (12.8%) | 0.00 | 2,017 (17.8%) | 1,993 (17.6%) | 0.01 | 3,144 (15.7%) | 3,112 (15.5%) | 0.01 |
| Use of anxiolytics/hypnotics-; n (%) | 584 (6.7%) | 609 (7.0%) | -0.01 | 1,176 (10.4%) | 1,141 (10.1%) | 0.01 | 1,760 (8.8%) | 1,750 (8.7%) | 0.00 |
| Use of dementia meds-; n (%) | 281 (3.2%) | 279 (3.2%) | 0.00 | 341 (3.0%) | 345 (3.0%) | 0.00 | 622 (3.1%) | 624 (3.1%) | 0.00 |
| Use of antiparkinsonian meds-; n (%) | 255 (2.9%) | 245 (2.8%) | 0.01 | 375 (3.3%) | 358 (3.2%) | 0.01 | 0,630 (3.1%) | 0,603 (3.0%) | 0.01 |
| Entresto (sacubitril/valsartan); n (%) | 24 (0.3%) | 1 (0.0%) | 0.08 | 4 (0.0%) | 0 (0.0%) | #DIV/0! | 28 (0.1%) | 1 (0.0%) | 0.04 |
| Labs | | | | | | | | | |
| Lab values- HbA1c (%); n (%) | 2,219 (25.5%) | 2,160 (24.8%) | 0.02 | 141 (1.2%) | 113 (1.0%) | 0.02 | 2,360 (11.8%) | 2,273 (11.4%) | 0.01 |
| Lab values- HbA1c (%) (within 3 months); n<br>(%) | 1,546 (17.7%) | 1,488 (17.1%) | 0.02 | 104 (0.9%) | 70 (0.6%) | 0.03 | 1,650 (8.2%) | 1,558 (7.8%) | 0.01 |
| Lab values- HbA1c (%) (within 6 months); n<br>(%) | 2,219 (25.5%) | 2,160 (24.8%) | 0.02 | 141 (1.2%) | 113 (1.0%) | 0.02 | 2,360 (11.8%) | 2,273 (11.4%) | 0.01 |
| Lab values- BNP; n (%) | 103 (1.2%) | 99 (1.1%) | 0.01 | 3 (0.0%) | 4 (0.0%) | #DIV/0! | 106 (0.5%) | 103 (0.5%) | 0.00 |
| Lab values- BNP (within 3 months); n (%) | 83 (1.0%) | 66 (0.8%) | 0.02 | 3 (0.0%) | 1 (0.0%) | #DIV/0! | 86 (0.4%) | 67 (0.3%) | 0.02 |
| Lab values-BNP (within 6 months); n (%) | 103 (1.2%) | 99 (1.1%) | 0.01 | 3 (0.0%) | 4 (0.0%) | #DIV/0! | 106 (0.5%) | 103 (0.5%) | 0.00 |
| Lab values- BUN (mg/dl); n (%) | 3,095 (35.5%) | 3,059 (35.1%) | 0.01 | 118 (1.0%) | 139 (1.2%) | -0.02 | 3,213 (16.0%) | 3,198 (16.0%) | 0.00 |
| Lab values-BUN (mg/dl) (within 3 months); | 2,258 (25.9%) | 2,203 (25.3%) | 0.01 | 83 (0.7%) | 96 (0.8%) | -0.01 | 2,341 (11.7%) | 2,299 (11.5%) | 0.01 |
| n (%) | | | | | | | | | |
| Lab values-BUN (mg/dl) (within 6 months); | 3,095 (35.5%) | 3,059 (35.1%) | 0.01 | 118 (1.0%) | 139 (1.2%) | -0.02 | 3,213 (16.0%) | 3,198 (16.0%) | 0.00 |
| n (%) | | | | | | | | | |
| Lab values-Creatinine (mg/dl); n (%) | 3,209 (36.8%) | 3,164 (36.3%) | 0.01 | 122 (1.1%) | 150 (1.3%) | -0.02 | 3,331 (16.6%) | 3,314 (16.6%) | 0.00 |
| Lab values- Creatinine (mg/dl) (within 3 | 2,349 (27.0%) | 2,272 (26.1%) | 0.02 | 85 (0.8%) | 106 (0.9%) | -0.01 | 2,434 (12.2%) | 2,378 (11.9%) | 0.01 |
| months); n (%) | | | | | | | | | |
| Lab values- Creatinine (mg/dl) (within 6 | 3,209 (36.8%) | 3,164 (36.3%) | 0.01 | 122 (1.1%) | 150 (1.3%) | -0.02 | 3,331 (16.6%) | 3,314 (16.6%) | 0.00 |
| months); n (%) | | | | | | | | | |
| Lab values- HDL level (mg/dl); n (%) | 2,385 (27.4%) | 2,343 (26.9%) | 0.01 | 117 (1.0%) | 101 (0.9%) | 0.01 | 2,502 (12.5%) | 2,444 (12.2%) | 0.01 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 1,570 (18.0%) | 1,511 (17.3%) | 0.02 | 81 (0.7%) | 60 (0.5%) | 0.03 | 1,651 (8.2%) | 1,571 (7.8%) | 0.01 |
| Lab values- HDL level (mg/dl) (within 6<br>months); n (%) | 2,385 (27.4%) | 2,343 (26.9%) | 0.01 | 117 (1.0%) | 101 (0.9%) | 0.01 | 2,502 (12.5%) | 2,444 (12.2%) | 0.01 |
| Lab values-LDL level (mg/dl); n (%) | 2,504 (28.7%) | 2,452 (28.2%) | 0.01 | 130 (1.1%) | 106 (0.9%) | 0.02 | 2,634 (13.2%) | 2,558 (12.8%) | 0.01 |
| Lab values-LDL level (mg/dl) (within 3 months); n (%) | 1,640 (18.8%) | 1,587 (18.2%) | 0.02 | 94 (0.8%) | 61 (0.5%) | 0.04 | 1,734 (8.7%) | 1,648 (8.2%) | 0.02 |
| Lab values-LDL level (mg/dl) (within 6 | 2,504 (28.7%) | 2,452 (28.2%) | 0.01 | 130 (1.1%) | 106 (0.9%) | 0.02 | 2,634 (13.2%) | 2,558 (12.8%) | 0.01 |
| months); n (%) | | | | | | | | | |
| Lab values- NT-proBNP; n (%) | 17 (0.2%) | 18 (0.2%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 17 (0.1%) | 18 (0.1%) | 0.00 |
| Lab values- NT-proBNP (within 3 months); | 12 (0.1%) | 9 (0.1%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 12 (0.1%) | 9 (0.0%) | 0.04 |
| n (%) | • | | | • | | - | • | | |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Lab values-NT-proBNP (within 6 months);<br>n (%) | 17 (0.2%) | 18 (0.2%) | 0.00 | 0 (0.0%) | 0 (0.0%) | #DIV/0! | 17 (0.1%) | 18 (0.1%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Lab values-Total cholesterol (mg/dl); n (%) | 2,465 (28.3%) | 2,426 (27.9%) | 0.01 | 127 (1.1%) | 106 (0.9%) | 0.02 | 2,592 (12.9%) | 2,532 (12.6%) | 0.01 |
| Lab values-Total cholesterol (mg/dl)<br>(within 3 months); n (%) | 1,611 (18.5%) | 1,569 (18.0%) | 0.01 | 89 (0.8%) | 61 (0.5%) | 0.04 | 1,700 (8.5%) | 1,630 (8.1%) | 0.01 |
| Lab values-Total cholesterol (mg/dl)<br>(within 6 months); n (%) | 2,465 (28.3%) | 2,426 (27.9%) | 0.01 | 127 (1.1%) | 106 (0.9%) | 0.02 | 2,592 (12.9%) | 2,532 (12.6%) | 0.01 |
| Lab values-Triglyceride level (mg/dl); n (%) | 2,424 (27.8%) | 2,396 (27.5%) | 0.01 | 125 (1.1%) | 106 (0.9%) | 0.02 | 2,549 (12.7%) | 2,502 (12.5%) | 0.01 |
| Lab values-Triglyceride level (mg/dl)<br>(within 3 months); n (%) | 1,590 (18.3%) | 1,552 (17.8%) | 0.01 | 87 (0.8%) | 61 (0.5%) | 0.04 | 1,677 (8.4%) | 1,613 (8.1%) | 0.01 |
| Lab values-Triglyceride level (mg/dl)<br>(within 6 months); n (%) | 2,424 (27.8%) | 2,396 (27.5%) | 0.01 | 125 (1.1%) | 106 (0.9%) | 0.02 | 2,549 (12.7%) | 2,502 (12.5%) | 0.01 |
| Lab result number- HbA1c (%) mean (only 2 to 20 included) | 2,183 | 2,127 | | 112 | 113 | | 0 | 0 | |
| mean (sd) | 7.00 (1.50) | 6.86 (1.38) | 0.10 | 7.64 (1.66) | 7.31 (1.77) | 0.19 | 7.36 (1.59) | 7.11 (1.61) | 0.16 |
| median [IQR] | 6.60 [6.00, 7.70] | 6.50 [5.90, 7.47] | 0.07 | 7.10 [6.40, 8.50] | 6.90 [6.10, 7.80] | 0.12 | 6.88 (1.59) | 6.73 (1.61) | 0.09 |
| Missing; n (%) | 6,527 (74.9%) | 6,583 (75.6%) | -0.02 | 11,202 (99.0%) | 11,201 (99.0%) | 0.00 | 17,729 (88.5%) | 17,784 (88.8%) | -0.01 |
| Lab result number- BNP mean | 103 | 99 | | 3 | 4 | | 0 | 0 | |
| mean (sd) | 159.45 (288.42) | 142.08 (206.91) | 0.07 | 169.00 (139.82) | 66.00 (28.53) | 1.02 | 164.85 (217.32) | 99.09 (138.14) | 0.36 |
| median [IQR] | 74.00 [37.00,<br>196.00] | 69.85 [37.00,<br>147.97] | 0.02 | 239.00 [8.00,<br>260.00] | 62.50 [41.25,<br>94.25] | 1.75 | 167.23 (217.32) | 65.70 (138.14) | 0.56 |
| Missing; n (%) | 8,607 (98.8%) | 8,611 (98.9%) | -0.01 | 11,311 (100.0%) | 11,310 (100.0%) | #DIV/0! | 19,918 (99.5%) | 19,921 (99.5%) | 0.00 |
| Lab result number- BUN (mg/dl) mean | 3,095 | 3,059 | | 118 | 139 | | 0 | 0 | |
| mean (sd) | 20.21 (10.19) | -88.29 (6,026.94) | 0.03 | 20.87 (12.48) | 22.01 (13.02) | -0.09 | 20.58 (11.54) | -25.97 (3974.92) | 0.02 |
| median [IQR] | 18.00 [14.00, 24.00] | 18.00 [14.00, 24.00] | 0.00 | 18.00 [13.97,<br>23.54] | 19.00 [14.50,<br>25.50] | -0.08 | 18.00 (11.54) | 18.57 (3974.92) | 0.00 |
| Missing; n (%) | 5,615 (64.5%) | 5,651 (64.9%) | -0.01 | 11,196 (99.0%) | 11,175 (98.8%) | 0.02 | 16,811 (84.0%) | 16,826 (84.0%) | 0.00 |
| Lab result number- Creatinine (mg/dl)<br>mean (only 0.1 to 15 included) | 3,129 | 3,079 | | 116 | 139 | | 3,245 | 3,218 | |
| mean (sd) | 1.17 (0.70) | 1.16 (0.62) | 0.02 | 1.22 (0.92) | 1.29 (1.13) | -0.07 | 1.20 (0.83) | 1.23 (0.94) | -0.03 |
| median [IQR] | 1.01 [0.82, 1.29] | 1.02 [0.84, 1.30] | -0.02 | 1.00 [0.84, 1.25] | 1.00 [0.83, 1.33] | 0.00 | 1.00 (0.83) | 1.01 (0.94) | -0.01 |
| Missing; n (%) | 5,581 (64.1%) | 5,631 (64.6%) | -0.01 | 11,198 (99.0%) | 11,175 (98.8%) | 0.02 | 16,779 (83.8%) | 16,806 (83.9%) | 0.00 |
| Lab result number- HDL level (mg/dl) mean<br>(only =<5000 included) | 2,385 | 2,343 | | 117 | 101 | | 2,502 | 2,444 | |
| mean (sd) | 49.89 (17.01) | 50.86 (17.23) | -0.06 | 46.19 (13.54) | 46.22 (13.42) | 0.00 | 47.80 (15.15) | 48.24 (15.20) | -0.03 |
| median [IQR] | | 49.00 [40.00, 60.00] | -0.06 | 44.00 [36.00,<br>54.00] | 44.00 [36.00,<br>53.50] | 0.00 | 45.74 (15.15) | 46.17 (15.20) | -0.03 |
| Missing; n (%) | 6,325 (72.6%) | 6,367 (73.1%) | -0.01 | 11,197 (99.0%) | 11,213 (99.1%) | -0.01 | 17,522 (87.5%) | 17,580 (87.8%) | -0.01 |
| Lab result number-LDL level (mg/dl) mean<br>(only =<5000 included) | 2,464 | 2,422 | | 121 | 103 | | 2,585 | 2,525 | |
| mean (sd) | -320.39 (20,147.33) | -1,566.06<br>(40,617.30) | 0.04 | 86.82 (39.78) | 85.48 (41.86) | 0.03 | -90.31 (13287.68) | -632.90 (26788.09) | 0.03 |
| median [IQR] | 83.00 [62.00,<br>108.00] | 82.00 [63.00,<br>106.00] | 0.00 | 81.00 [62.00,<br>110.00] | 77.00 [57.00,<br>118.00] | 0.10 | 81.87 (13287.68) | 79.17 (26788.09) | 0.00 |
| Missing; n (%) | 6,246 (71.7%) | 6,288 (72.2%) | -0.01 | 11,193 (98.9%) | 11,211 (99.1%) | -0.02 | 17,439 (87.1%) | 17,499 (87.4%) | -0.01 |
| Lab result number- Total cholesterol | 2,464 | 2,422 | | 127 | 106 | | 2,591 | 2,528 | |
| (mg/dl) mean (only =<5000 included) | | - | | | | | - | - | |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| | 1 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Maining n (N 191.00 191.50 | mean (sd) | 163.82 (48.07) | 165.75 (48.76) | -0.04 | 167.44 (40.25) | 171.71 (59.13) | -0.08 | 165.87 (43.82) | 169.12 (54.86) | -0.07 |
| Lab result number - Trigly cardie level (might) man (m | median [IQR] | | | -0.02 | | | 0.08 | 163.13 (43.82) | 161.30 (54.86) | 0.04 |
| | Missing; n (%) | 6,246 (71.7%) | 6,288 (72.2%) | -0.01 | 11,187 (98.9%) | 11,208 (99.1%) | -0.02 | 17,433 (87.1%) | 17,496 (87.4%) | -0.01 |
| mean (al) 143,07 91,94 142,08 90,61 100,18 100,00 122,05 100,00 121,00 171,00 171,00 172,00 171,00 171,00 172,00 171,00 172,00 172,00 172,00 172,00 171,00 172,00 | Lab result number-Triglyceride level | 2,424 | 2,396 | | 125 | 106 | | 2,549 | 2,502 | |
| | (mg/dl) mean (only =<5000 included) | | | | | | | | | |
| Missing_n N | mean (sd) | 143.07 (91.94) | 142.08 (90.61) | 0.01 | 165.02 (106.63) | 203.39 (411.31) | -0.13 | 155.47 (100.50) | 176.72 (314.90) | -0.09 |
| Lab result number - Hemoglobin mean (only \( \) 1.29 \( \) 1.85 \\ 2.321 \\ 2.3231 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ | median [IQR] | | | 0.02 | • | | 0.00 | 131.82 (100.50) | 132.02 (314.90) | 0.00 |
| Lab result number - Hemoglobin mean (only \( \) 1.29 \( \) 1.85 \\ 2.321 \\ 2.3231 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ 2.321 \\ | Missing: n (%) | 6.286 (72.2%) | 6.314 (72.5%) | -0.01 | 11.189 (98.9%) | 11.208 (99.1%) | -0.02 | 17.475 (87.3%) | 17.522 (87.5%) | -0.01 |
| | Lab result number- Hemoglobin mean | | | | 82 | 101 | | 2,436 | 2,422 | |
| | (only >0 included) | | • | | | | | | | |
| Missing n (%) | mean (sd) | 12.99 (1.68) | 12.92 (1.72) | 0.04 | 13.04 (1.78) | • | -0.14 | 13.02 (1.74) | | -0.11 |
| Lab result number - Serum sodium mean (only >0 and <190 included) mean (sd) | median [IQR] | 13.00 [11.90, 14.10] | 12.93 [11.75, 14.05] | 0.04 | • • | • • | 0.00 | 13.00 (1.74) | 13.03 (747952.25) | 0.00 |
| Conty-90 and <190 included | Missing; n (%) | 6,356 (73.0%) | 6,389 (73.4%) | -0.01 | 11,232 (99.3%) | 11,213 (99.1%) | 0.02 | 17,588 (87.8%) | 17,602 (87.9%) | 0.00 |
| 140.50 139.00 | Lab result number-Serum sodium mean<br>(only > 90 and < 190 included) | 3,059 | 3,040 | | 110 | 125 | | 3,169 | 3,165 | |
| 142.00 142.00 142.00 141.00 141.42 | mean (sd) | 140.35 (3.02) | 140.39 (2.92) | -0.01 | 139.32 (2.59) | 139.72 (2.65) | -0.15 | 139.77 (2.79) | 140.01 (2.77) | -0.09 |
| Lab result number- Albumin mean (only >0 and <=10 included) and <=10 included)mean (sd)median [IQR] 4.16 (0.36) 4.20 [4.00, 4.40] 5.828 (67.0%) 5.82 | median [IQR] | | | -0.15 | | | -0.19 | 139.93 (2.79) | 140.41 (2.77) | -0.17 |
| | Missing; n (%) | 5,651 (64.9%) | 5,670 (65.1%) | 0.00 | 11,204 (99.0%) | 11,189 (98.9%) | 0.01 | 16,855 (84.2%) | 16,859 (84.2%) | 0.00 |
| mean (sd) | Lab result number- Albumin mean (only >0 | 2,872 | 2,834 | | 102 | 124 | | 2,974 | 2,958 | |
| median [OR] | and <=10 included) | | | | | | | | | |
| 1,000 1,00 | mean (sd) | 4.16 (0.36) | 4.20 (0.36) | -0.11 | 4.15 (0.38) | 4.12 (0.40) | 0.08 | 4.15 (0.37) | 4.15 (0.38) | 0.00 |
| Lab result number - Glucose (fasting or random) mean (only 10-1000 included)mean (sd) 128.09 (53.05) 123.35 (46.88) 0.09 153.54 (67.14) 145.57 (62.13) 0.12 142.47 (61.41) 135.90 (56.01) 0.11 1median [toR] 111.00 [95.00, 146.00] 138.00] 178.50] 165.00] 165.00] 178.50] 165.00] 178.50] 165.00] 178.50] 165.00] 178.50] 165.00] | median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 0.00 | 4.18 [4.00, 4.40] | 4.13 [3.95, 4.37] | 0.13 | 4.19 (0.37) | 4.16 (0.38) | 0.08 |
| random) mean (only 10-1000 included)mean (sd)mean | Missing; n (%) | 5,838 (67.0%) | 5,876 (67.5%) | -0.01 | 11,212 (99.1%) | 11,190 (98.9%) | 0.02 | 17,050 (85.1%) | 17,066 (85.2%) | 0.00 |
| 128.09 (53.05) 123.35 (46.88) 0.09 153.54 (67.14) 145.57 (62.13) 0.12 142.47 (61.41) 135.90 (56.01) 0.11 | Lab result number- Glucose (fasting or | 3,051 | 3,028 | | 102 | 123 | | 3,153 | 3,151 | |
| 111.00 [95.00, 108.50 [95.00, 0.05 135.25 [103.81, 133.00 [104.00, 0.03 124.70 [61.41] 122.34 [56.01] 0.04 146.00] 138.00] 138.00] 178.50] 165.00] 178.50] 166.00] 178.50] 178.50] 178.50] 165.00] 178.50] 178.50] 165.00] 178.50] 178 | random) mean (only 10-1000 included) | | | | | | | | | |
| 146.00] 138.00] 178.50] 165.00] 165.00 | mean (sd) | 128.09 (53.05) | 123.35 (46.88) | 0.09 | 153.54 (67.14) | 145.57 (62.13) | 0.12 | 142.47 (61.41) | 135.90 (56.01) | 0.11 |
| Lab result number- Potassium mean (only 1-7 included)mean (sd)mean (sd)median [IQR]median [IQR | median [IQR] | | | 0.05 | | • | 0.03 | 124.70 (61.41) | 122.34 (56.01) | 0.04 |
| 1-7 included)mean (sd)mean (sd)median [IQR]median [IQR]mean (sd)median [IQR]median | Missing; n (%) | 5,659 (65.0%) | 5,682 (65.2%) | 0.00 | 11,212 (99.1%) | 11,191 (98.9%) | 0.02 | 16,871 (84.3%) | 16,873 (84.3%) | 0.00 |
| median [IQR] 4.40 [4.10, 4.70] 4.35 [4.07, 4.65] 0.11 4.27 [4.00, 4.55] 4.30 [4.00, 4.60] -0.06 4.33 (0.48) 4.32 (0.50) 0.02 median [IQR] 4.40 [4.10, 4.70] 5,590 (64.2%) 5,619 (64.5%) -0.01 11,196 (99.0%) 11,176 (98.8%) 0.02 16,786 (83.8%) 16,795 (83.9%) 0.00 mean (sd) 3.09 (2.05) 3.06 (2.02) 0.01 2.11 (1.74) 2.09 (1.70) 0.01 2.54 (1.88) 2.51 (1.85) 0.02 median [IQR] 3.00 [1.00, 4.00] 3.00 [1.00, 4.00] 0.00 2.00 [1.00, 3.00] 0.00 2.43 (1.88) 2.43 (1.85) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.18 (0.06) 0.18 (0.06) 0.00 0.17 (0.05) 0.17 (0.05) 0.00 0.17 (0.05) 0.17 (0.05) 0.00 median [IQR] 0.17 [0.14, 0.21] 0.17 [0.14, 0.21] 0.00 0.16 [0.14, 0.20] 0.16 [0.14, 0.20] 0.00 0.16 (0.05) 0.16 (0.05) 0.00 Healthcare Utilization | Lab result number- Potassium mean (only 1-7 included) | 3,120 | 3,091 | | 118 | 138 | | 3,238 | 3,229 | |
| Missing, n (%) Comorbidity Scores CCI (180 days)- ICD9 and ICD10mean (sd)median [IQR] Frailty Score (mean): Empirical Version 365 days,mean (sd)mean (sd) . | mean (sd) | 4.41 (0.46) | 4.37 (0.48) | 0.09 | 4.29 (0.49) | 4.30 (0.51) | -0.02 | 4.34 (0.48) | 4.33 (0.50) | 0.02 |
| Comorbidity Scores CCI (180 days)-ICD9 and ICD10mean (sd)mean (sd)median [IQR] Strailty Score (mean): Empirical Version 365 days,mean (sd)mean (sd) 0.18 (0.06) 0.18 (0.06) 0.17 [0.14, 0.21] 0.17 [0.14, 0.21] 0.17 [0.14, 0.21] 0.18 (0.05) 0.19 (0.05) 0.10 (0.05) 0.10 (0.14, 0.20) 0.10 (0.14, 0.20) 0.10 (0.14, 0.20) 0.11 (1.74) 0.10 (1.00, 3.00) 0.10 (1.00, | median [IQR] | 4.40 [4.10, 4.70] | 4.35 [4.07, 4.65] | 0.11 | 4.27 [4.00, 4.55] | 4.30 [4.00, 4.60] | -0.06 | 4.33 (0.48) | 4.32 (0.50) | 0.02 |
| CCI (180 days)-ICD9 and ICD10mean (sd) 3.09 (2.05) 3.06 (2.02) 0.01 2.11 (1.74) 2.09 (1.70) 0.01 2.54 (1.88) 2.51 (1.85) 0.02 2.00 [1.00, 3.00] 0.00 2.01 (0.05) 0.00 0.00 0.00 0.00 0.00 0.00 0.00 | Missing; n (%) | 5,590 (64.2%) | 5,619 (64.5%) | -0.01 | 11,196 (99.0%) | 11,176 (98.8%) | 0.02 | 16,786 (83.8%) | 16,795 (83.9%) | 0.00 |
| mean (sd) 3.09 (2.05) 3.06 (2.02) 0.01 2.11 (1.74) 2.09 (1.70) 0.01 2.54 (1.88) 2.51 (1.85) 0.02median [IQR] 3.00 [1.00, 4.00] 3.00 [1.00, 3.00] 3.00 | Comorbidity Scores | I | | | | | | | | |
| median [IQR] 3.00 [1.00, 4.00] 3.00 [1.00, 4.00] 0.00 2.00 [1.00, 3.00] 0.00 2.43 (1.88) 2.43 (1.85) 0.00 Frailty Score (mean): Empirical Version 365 days,mean (sd) 0.18 (0.06) 0.18 (0.06) 0.00 0.17 (0.05) 0.17 (0.05) 0.00 0.17 (0.05) 0.17 (0.05) 0.00 median [IQR] 0.17 [0.14, 0.21] 0.17 [0.14, 0.21] 0.00 0.16 [0.14, 0.20] 0.16 [0.14, 0.20] 0.00 0.16 (0.05) 0.16 (0.05) 0.00 Healthcare Utilization | CCI (180 days)-ICD9 and ICD10 | | | | | | | | | |
| Frailty Score (mean): Empirical Version 365 days, mean (sd) 0.18 (0.06) 0.18 (0.06) 0.17 (0.05) 0.17 (0.05) 0.17 (0.05) 0.17 (0.05) 0.17 (0.05) 0.17 (0.05) 0.17 (0.05) 0.16 (0.05) 0.16 (0.05) 0.16 (0.05) 0.17 (0.05) | mean (sd) | 3.09 (2.05) | 3.06 (2.02) | 0.01 | 2.11 (1.74) | 2.09 (1.70) | 0.01 | 2.54 (1.88) | 2.51 (1.85) | 0.02 |
| days,mean (sd)mean (sd) 0.18 (0.06) 0.18 (0.06) 0.17 (0.05) 0.18 (0.05) 0.19 (0.05) 0.19 (0.05) 0.10 (0.05) 0.10 (0.05) 0.10 (0.05) 0.10 (0.05) 0.10 (0.05) 0.10 (0.05) | median [IQR] | 3.00 [1.00, 4.00] | 3.00 [1.00, 4.00] | 0.00 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 2.43 (1.88) | 2.43 (1.85) | 0.00 |
| mean (sd) 0.18 (0.06) 0.18 (0.06) 0.00 0.17 (0.05) 0.17 (0.05) 0.00 0.17 (0.05) 0.17 (0.05) 0.00median [IQR] 0.17 [0.14, 0.21] 0.17 [0.14, 0.21] 0.00 0.16 [0.14, 0.20] 0.16 [0.14, 0.20] 0.00 0.16 (0.05) 0.16 (0.05) 0.00 0.16 (0.05) | Frailty Score (mean): Empirical Version 365 | | | | | | | | | |
| median [IQR] 0.17 [0.14, 0.21] 0.17 [0.14, 0.21] 0.00 0.16 [0.14, 0.20] 0.16 [0.14, 0.20] 0.00 0.16 (0.05) 0.16 (0.05) 0.00 Healthcare Utilization | days, | | | | | | | | | |
| Healthcare Utilization | mean (sd) | | | | | | | | | |
| | | 0.17 [0.14, 0.21] | 0.17 [0.14, 0.21] | 0.00 | 0.16 [0.14, 0.20] | 0.16 [0.14, 0.20] | 0.00 | 0.16 (0.05) | 0.16 (0.05) | 0.00 |
| Any hospitalization; n (%) 894 (10.3%) 868 (10.0%) 0.01 1,833 (16.2%) 1,769 (15.6%) 0.02 2,727 (13.6%) 2,637 (13.2%) 0.01 | | | | | | | | | | |
| | Any hospitalization; n (%) | 894 (10.3%) | 868 (10.0%) | 0.01 | 1,833 (16.2%) | 1,769 (15.6%) | 0.02 | 2,727 (13.6%) | 2,637 (13.2%) | 0.01 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Any hospitalization during prior 31-180 | 706 (8.1%) | 680 (7.8%) | 0.01 | 1,440 (12.7%) | 1,401 (12.4%) | 0.01 | 2,146 (10.7%) | 2,081 (10.4%) | 0.01 | I |
|---|---|---|---|---|---|---|---|---|---|---|
| days; n (%) | | | | | | | | | | ı |
| Endocrinologist Visit; n (%) | 726 (8.3%) | 711 (8.2%) | 0.00 | 711 (6.3%) | 736 (6.5%) | -0.01 | 1,437 (7.2%) | 1,447 (7.2%) | 0.00 | ı |
| Endocrinologist Visit (30 days prior); n (%) | 250 (2.9%) | 246 (2.8%) | 0.01 | 254 (2.2%) | 271 (2.4%) | -0.01 | 0,504 (2.5%) | 0,517 (2.6%) | -0.01 | ı |
| Endocrinologist Visit (31 to 180 days | 644 (7.4%) | 636 (7.3%) | 0.00 | 647 (5.7%) | 664 (5.9%) | -0.01 | 1,291 (6.4%) | 1,300 (6.5%) | 0.00 | ı |
| prior); n (%) | | | | | | | | | | ı |
| Internal medicine/family medicine visits; n | 7,403 (85.0%) | 7,353 (84.4%) | 0.02 | 9,048 (80.0%) | 9,046 (80.0%) | 0.00 | 16,451 (82.2%) | 16,399 (81.9%) | 0.01 | ı |
| (%) | | | | | | | | | | ı |
| Internal medicine/family medicine visits<br>(30 days prior); n (%) | 4,534 (52.1%) | 4,888 (56.1%) | -0.08 | 5,619 (49.7%) | 5,985 (52.9%) | -0.06 | 10,153 (50.7%) | 10,873 (54.3%) | -0.07 | l |
| Internal medicine/family medicine visits | 6,958 (79.9%) | 6,800 (78.1%) | 0.04 | 8,457 (74.7%) | 8,353 (73.8%) | 0.02 | 15,415 (77.0%) | 15,153 (75.7%) | 0.03 | ı |
| (31 to 180 days prior); n (%) | | | | | | | | | | ı |
| Cardiologist visit; n (%) | 3,601 (41.3%) | 3,542 (40.7%) | 0.01 | 4,416 (39.0%) | 4,297 (38.0%) | 0.02 | 8,017 (40.0%) | 7,839 (39.1%) | 0.02 | ı |
| Number of Cardiologist visits (30 days | 1,590 (18.3%) | 1,519 (17.4%) | 0.02 | 1,996 (17.6%) | 1,963 (17.4%) | 0.01 | 3,586 (17.9%) | 3,482 (17.4%) | 0.01 | ı |
| prior); n (%) | | | | | | | | | | |
| Number of Cardiologist visits (31 to 180 | 2,997 (34.4%) | 2,934 (33.7%) | 0.01 | 3,665 (32.4%) | 3,605 (31.9%) | 0.01 | 6,662 (33.3%) | 6,539 (32.7%) | 0.01 | 1 |
| days prior); n (%) | , , , | | | | | | | | | ı |
| Electrocardiogram ; n (%) | 3,482 (40.0%) | 3,419 (39.3%) | 0.01 | 4,861 (43.0%) | 4,862 (43.0%) | 0.00 | 8,343 (41.7%) | 8,281 (41.4%) | 0.01 | ı |
| Use of glucose test strips; n (%) | 218 (2.5%) | 234 (2.7%) | -0.01 | 247 (2.2%) | 230 (2.0%) | 0.01 | 0,465 (2.3%) | 0,464 (2.3%) | 0.00 | |
| Dialysis; n (%) | 30 (0.3%) | 27 (0.3%) | 0.00 | 66 (0.6%) | 50 (0.4%) | 0.03 | 96 (0.5%) | 77 (0.4%) | 0.01 | ı |
| number of different/distinct medication | | | | | | | | | | ı |
| prescriptions | | | | | | | | | | ı |
| mean (sd) | 11.69 (5.68) | 11.56 (5.05) | 0.02 | 11.97 (5.71) | 11.79 (5.20) | 0.03 | 11.85 (5.70) | 11.69 (5.14) | 0.03 | ı |
| median [IQR] | 11.00 [8.00, 15.00] | 11.00 [8.00, 14.00] | 0.00 | 11.00 [8.00, 15.00] | 11.00 [8.00, 15.00] | 0.00 | 11.00 (5.70) | 11.00 (5.14) | 0.00 | ı |
| Number of Hospitalizations | | | | | | | | | | ı |
| mean (sd) | 0.12 (0.41) | 0.12 (0.39) | 0.00 | 0.19 (0.46) | 0.18 (0.45) | 0.02 | 0.16 (0.44) | 0.15 (0.42) | 0.02 | ı |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.44) | 0.00 (0.42) | 0.00 | ı |
| Number of hospital days | | | | ,, | | | | | | ı |
| mean (sd) | 0.67 (2.94) | 0.62 (2.67) | 0.02 | 1.02 (3.48) | 0.99 (3.54) | 0.01 | 0.87 (3.26) | 0.83 (3.19) | 0.01 | ı |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (3.26) | 0.00 (3.19) | 0.00 | ı |
| Number of Emergency Department (ED) | 0.00 [0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (3.20) | 0.00 (5.25) | 0.00 | ı |
| visits | | | | | | | | | | I |
| mean (sd) | 0.46 (1.16) | 0.45 (1.44) | 0.01 | 0.16 (0.94) | 0.15 (1.17) | 0.01 | 0.29 (1.04) | 0.28 (1.29) | 0.01 | ı |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.04) | 0.00 (1.29) | 0.00 | |
| Number of Office visits | | | | , | | | ,—— , | ,, | | ı |
| mean (sd) | 6.23 (4.59) | 6.10 (4.55) | 0.03 | 6.68 (5.39) | 6.59 (5.03) | 0.02 | 6.48 (5.06) | 6.38 (4.83) | 0.02 | |
| median [IQR] | 5.00 [3.00, 8.00] | 5.00 [3.00, 8.00] | 0.00 | 6.00 [3.00, 9.00] | 6.00 [3.00, 9.00] | 0.00 | 5.57 (5.06) | 5.57 (4.83) | 0.00 | ı |
| Number of Endocrinologist visits | | | | | | | (/ | | | ı |
| mean (sd) | 0.39 (1.97) | 0.39 (2.06) | 0.00 | 0.31 (1.84) | 0.33 (1.88) | -0.01 | 0.38 (1.58) | 0.38 (1.70) | 0.00 | |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.58) | 0.00 (1.70) | 0.00 | |
| Number of internal medicine/family | 2.2.2 (2.2.2) | | | | | | | () | | |
| medicine visits | | | | | | | | | | |
| mean (sd) | 10.92 (15.41) | 10.78 (15.39) | 0.01 | 7.49 (11.92) | 7.40 (10.47) | 0.01 | 8.98 (13.55) | 8.87 (12.84) | 0.01 | |
| median [IQR] | 6.00 [2.00, 14.00] | 6.00 [2.00, 14.00] | 0.00 | 4.00 [1.00, 9.00] | 4.00 [1.00, 9.00] | 0.00 | 4.87 (13.55) | 4.87 (12.84) | 0.00 | |
| Number of Cardiologist visits | | | | | [2.20, 2.00] | | (22.22) | (22.2.) | | |
| mean (sd) | 2.19 (4.98) | 2.13 (4.57) | 0.01 | 2.13 (4.59) | 2.09 (4.48) | 0.01 | 2.16 (4.76) | 2.11 (4.52) | 0.01 | ı |
| median [IQR] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 (4.76) | 0.00 (4.52) | 0.00 | |
| meatan [rejv] | 0.00 [0.00, 2.00] | J.00 [J.00, 2.00] | 0.00 | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | 0.00 | 0.00 (4.70) | 0.00 (4.32) | 0.00 | |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Number electrocardiograms received | I | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 0.78 (1.39) | 0.77 (1.45) | 0.01 | 0.81 (1.36) | 0.79 (1.32) | 0.01 | 0.80 (1.37) | 0.78 (1.38) | 0.01 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 (1.37) | 0.00 (1.38) | 0.00 |
| Number of HbA1c tests ordered | | | | | | | | | |
| mean (sd) | 0.80 (0.93) | 0.80 (0.92) | 0.00 | 0.35 (0.71) | 0.34 (0.72) | 0.01 | 0.55 (0.81) | 0.54 (0.81) | 0.01 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.43 (0.81) | 0.43 (0.81) | 0.00 |
| Number of glucose tests ordered | | | | | | | | | |
| mean (sd) | 0.37 (2.28) | 0.35 (2.21) | 0.01 | 0.23 (0.93) | 0.22 (0.92) | 0.01 | 0.29 (1.66) | 0.28 (1.61) | 0.01 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.66) | 0.00 (1.61) | 0.00 |
| Number of lipid tests ordered | | | | | | | | | |
| mean (sd) | 0.86 (1.05) | 0.85 (0.95) | 0.01 | 0.43 (0.91) | 0.43 (0.90) | 0.00 | 0.62 (0.97) | 0.61 (0.92) | 0.01 |
| median [IQR] | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.43 (0.97) | 0.43 (0.92) | 0.00 |
| Number of creatinine tests ordered | | | | | | | | | |
| mean (sd) | 0.09 (0.49) | 0.08 (0.41) | 0.02 | 0.08 (0.49) | 0.07 (0.39) | 0.02 | 0.08 (0.49) | 0.07 (0.40) | 0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.49) | 0.00 (0.40) | 0.00 |
| Number of BUN tests ordered | | | | | | | | | |
| mean (sd) | 0.06 (0.56) | 0.06 (0.52) | 0.00 | 0.05 (0.46) | 0.06 (0.46) | -0.02 | 0.05 (0.51) | 0.06 (0.49) | -0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.51) | 0.00 (0.49) | 0.00 |
| Number of tests for microal buminuria | | | | | | | | | |
| mean (sd) | 0.59 (1.28) | 0.58 (1.14) | 0.01 | 0.20 (0.69) | 0.19 (0.66) | 0.01 | 0.37 (0.99) | 0.36 (0.90) | 0.01 |
| median [IQR] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.99) | 0.00 (0.90) | 0.00 |
| Total N distinct ICD9/ICD10 diagnoses at | | | | | | | | | |
| the 3rd digit level | | | | | | | | | |
| mean (sd) | 7.82 (9.19) | 7.74 (8.80) | 0.01 | 1.51 (3.92) | 1.44 (3.83) | 0.02 | 4.25 (6.74) | 4.18 (6.48) | 0.01 |
| median [IQR] | 5.00 [0.00, 12.00] | 6.00 [0.00, 12.00] | -0.11 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 2.17 (6.74) | 2.61 (6.48) | -0.07 |
| For PS | 244 (2 004) | 24.4(2.50) | | 250 (2.00) | 254 (2 404) | | 500 (2 50) | 555 (2.204) | |
| Hemorrhagic stroke+Other | 341 (3.9%) | 314 (3.6%) | 0.02 | 358 (3.2%) | 351 (3.1%) | 0.01 | 699 (3.5%) | 665 (3.3%) | 0.01 |
| cerebrovascular disease+Cerebrovascular<br>procedure (for PS); n (%) | | | | | | | | | |
| Occurrence of creatinine tests ordered (for PS); n (%) | 502 (5.8%) | 490 (5.6%) | 0.01 | 520 (4.6%) | 527 (4.7%) | 0.00 | 1,022 (5.1%) | 1,017 (5.1%) | 0.00 |
| Occurrence of BUN tests ordered (for PS); n<br>(%) | 287 (3.3%) | 308 (3.5%) | -0.01 | 336 (3.0%) | 387 (3.4%) | -0.02 | 0,623 (3.1%) | 0,695 (3.5%) | -0.02 |
| Occurrence of chronic renal insufficiency<br>w/o CKD (for PS); n (%) | 756 (8.7%) | 729 (8.4%) | 0.01 | 566 (5.0%) | 550 (4.9%) | 0.00 | 1,322 (6.6%) | 1,279 (6.4%) | 0.01 |
| Chronic kidney disease Stage 1-2 (for PS); n<br>(%) | 421 (4.8%) | 415 (4.8%) | 0.00 | 168 (1.5%) | 178 (1.6%) | -0.01 | 589 (2.9%) | 593 (3.0%) | -0.01 |
| Chronic kidney disease Stage 3-6 (for PS); n | 1,557 (17.9%) | 1,579 (18.1%) | -0.01 | 968 (8.6%) | 941 (8.3%) | 0.01 | 2,525 (12.6%) | 2,520 (12.6%) | 0.00 |
| (%) | 196 (2.3%) | 106 /2 294 | 0.00 | 194 (1.7%) | 193 (1.7%) | 0.00 | 0,390 (1.9%) | 0,389 (1.9%) | 0.00 |
| Bladder stones+Kidney stones (for PS); n<br>(%) | | 196 (2.3%) | | | | | | | |
| Diabetes with peripheral circulatory<br>disorders+Gangrene+Osteomyelitis(for PS)<br>with ICD10; n (%) | 639 (7.3%) | 610 (7.0%) | 0.01 | 303 (2.7%) | 326 (2.9%) | -0.01 | 0,942 (4.7%) | 0,936 (4.7%) | 0.00 |
| Alcohol abuse or dependence+Drug abuse or dependence (for PS); n (%) | 221 (2.5%) | 213 (2.4%) | 0.01 | 70 (0.6%) | 65 (0.6%) | 0.00 | 291 (1.5%) | 278 (1.4%) | 0.01 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Diabetes with other ophthalmic<br>manifestations+Retinal detachment,<br>vitreous hemorrhage, vitrectomy+Retinal | 216 (2.5%) | 213 (2.4%) | 0.01 | 540 (4.8%) | 528 (4.7%) | 0.00 | 0,756 (3.8%) | 0,741 (3.7%) | 0.01 |
|---|---|---|---|---|---|---|---|---|---|
| laser coagulation therapy (for PS); n (%) | () | | | () | | | () | () | |
| Other atherosclerosis+Cardiac conduction<br>disorders+Other CVD (for PS); n (%) | 1,237 (14.2%) | 1,211 (13.9%) | 0.01 | 2,055 (18.2%) | 2,042 (18.0%) | 0.01 | 3,292 (16.4%) | 3,253 (16.2%) | 0.01 |
| Previous cardiac procedure (CABG or PTCA<br>or Stent) + History of CABG or PTCA (for PS)<br>; n (%) | 691 (7.9%) | 675 (7.7%) | 0.01 | 480 (4.2%) | 472 (4.2%) | 0.00 | 1,171 (5.8%) | 1,147 (5.7%) | 0.00 |
| Hyperthyroidism + Hypothyroidism +<br>Other disorders of thyroid gland (for PS); n<br>(%) | 1,914 (22.0%) | 1,834 (21.1%) | 0.02 | 1,123 (9.9%) | 1,165 (10.3%) | -0.01 | 3,037 (15.2%) | 2,999 (15.0%) | 0.01 |
| Delirium + Psychosis (for PS); n (%) | 180 (2.1%) | 186 (2.1%) | 0.00 | 174 (1.5%) | 167 (1.5%) | 0.00 | 354 (1.8%) | 353 (1.8%) | 0.00 |
| Any use of Meglitinides (for PS); n (%) | 72 (0.8%) | 66 (0.8%) | 0.00 | 142 (1.3%) | 164 (1.4%) | -0.01 | 214 (1.1%) | 230 (1.1%) | 0.00 |
| Any use of AGIs (for PS); n (%) | 23 (0.3%) | 13 (0.1%) | 0.04 | 2,055 (18.2%) | 2,042 (18.0%) | 0.01 | 3,292 (16.4%) | 3,253 (16.2%) | 0.01 |
| CKD stage 3-6 + dialysis (for PS); n (%) | 1,560 (17.9%) | 1,580 (18.1%) | -0.01 | 977 (8.6%) | 947 (8.4%) | 0.01 | 2,537 (12.7%) | 2,527 (12.6%) | 0.00 |
| Use of thiazide; n (%) | 2,793 (32.1%) | 2,788 (32.0%) | 0.00 | 3,575 (31.6%) | 3,582 (31.7%) | 0.00 | 11,209 (56.0%) | 11,107 (55.5%) | 0.01 |
| Use of beta blockers; n (%) | 4,837 (55.5%) | 4,821 (55.4%) | 0.00 | 6,372 (56.3%) | 6,286 (55.6%) | 0.01 | 13,631 (68.1%) | 13,607 (68.0%) | 0.00 |
| Use of calcium channel blockers; n (%) | 6,196 (71.1%) | 6,156 (70.7%) | 0.01 | 7,435 (65.7%) | 7,451 (65.9%) | 0.00 | 7,859 (39.2%) | 7,759 (38.7%) | 0.01 |
| All antidiabetic medications except<br>Insulin; n (%) | 3,652 (41.9%) | 3,607 (41.4%) | 0.01 | 4,207 (37.2%) | 4,152 (36.7%) | 0.01 | 6,368 (31.8%) | 6,370 (31.8%) | 0.00 |
| DM Medications - Insulin ; n (%) | 1,491 (17.1%) | 1,467 (16.8%) | 0.01 | 1,865 (16.5%) | 1,861 (16.4%) | 0.00 | 3,356 (16.8%) | 3,328 (16.6%) | 0.01 |
| Use of Low Intensity Statins; n (%) | 2,845 (32.7%) | 2,886 (33.1%) | -0.01 | 3,842 (34.0%) | 3,834 (33.9%) | 0.00 | 6687 (33.4%) | 6,720 (33.6%) | 0.00 |
| Use of High Intensity Statins; n (%) | 2,931 (33.7%) | 2,856 (32.8%) | 0.02 | 2,976 (26.3%) | 2,846 (25.2%) | 0.03 | 5907 (29.5%) | 5,702 (28.5%) | 0.02 |
| Malignant hypertension; n (%) | 288 (3.3%) | 271 (3.1%) | 0.01 | 5,093 (45.0%) | 5,127 (45.3%) | -0.01 | 5381 (26.9%) | 5,398 (27.0%) | 0.00 |
| Cardiovascular stress test; n (%) | 21 (0.2%) | 23 (0.3%) | -0.02 | 49 (0.4%) | 50 (0.4%) | 0.00 | 0,070 (0.3%) | 73 (0.4%) | -0.02 |
| Echocardiogram; n (%) | 1,165 (13.4%) | 1,125 (12.9%) | 0.01 | 2,534 (22.4%) | 2,440 (21.6%) | 0.02 | 3,699 (18.5%) | 3565 (17.8%) | 0.02 |
| Number of BNP tests | | | | | | | | | |
| mean (sd) | 0.07 (0.33) | 0.07 (0.34) | 0.00 | 0.05 (0.28) | 0.04 (0.27) | 0.04 | 0.06 (0.30) | 0.05 (0.30) | 0.03 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.30) | 0.00 (0.30) | 0.00 |
| Number of Cardiac biomarkers tests | | | | | | | | | |
| (tropnin, CK-MBs, Myoglobin, CPK) | | | | | | | | | |
| mean (sd) | 0.22 (0.90) | 0.21 (0.88) | 0.01 | 0.19 (0.98) | 0.19 (0.97) | 0.00 | 0.20 (0.95) | 0.20 (0.93) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.95) | 0.00 (0.93) | 0.00 |
| Number of Ambulatory Blood pressure<br>monitoring tests | | | | | | | | | |
| mean (sd) | 0.00 (0.05) | 0.00 (0.05) | 0.00 | 0.00 (0.09) | 0.00 (0.07) | 0.00 | 0.00 (0.08) | 0.00 (0.06) | 0.00 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.08) | 0.00 (0.06) | 0.00 |
| N of days on antihypertensive medications | | | | | | | | | |
| during baseline | | | | | | | | | |
| mean (sd) | 155.87 (43.03) | 156.52 (45.30) | -0.01 | 152.05 (46.71) | 151.49 (48.30) | 0.01 | 153.71 (45.15) | 153.68 (47.02) | 0.00 |
| median [IQR] | 176.00 [154.00,<br>181.00] | 179.00 [158.00,<br>181.00] | -0.07 | 175.00 [147.00,<br>181.00] | 177.00 [145.00,<br>181.00] | -0.04 | 175.43 (45.15) | 177.87 (47.02) | -0.05 |
| N of days in database anytime prior | | | | | | | | | |
| mean (sd) | 1,982.37 (1,425.64) | 2,002.50 (1,451.47) | -0.01 | 1,709.38<br>(1,080.10) | 1,702.87<br>(1,073.43) | 0.01 | 1828.12 (1242.27) | 1833.20 (1251.97) | 0.00 |
| median [IQR] | 1,617.50 [867.00,<br>2,699.25] | 1,612.00 [873.75,<br>2,761.00] | 0.00 | 1,508.50 [840.00,<br>2,387.00] | 1,520.50 [821.75,<br>2,445.25] | -0.01 | 1555.91 (1242.27) | 1560.30 (1251.97) | 0.00 |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| Mean Copay for per prescription cost | ı | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| (charges in U.S. \$) (180-1 day prior) | | | | | | | | | |
| mean (sd) | 27.14 (36.65) | 27.51 (33.53) | -0.01 | 25.60 (26.67) | 25.50 (26.82) | 0.00 | 26.27 (31.40) | 26.37 (29.92) | 0.00 |
| median [IQR] | | 18.64 [7.23, 35.71] | 0.00 | | 20.00 [7.97, 35.00] | 0.00 | 19.49 (31.40) | 19.41 (29.92) | 0.00 |
| median [idk] | 18.62 [7.00, 35.26] | 18.64 [7.23, 35.71] | 0.00 | 20.16 [8.57, 35.34] | 20.00 [7.57, 35.00] | 0.01 | 19.49 (31.40) | 19.41 (29.92) | 0.00 |
| Missing; n (%) | 33 (0.4%) | 40 (0.5%) | -0.01 | 25 (0.2%) | 28 (0.2%) | 0.00 | 0,058 (0.3%) | 68 (0.3%) | 0.00 |
| Colonos; n (%) | 427 (4.9%) | 434 (5.0%) | 0.00 | 637 (5.6%) | 607 (5.4%) | 0.01 | 1,064 (5.3%) | 1041 (5.2%) | 0.00 |
| Fecal occult blood (FOB) test; n (%) | 388 (4.5%) | 390 (4.5%) | 0.00 | 345 (3.0%) | 368 (3.3%) | -0.02 | 0,733 (3.7%) | 758 (3.8%) | -0.01 |
| Flu vaccine; n (%) | 1,619 (18.6%) | 1,601 (18.4%) | 0.01 | 1,188 (10.5%) | 1,207 (10.7%) | -0.01 | 2,807 (14.0%) | 2808 (14.0%) | 0.00 |
| Mammogram; n (%) | 1,128 (13.0%) | 1,166 (13.4%) | -0.01 | 1,297 (11.5%) | 1,371 (12.1%) | -0.02 | 2,425 (12.1%) | 2537 (12.7%) | -0.02 |
| Pap smear; n (%) | 278 (3.2%) | 281 (3.2%) | 0.00 | 445 (3.9%) | 458 (4.0%) | -0.01 | 0,723 (3.6%) | 739 (3.7%) | -0.01 |
| Pneumonia vaccine; n (%) | 1,425 (16.4%) | 1,411 (16.2%) | 0.01 | 326 (2.9%) | 322 (2.8%) | 0.01 | 1,751 (8.7%) | 1733 (8.7%) | 0.00 |
| PSA test or Prostate exam for DRE; n (%) | 1,117 (12.8%) | 1,120 (12.9%) | 0.00 | 827 (7.3%) | 861 (7.6%) | -0.01 | 1,944 (9.7%) | 1981 (9.9%) | -0.01 |
| Bone mineral density; n (%) | 425 (4.9%) | 431 (4.9%) | 0.00 | 352 (3.1%) | 353 (3.1%) | 0.00 | 0,777 (3.9%) | 784 (3.9%) | 0.00 |
| Use of Sympatomimetic agents; n (%) | 72 (0.8%) | 80 (0.9%) | -0.01 | 230 (2.0%) | 219 (1.9%) | 0.01 | 0,302 (1.5%) | 299 (1.5%) | 0.00 |
| Use of CNS stimulants; n (%) | 59 (0.7%) | 54 (0.6%) | 0.01 | 92 (0.8%) | 98 (0.9%) | -0.01 | 0,151 (0.8%) | 152 (0.8%) | 0.00 |
| Use of estrogens, progestins, androgens; n | 390 (4.5%) | 382 (4.4%) | 0.00 | 791 (7.0%) | 805 (7.1%) | 0.00 | 1,181 (5.9%) | 1187 (5.9%) | 0.00 |
| (%) | | | | | | | | | |
| Use of Angiogenesis inhibitors; n (%) | 5 (0.1%) | 1 (0.0%) | 0.04 | 20 (0.2%) | 6 (0.1%) | 0.03 | 0,025 (0.1%) | 7 (0.0%) | 0.04 |
| Use of Oral Immunosuppressants; n (%) | 54 (0.6%) | 31 (0.4%) | 0.03 | 137 (1.2%) | 54 (0.5%) | 0.08 | 0,191 (1.0%) | 85 (0.4%) | 0.07 |
| Cardiomegaly, LVH, and other cardiopathy | | 1,120 (12.9%) | 0.02 | 1,219 (10.8%) | 1,179 (10.4%) | 0.01 | 2,406 (12.0%) | 2299 (11.5%) | 0.02 |
| due to hypertension; n (%) | , , , | , , , | | , , , | , , , | | , , , | | |
| Ultrasound; n (%) | 1,728 (19.8%) | 1,704 (19.6%) | 0.01 | 2,845 (25.1%) | 2,813 (24.9%) | 0.00 | 4,573 (22.8%) | 4517 (22.6%) | 0.00 |
| Symptomatic hypotension; n (%) | 154 (1.8%) | 149 (1.7%) | 0.01 | 158 (1.4%) | 146 (1.3%) | 0.01 | 0,312 (1.6%) | 295 (1.5%) | 0.01 |
| Syncopal episodes; n (%) | 208 (2.4%) | 220 (2.5%) | -0.01 | 186 (1.6%) | 187 (1.7%) | -0.01 | 0,394 (2.0%) | 407 (2.0%) | 0.00 |
| N of Generic name drugs only | ` ' | . , | | . , | . , | | | | |
| mean (sd) | 19.00 (13.93) | 18.89 (14.40) | 0.01 | 13.94 (10.10) | 13.66 (10.69) | 0.03 | 16.14 (11.92) | 15.93 (12.44) | 0.02 |
| median [IQR] | | 16.00 [10.00, 24.00] | 0.00 | 12.00 [7.00, 18.00] | | 0.10 | 13.74 (11.92) | 13.17 (12.44) | 0.05 |
| N of Brand name drugs only | | | | | | | | | |
| mean (sd) | 5.64 (7.16) | 5.56 (7.28) | 0.01 | 8.82 (7.98) | 8.68 (8.29) | 0.02 | 7.44 (7.63) | 7.32 (7.87) | 0.02 |
| median [IQR] | 3.00 [1.00, 8.00] | 3.00 [0.00, 8.00] | 0.00 | 7.00 [3.00, 12.00] | 7.00 [3.00, 12.00] | 0.00 | 5.26 (7.63) | 5.26 (7.87) | 0.00 |
| Number of distinct antihypertensive | | | | | | | | | |
| generic medications (180-1 days before | | | | | | | | | |
| index) | | | | | | | | | |
| mean (sd) | 3.06 (1.28) | 3.04 (1.51) | 0.01 | 2.95 (1.26) | 2.90 (1.58) | 0.03 | 3.00 (1.27) | 2.96 (1.55) | 0.03 |
| median [IQR] | 3.00 [2.00, 4.00] | 3.00 [2.00, 4.00] | 0.00 | 3.00 [2.00, 4.00] | 3.00 [2.00, 4.00] | 0.00 | 3.00 (1.27) | 3.00 (1.55) | 0.00 |
| Number of distinct antihypertensive | | | | | | | | | |
| generic medications on CED | | | | | | | | | _ |
| mean (sd) | 0.10 (0.39) | 1.39 (0.74) | -2.18 | 0.12 (0.44) | 1.47 (0.80) | -2.09 | 0.11 (0.42) | 1.44 (0.77) | -2.14 |
| median [IQR] | 0.00 [0.00, 0.00] | 1.00 [1.00, 2.00] | -1.69 | 0.00 [0.00, 0.00] | 1.00 [1.00, 2.00] | -1.55 | 0.00 (0.42) | 1.00 (0.77) | -1.61 |
| Hypertensive retinopathy; n (%) | 142 (1.6%) | 142 (1.6%) | 0.00 | 69 (0.6%) | 65 (0.6%) | 0.00 | 0 | 0 | #VALUE! |
| Commercial vs Medicare Advantage- | | | | | | | | | |
| Business Type Code - CORRECT ONE -<br>TRUVEN | | | | | | | | | |
| Commercial; n (%) | 2,354 (27.0%) | 2,352 (27.0%) | 0.00 | 7,423 (65.6%) | 7,408 (65.5%) | 0.00 | 9,777 (48.8%) | 9760 (48.7%) | 0.00 |
| Medicare Advantage; n (%) | 6,356 (73.0%) | 6,358 (73.0%) | 0.00 | 3,891 (34.4%) | 3,906 (34.5%) | 0.00 | 10,247 (51.2%) | 10264 (51.3%) | 0.00 |
| Commercial vs Medicare Advantage- | | - | | • | - | | | | |
| Business Type Code | | | | | | | | | |
| | • | | | | | | | | |

Table 1: Telmisartan vs Loop/Dihydropyridines/Thiazides

| COM = COMMERCIAL; n (%) | 2,354 (27.0%) | 2,352 (27.0%) | 0.00 | - | - | #VALUE! | 2,354 (27.0%) | 2,352 (27.0%) | 0.00 |
|---|---|---|---|---|---|---|---|---|---|
| MCR = MEDICARE; n (%) | 6,356 (73.0%) | 6,358 (73.0%) | 0.00 | - | - | #VALUE! | 6,356 (73.0%) | 6,358 (73.0%) | 0.00 |
| MCD = MEDICAID; n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| NONE = NO BUSINESS LINE CODE (added | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| in 2015); n (%) | | | | | | | | | |
| UNK = UNKNOWN (added in 2015); n (%) | 0 (0.0%) | 0 (0.0%) | #DIV/0! | - | - | #VALUE! | 0 (0.0%) | 0 (0.0%) | #DIV/0! |
| Commercial vs Medicare Advantage- Data | _ | _ | #VALUE! | 0 | 0 | #VALUE! | 0 | 0 | #VALUE! |
| Type | | | | | | | | | |
| 1 - Fee For Service; n (%) | - | - | #VALUE! | 3,524 (31.1%) | 3,538 (31.3%) | 0.00 | 3,524 (31.1%) | 3,538 (31.3%) | 0.00 |
| 2 - Encounter; n (%) | - | - | #VALUE! | 367 (3.2%) | 368 (3.3%) | -0.01 | 367 (3.2%) | 368 (3.3%) | -0.01 |
| 3 - Medicare; n (%) | - | - | #VALUE! | 6,985 (61.7%) | 6,939 (61.3%) | 0.01 | 6,985 (61.7%) | 6,939 (61.3%) | 0.01 |
| 4 - Medicare Encounter; n (%) | - | - | #VALUE! | 438 (3.9%) | 469 (4.1%) | -0.01 | 438 (3.9%) | 469 (4.1%) | -0.01 |
| Metropolitan Statistical Area - Urban (any | | | | | | | | | |
| MSA) vs Rural (non-MSA) | | | | | | | | | |
| Urban; n (%) | - | - | #VALUE! | 8,502 (75.1%) | 8,576 (75.8%) | -0.02 | 8,502 (75.1%) | 8,576 (75.8%) | -0.02 |
| Rural; n (%) | - | - | #VALUE! | 68 (0.6%) | 68 (0.6%) | 0.00 | 68 (0.6%) | 68 (0.6%) | 0.00 |
| Unknown/Missing; n (%) | - | - | #VALUE! | 2,744 (24.3%) | 2,670 (23.6%) | 0.02 | 2,744 (24.3%) | 2,670 (23.6%) | 0.02 |